#### The GlaxoSmithKline group of companies

207660

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title

: Reporting and Analysis Plan for A phase III study (a placebo controlled, randomized, double-blind comparative study and an open-label, uncontrolled study) to evaluate the efficacy and safety of GSK1358820 in patients with post-stroke upper limb spasticity.

Compound Number

: GSK1358820

Effective Date

: 02-APR-2018

# **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 207660.
- This RAP is intended to describe the efficacy and safety analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the interim and final Statistical Analysis Complete (SAC) deliverable.

#### **RAP Author(s):**

| Approver | Date | Approval Method |
|-------------------------------------------|------|-----------------|
| PPD | | |
| Lead Statistician (Biostatistics Group 2, | | |
| Biomedical Data Sciences Dept., Japan) | | |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

207660

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Japan Project Lead (Future Pipelines Discovery Office, Medicines Development, Japan) | 23-MAR-2018 | eSignature |
| Clinical Investigations Lead (Future Pipelines Discovery Office, Medicines Development, Japan) | 23-MAR-2018 | eSignature |
| Operations and Science Lead (6, Clinical Operations Dept., Japan) | 23-MAR-2018 | eSignature |
| Data Quality Lead (Data Practice Group,<br>Biomedical Data Sciences Dept., Japan) | 28-MAR-2018 | eSignature |
| Medical Writer (2, Medical Writing Office, Medicines Development, Japan) | 27-MAR-2018 | eSignature |
| Lead Programmer (Statistical Programming & Reporting Group, Biomedical Data Sciences Dept., Japan) | 28-MAR-2018 | eSignature |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Manager (Biostatistics Group 2, Biomedical Data Sciences Dept., Japan) | 28-MAR-2018 | eSignature |
| Department Manager (Biomedical Data Sciences | 02-APR-2018 | eSignature |
| Dept., Japan) | | |

207660

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | DDUCTION | 6 |
| | 1.1. | Summary of Key Protocol Information | |
| | | 1.1.1. Changes to the Protocol Defined Statistical Analysis Plan | |
| | | 1.1.2. Study Objective(s) and Endpoint(s) | |
| | | 1.1.3. Study Design | <mark>7</mark> |
| | | 1.1.4. Statistical Hypotheses / Statistical Analyses | 8 |
| _ | | | |
| 2. | | NED ANALYSES | |
| | 2.1. | Interim Analyses | |
| | 2.2. | Final Analyses | 9 |
| 3. | ANAL | YSIS POPULATIONS | 9 |
| | 3.1. | Protocol Deviations | 10 |
| | 00110 | | |
| 4. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING<br>/ENTIONS | 11 |
| | 4.1. | Study Treatment & Sub-group Display Descriptors | |
| | 4.1.<br>4.2. | Baseline Definitions | 11 |
| | 4.3. | Multicentre Studies | |
| | 4.4. | Examination of Covariates, Other Strata and Subgroups | |
| | 7.7. | 4.4.1. Covariates and Other Strata | |
| | | 4.4.2. Examination of Subgroups | |
| | 4.5. | Multiple Comparisons and Multiplicity | |
| | 4.6. | Other Considerations for Data Analyses and Data Handling | |
| | | Conventions | 12 |
| _ | CTUD | NY DODUH ATION ANALYSES | 40 |
| 5. | 5.1. | Y POPULATION ANALYSES Overview of Planned Study Population Analyses | 13 |
| | 5.1.<br>5.2. | Participant Disposition and Population | |
| | 5.2.<br>5.3. | Protocol Deviation | |
| | 5.3.<br>5.4. | Demographic and Baseline Characteristics | |
| | 5. <del>4</del> .<br>5.5. | Prior and Concomitant Medications | |
| | 5.6. | Rehabilitation | |
| | 5.0. | Tonabilitation | |
| 6. | EFFIC | CACY ANALYSES | 15 |
| | 6.1. | Primary Efficacy Analyses | 15 |
| | | 6.1.1. Endpoint / Variables | 15 |
| | | 6.1.2. Summary Measure | 15 |
| | | 6.1.3. Population of Interest | |
| | | 6.1.4. Strategy for Intercurrent (Post-Randomization) Events | 15 |
| | | 6.1.5. Statistical Analyses / Methods | |
| | | 6.1.5.1. Statistical Methodology Specification | |
| | 6.2. | Secondary Efficacy Analyses | |
| | | 6.2.1. Endpoint / Variables | |
| | | 6.2.2. Summary Measure | |
| | | 6.2.3. Population of Interest | |
| | | 6.2.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 6.2.5 Statistical Analyses / Methods | 17 |

| | | 2 | 207660 |
|---|---|---|---|
| | | 6.2.5.1. Statistical Methodology Specification | 18 |
| | 6.3. | Exploratory Efficacy Analyses | |
| | | 6.3.1. Modified Ashworth Scale (MAS) | 18 |
| | | 6.3.2. Numeric Rating Scale (NRS) for pain | |
| | | 6.3.3. Disability Assessment Scale (DAS) | 19 |
| | | 6.3.4. Clinical Global Impression of Change (CGI) of functional | |
| | | disability | |
| | | 6.3.5. Patient-Reported Benefit of Injection | 19 |
| | | 6.3.6. Time to Patient-Reported Onset of Spasticity Symptom | |
| | | Relief | |
| | | 6.3.7. Time to Qualification for Retreatment | 20 |
| 7. | SAFE | TY ANALYSES | 20 |
| | 7.1. | Adverse Events Analyses | |
| | 7.2. | Adverse Events of Special Interest Analyses | |
| | 7.3. | Clinical Laboratory Analyses | |
| | 7.4. | Other Safety Analyses | |
| | 7.5. | Exposure | |
| | | · | |
| 8. | REFE | RENCES | 25 |
| 9. | APPE | NDICES | 26 |
| - | 9.1. | Appendix 1: Protocol Deviation Management and Definitions for Per | |
| | 0 | Protocol Population | 26 |
| | 9.2. | Appendix 2: Schedule of Activities | |
| | 0.2. | 9.2.1. Protocol Defined Schedule of Events | |
| | 9.3. | Appendix 3: Assessment Windows | |
| | 9.4. | Appendix 4: Study Phases and Treatment Emergent Adverse | |
| | 0 | Events | 31 |
| | | 9.4.1. Study Phases for Concomitant Medication | |
| | | 9.4.2. Study Phases for Adverse Events | 31 |
| | | 9.4.2.1. Definition of Adverse Events of Special Interest | |
| | 9.5. | Appendix 5: Data Display Standards & Handling Conventions | |
| | 0.0. | 9.5.1. Reporting Process | 32 |
| | | 9.5.2. Reporting Standards | |
| | 9.6. | Appendix 6: Derived and Transformed Data | |
| | 0.0. | 9.6.1. General | |
| | | 9.6.2. Study Population | |
| | | 9.6.3. Efficacy | |
| | 9.7. | Appendix 7: Reporting Standards for Missing Data | |
| | 0.7. | 9.7.1. Premature Withdrawals | |
| | | 9.7.2. Handling of Missing Data | |
| | | 9.7.2.1. Handling of Missing and Partial Dates | |
| | 9.8. | Appendix 8: Values of Potential Clinical Importance | |
| | 9.9. | Appendix 9: Population Pharmacokinetic (PopPK) Analyses | |
| | 9.9.<br>9.10. | Appendix 9: Population Pharmacokinetic (PopPK) Analyses | |
| | 9.10.<br>9.11. | Appendix 10: Pharmacokinetic / Pharmacodynamic Arialyses | ۸۵ |
| | y. 11. | 9.11.1. Abbreviations | |
| | 0.40 | | |
| | 9.12. | 11 | |
| | | 9.12.1. Data Display Numbering | |
| | | 9.12.2. Mock Example Shell Referencing | 42 |

| | | | 207660 |
|---|---|---|---|
| | 9.12.3. | Deliverables | 42 |
| | 9.12.4. | Study Population Tables | 43 |
| | | 9.12.4.1. Interim Analyses | 43 |
| | | 9.12.4.2. Final Analyses | 44 |
| | 9.12.5. | | |
| | | 9.12.5.1. Interim Analyses | 45 |
| | | 9.12.5.2. Final Analyses | |
| | 9.12.6. | Efficacy Figures | 53 |
| | | 9.12.6.1. Interim Analyses | |
| | | 9.12.6.2. Final Analyses | 57 |
| | 9.12.7. | | 61 |
| | | 9.12.7.1. Interim Analyses | 61 |
| | | 9.12.7.2. Final Analyses | |
| | 9.12.8. | Safety Figures | 79 |
| | | 9.12.8.1. Interim Analyses | 79 |
| | 9.12.9. | ICH Listings | 80 |
| | | 9.12.9.1. Interim Analyses | |
| | | 9.12.9.2. Final Analyses | 83 |
| 9.13. | Appendi | x 13: List of Preferred Terms / System Organ Class of | |
| | Adverse | Events of Special Interest | 87 |
| | | Convulsions and Seizures | |
| | 9.13.2. | | |
| | 9.13.3. | Possible Distant Spread of Toxin | 87 |

207660

# 1. INTRODUCTION

# 1.1. Summary of Key Protocol Information

# 1.1.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol amendment 02 [(Dated: 06OCT2017)].

# 1.1.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate the efficacy of the injections of 400 units of the product at Week 6 (finger/ wrist flexors: 240 units, elbow flexors: 160 units), comparing to that of 240 units (finger/ wrist flexors: 240 units, elbow flexors: placebo). | The responder rate: The rate of the participants that Modified Ashworth Scale (MAS) score was reduced at least 1 from baseline in the elbow flexors. |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the efficacy of 400 units of the product, comparing to 240 units of the product | <ul> <li>The responder rate of MAS score from baseline in the finger, thumb and wrist flexors</li> <li>Changes in MAS score from baseline in the finger, thumb, wrist and elbow flexors</li> <li>Changes in Disability Assessment Scale (DAS) from baseline</li> </ul> |
| To evaluate the safety and | Adverse events |
| tolerability of the product of 400 | Physical examinations |
| units, comparing to 240 units of the product/ To evaluate the safety and | Clinical laboratory tests (haematology, blood biochemistry, urinalysis) |
| tolerability of 400 units of the product | <ul> <li>Vital signs (heart rate, blood pressure, body temperature)</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| To evaluate the efficacy of 400 units of the product | <ul> <li>Changes in MAS score from baseline in finger,<br/>thumb, wrist, elbow, pronation of the forearm and<br/>shoulder flexors</li> </ul> |
| To evaluate the other efficacy of<br>the product of 400 units, comparing | Changes in Numeric Rating Scale (NRS) for pain from baseline |
| to 240 units of the product/ To | Changes in other items of DAS from baseline |
| evaluate the other efficacy of 400 | Clinical Global Impression of Change (CGI) of |
| units of the product | functional disability by an investigator |
| | CGI of functional disability by a patient |
| | Time to patient-reported onset of spasticity symptom relief |
| | Patient-reported benefit of injection |
| | Time to qualification for retreatment |

207660

| Objectives | Endpoints |
|-----------------------------------|-----------------------------------|
| To evaluate neutralizing antibody | Testing for neutralizing antibody |
| production | |

## 1.1.3. Study Design



207660

| Overview of S | Overview of Study Design and Key Features |
|---|---|
| Treatment<br>Assignment | <ul> <li>Number of participants (randomized participants): 120 (60 per group)</li> <li>GSK RandAll NG will be used to generate the randomization schedule.</li> <li>The randomization will be stratified by the MAS score (3 or 4) in the elbow flexors at Day1</li> </ul> |
| Interim<br>Analysis | Interim analysis is planned in this study as described in 3.1. |

# 1.1.4. Statistical Hypotheses / Statistical Analyses

No formal hypothesis will not be tested.

# 2. PLANNED ANALYSES

# 2.1. Interim Analyses

The interim planned primary analyses will be performed after the completion of the following sequential steps:

1. All participants (except for early termination) complete the visit at Week 24 of the initial dose as defined in the protocol. The participants who complete that visit are defined as below.

The participant is re-treated at Week 12 visit in Blind Phase and completes the Week 12 visit in Open-label Phase.

The participant is re-treated at Week 16 visit in Blind Phase and completes the Week 12 visit in Open-label Phase.

The participant is re-treated at Week 20 visit in Blind Phase and completes the Week 4 visit in Open-label Phase.

The participant completes the Week 24 visit in Blind Phase.

- 2. All required database cleaning activities have been completed and interim database release and database freeze has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG procedures.
- 5. Interim analyses will be performed.

The interim analyses will be performed for regulatory submission. However subject level data will not be disclosed to people who work at the sites including investigators.

All planned interim analyses (i.e. Study population, Efficacy and Safety analyses) will be performed using data up to Week 24 visit for all participants.

For Adverse Events, Cardiovascular Events, Liver Events and Medication, the data up to Week 24 visit is defined by using the start date. If the start date of these data is earlier

207660

than or same as the date of Week 24 visit defined above, these data will be included in the data up to Week 24 visit. Otherwise the data will not.

# 2.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. Final analyses will be performed.

# 3. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | Comprise of all screened participants | Study Population |
| Enrolled | Comprise of all participants who meet the eligibility criteria at a screening and Day 1 visit. | Study Population |
| Intent-To-Treat 1 | This population consists of all participants who | Study Population |
| (ITT1) | are randomized in the study and who have at least 1 post-baseline efficacy assessment: | Efficacy |
| | ITT is the primary efficacy analysis population,<br>and the participants will be analyzed in line<br>with the randomized treatment group | |
| | Any participant who receives a study treatment<br>randomization number will be considered to<br>have been randomized. | |
| ITT2 | This population consists of all participants in | Study Population |
| | ITT1 population, who have at least 2 study treatments and who have at least 1 efficacy assessment after the 2nd treatment. | Efficacy |
| ITT3 | This population consists of all participants in | Study Population |
| | ITT2 population, who have at least 3 study treatments and who have at least 1 efficacy assessment after the 3rd treatment. | Efficacy |
| ITT4 | This population consists of all participants in | Study Population |
| | ITT3 population, who have <b>4</b> study treatments and who have at least 1 efficacy assessment after the 4th treatment. | Efficacy |

207660

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Safety1 | This population consists of all participants who are randomized in the study and who receive study treatment at least once | Safety |
| | The participants will be analyzed based on the treatment actually given. | |
| Safety2 | This population consists of all participants in<br>Safety1 population, who receive study<br>treatment at least twice. | Safety |
| | The participants will be analyzed based on the treatment actually given. | |
| Safety3 | This population consists of all participants who are randomized in the study and who receive study treatment at least three times | Safety |
| | The participants will be analyzed based on the treatment actually given. | |
| Safety4 | This population consists of all participants in<br>Safety1 population, who receive study<br>treatment four times. | Safety |
| | The participants will be analyzed based on the treatment actually given. | |

#### NOTES:

 Please refer to Appendix 12: List of Data Displays which details the population to be used for each displays being generated.

#### 3.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided. This listing will be based on data as recorded on the inclusion/exclusion page of the eCRF.

207660

# 4. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 4.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| | RandAll NG Data Displays for Reporting | | |
| Code | Description | Description | Order in TLF |
| Α | GSK1358820 240U | GSK1358820 240U | 1 |
| В | GSK1358820 400U | GSK1358820 400U | 2 |

Treatment comparisons will be displayed as follows using the descriptors as specified:

1. GSK1358820 400U vs GSK1358820 240U

### 4.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline. These baseline values will be used for all analyses in both Blind Phase and Open Label Phase.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

#### 4.3. Multicentre Studies

No data will be analysed by center.

## 4.4. Examination of Covariates, Other Strata and Subgroups

#### 4.4.1. Covariates and Other Strata

The list of covariates and other strata may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses. Additional covariates and other strata of clinical interest may also be considered.

| Category | Details |
|-----------------------|-----------------------------|
| Strata and Covariates | Baseline MAS value (3 or 4) |

## 4.4.2. Examination of Subgroups

The list of subgroups may be used in descriptive summaries and statistical analyses. Additional subgroups of clinical interest may also be considered.

207660

- If the percentage of participants is small within a particular subgroup, then the subgroup categories may be refined prior to unblinding the trial.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.

| Subgroup | Categories |
|---|---|
| Baseline MAS value | 3 or 4 |
| Baseline Rehabilitation | |
| Task-specific practice | Yes, or No |
| Muscle strengthening exercise | The subgroup analyses will be conducted by each rehabilitation use. |
| Stretching/Range of motion | |
| exercise | |
| Splinting/Orthoses | |
| Taping | |
| Positioning aids | |

# 4.5. Multiple Comparisons and Multiplicity

No multiplicity adjustment is considered in this study because no statistical hypothesis will be tested.

# 4.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|-------------|----------------------------------------------------------------|
| Section 9.3 | Appendix 3: Assessment Windows |
| Section 9.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| Section 9.5 | Appendix 5: Data Display Standards & Handling Conventions |
| Section 9.6 | Appendix 6: Derived and Transformed Data |
| Section 9.7 | Appendix 7: Reporting Standards for Missing Data |
| Section 9.8 | Appendix 8: Values of Potential Clinical Importance |

207660

#### 5. STUDY POPULATION ANALYSES

# 5.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Screened, Enrolled and ITT populations, unless otherwise specified.

Study population analyses including analyses of participant's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and rehabilitations will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 12: List of Data Displays.

# 5.2. Participant Disposition and Population

The number and percentage of those participants below will be presented by treatment group and total.

- Participants who completed the Week 24 and who withdrew early from study by Week 24 (including the reasons for early withdrawal)
- Participants who completed the study and who withdrew early from study (including the reasons for early withdrawal)
- Participants who passed screening and who failed screening (including the reasons for screen failure)
- Participants at each centre
- Participants included in each population defined in the Section 3.

These items below will be listed.

- The reasons for early withdrawal and screen failure.
- Participants who were rescreened.
- Participants for whom the treatment blind was broken.
- Planned and actual treatments
- Participants excluded from any population defined in the Section 3.

#### 5.3. Protocol Deviation

The number and percentage of participants with important protocol deviation will be presented by treatment group. This summary will not include subcategories

Important protocol deviations and participants with inclusion/exclusion criteria deviation will be listed.

# 5.4. Demographic and Baseline Characteristics

These parameters as below will be summarized by treatment group and total.

• Demographic data (age, sex, ethnicity, weight, height, body mass index(BMI), race and racial combinations)

207660

- Baseline Efficacy Parameter
  - Modified Ashworth Scales in finger, thumb, wrist, elbow, pronation of forearm and shoulder flexors.
  - o Numeric Rating Scale for pain
  - o Disability Assessment Scale (Main Assessment Parameter)
  - o Disability Assessment Scale (Hygiene, Pain, Dressing and Limb posture)
  - The selected item as a Main Assessment Parameter of DAS out of the 4 items
    - Hygiene
    - Pain
    - Dressing
    - Limb posture

### 5.5. Prior and Concomitant Medications

All medication used in this study will be coded according to drug name as defined in the GSK Drug Dictionary. The relationship between the ATC level 1 and ingredient will be summarized for the all prior and concomitant medications, respectively.

## 5.6. Rehabilitation

Screening

The number and percentage of Rehabilitations will be presented.

• Treatment phase

The category and frequency of Rehabilitations will be collected on eCRF. The number and percentage of each Rehabilitation will be presented in Blind Phase. The category and frequency of Rehabilitations in all treatment phase will be listed.

• Category and Frequency

The categories of Rehabilitation are as below:

- Task-specific practice
- Muscle strengthening exercise
- Stretching/Range of motion exercise
- Splinting/Orthoses
- Taping
- Positioning aids

207660

#### • Other

The category of frequency which will be collected on CRF is defined as below:

- No practice
- $\circ$  > 8 days per month
- $\circ$  > 8 and  $\leq$  16 days per month
- $\circ$  > 16 and  $\leq$  24 days per month
- $\circ$  > 24 days per month

## 6. EFFICACY ANALYSES

# 6.1. Primary Efficacy Analyses

## 6.1.1. Endpoint / Variables

The primary endpoint is the responder rate of MAS score.

# 6.1.2. Summary Measure

The summary measure is the difference in the responder rate of MAS score.

#### 6.1.3. Population of Interest

The primary efficacy analyses will be based on the Intent-To-Treat 1 population, unless otherwise specified.

## 6.1.4. Strategy for Intercurrent (Post-Randomization) Events

Intercurrent event: early withdrawal from study

Strategy: if MAS score is missing because of an early withdrawal from the study, the participant will be regarded as a non-responder.

#### 6.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 6.1.1 will be summarised using descriptive statistics and listed.

207660

### 6.1.5.1. Statistical Methodology Specification

### **Endpoint / Variables**

Responder Rate of MAS in the elbow flexors at Week 6 of the initial dose

#### **Model Specification**

- To summarize the primary endpoint without statistical model
  - The primary endpoint will be calculated as the proportion of participants whose MAS score decreased by at least 1 level from the baseline in the ITT1 population.
  - The intergroup difference in the responder rate and its 95% confidence interval (Waldtype) will be computed.

#### **Data Convention**

• The MAS scores, 0, 1, 1+, 2, 3 and 4 will be encoded to 0, 1, 2, 3, 4 and 5, respectively, for the analyses.

# **Definition of Responder and Responder rate**

"Responder" is defined as a participant whose MAS score decrease by at least 1 level from the baseline.

Responder Rate will be calculated as below.

Responder Rate (%) = (Number of Respondersparticipant) / (Number of participants in ITT1 population) x 100

• If MAS score of a given participant is missing at Week 6, then this participants will be regarded as a non-responder.

#### **Model Results Presentation**

• The difference in the responder rate (400 units – 200 units) and its associated 95% CI will be presented.

### **Subgroup Analyses (Rehabilitation)**

- Subgroup analyses will be performed by baseline rehabilitation in the Section 4.4.
- The difference (400 units 200 units) and its 95% CI will be presented.

# Subgroup Analyses (baseline MAS score)

- Subgroup analyses will be performed by baseline MAS score (3 or 4).
- The difference (400 units 200 units) and its 95% CI will be presented.

#### **Supportive Analyses**

- The difference in the responder rate will be estimated using Mantel-Haenszel method to consider a stratification factor, that is baseline MAS score (3 or 4).
- Mantel-Haenszel rate difference (400 units 200 units) and its 95% CI will be calculated.

## 6.2. Secondary Efficacy Analyses

### 6.2.1. Endpoint / Variables

Secondary Efficacy Endpoints are the following items:

• MAS scores in the elbow, finger, thumb and wrist flexors.

207660

- Change from baseline in MAS scores
- Responder rate of MAS in the elbow, finger, thumb and wrist flexors.
- DAS score (Main Assessment Parameter)
- Change from baseline in DAS score (Main Assessment Parameter)

## 6.2.2. Summary Measure

Summary Measures are as below.

- The differences in the responder rate of MAS scores
- The differences in the least square means of changes from baseline in MAS scores
- The differences in the least square means of changes from baseline in DAS scores

# 6.2.3. Population of Interest

The secondary efficacy analyses will be based on the Intent-To-Treat 1 population, unless otherwise specified.

The secondary efficacy analyses will be performed for only double blind phase. All efficacy analyses for open -label phase and other endpoints for double blind phase will be done as exploratory.

Unless specified otherwise, the data up to Week 12 of treatment will be summarized during the double-blind period. This is because this study allows to re-treat. In other words, after 12 weeks, only participants who have a smaller MAS score would remain and the difference of the change from baseline in MAS between 240 units and 400 units would be attenuated. Therefore, the data up to Week 12 of initial treatment will be analysed as secondary statistical analyses. This is the case for exploratory analyses for open label period (i.e. the data up to week 12 of re-treatment will be summarized). Listing will include the data after week 12 of treatment/re-treatment.

# 6.2.4. Strategy for Intercurrent (Post-Randomization) Events

Intercurrent event: early withdrawal from study.

Strategy for dichotomous data: the participant will be regarded as a non-responder.

Strategy for continuous data: the missing data will be removed from the analyses.

#### 6.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 6.2.1 will be summarised using descriptive statistics, graphically presented and listed.

207660

### 6.2.5.1. Statistical Methodology Specification

### **Secondary Efficacy Analysis**

## **Endpoint / Variables**

Change from baseline in MAS and DAS scores

#### **Model Specification**

- The endpoint will be analyzed using a mixed model for repeated measures (MMRM)
- Terms fitted in the MMRM will include the items below as fixed and categorical effects.
  - Treatment
  - Visit
  - Treatment-by-visit interaction
  - Baseline value
  - Baseline-by-visit interaction
- An unstructured variance structure will be used to model the within-participant errors, shared across treatments.
- The empirical sandwich estimator will be used to estimate the standard errors.

## **Model Checking & Diagnostics**

• If the model will not converge with unstructured variance, AR(1) variance structure can be used.

#### **Model Results Presentation**

Adjusted means (least square means) and corresponding standard errors of means will be
presented for each treatment by visit, together with estimated treatment differences (400 units

– 240 units) and the corresponding 95% CI.

#### **Data included in Model**

• The dataset including only data until week 12 after the first treatment will be used.

#### **Endpoint / Variables**

Responder Rate of MAS score

#### **Model Specification**

See primary endpoint section.

#### **Data Convention**

See primary endpoint section.

## **Supportive Statistical Analyses**

See supportive statistical analyses for primary efficacy analyses section.

## 6.3. Exploratory Efficacy Analyses

## 6.3.1. Modified Ashworth Scale (MAS)

These analyses will be based on ITT 2, 3 and 4 populations.

207660

Values and changes from baseline in MAS scores in finger, thumb, wrist, elbow, pronation of the forearm and shoulder flexors will be summarised using descriptive statistics, graphically presented and listed by visit and treatment cycle. Data up to Week 12 in each treatment cycle will be used for summary tables and Figures, whereas all data will be listed.

### 6.3.2. Numeric Rating Scale (NRS) for pain

These analyses will be based on ITT 1, 2, 3 and 4 populations.

Values and changes from baseline in NRS for pain will be summarised using descriptive statistics, graphically presented and listed by visit and treatment cycle.

# 6.3.3. Disability Assessment Scale (DAS)

These analyses will be based on ITT 1, 2, 3 and 4 populations.

Values and changes from baseline in all items of DAS will be summarised using descriptive statistics, graphically presented and listed by visit and treatment cycle.

# 6.3.4. Clinical Global Impression of Change (CGI) of functional disability

These analyses will be based on ITT 1, 2, 3 and 4 populations.

Values of the variables below will be summarised using descriptive statistics, graphically presented and listed by visit and treatment cycle.

CGI of functional disability by an investigator

CGI of functional disability by a patient

#### 6.3.5. Patient-Reported Benefit of Injection

These analyses will be based on ITT 1, 2, 3 and 4 populations.

The number and percentage of patient-reported benefit of injection will be presented and listed by visit and treatment cycle.

## 6.3.6. Time to Patient-Reported Onset of Spasticity Symptom Relief

These analyses will be based on ITT 1, 2, 3 and 4 populations.

Time to event data will be summarized using the descriptive statistics below and listed.

- The number of events and censored cases.
- Median survival time with the associated 95% CI.
- 25% and 75% survival time.

207660

Survival analyses will be conducted using a Kaplan-Meier method. To graphically compare the survival functions between 400 units and 240 units, the analysis will be conducted based on ITT 1 population whereas the analyses will be based on ITT 2, 3 and 4 populations to assess the survival time by treatment cycle. Participants who are withdrawn from this study before Visit 2 are censored at the withdrawal date. All other participants who do not experience the event and is not withdrawn from study are censored at the Visit 2.

Survival function estimates will be summarized (survival probabilities and the number of participants at risk per time to event, and median in survival time) based on Kaplan Meier method. Kaplan Meier plots will be presented.

#### 6.3.7. Time to Qualification for Retreatment

These analyses will be based on ITT 1, 2, 3 and 4 populations.

The number and percentage of event of interest will be presented by visit. Time to event data will be summarized using the descriptive statistics below and listed.

- The number of events and censored cases.
- Median survival time with the associated 95% CI.
- 25% and 75% survival time.

Survival analyses will be conducted using a Kaplan-Meier method. To graphically compare the survival functions between 400 units and 240 units, the analysis will be conducted based on ITT 1 population whereas the analyses will be based on ITT 2, 3 and 4 populations to assess the survival time by treatment cycle. Participants who are withdrawn from this study before the event are censored at the withdrawal date. All other participants who do not experience the event and is not withdrawn from study are censored at the Last Observed Visit at the interim analyses or the final analyses.

Survival function estimates will be summarized (survival probabilities and the number of participants at risk per time to event, and median in survival time) based on Kaplan Meier method. Kaplan Meier plots will be presented.

Note that the retreatment is not allowed within 83 days from the previous treatment. Therefore, this event will not occur before 83 days later after the treatment/re-treatment.

# 7. SAFETY ANALYSES

The safety analyses will be based on the Safety 1, 2, 3 and 4 populations, unless otherwise specified.

# 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 12: List of Data Displays.

207660

Adverse events that occurred in the overall study period, blinded period and open-label period will be summarized for each treatment group. The treatment group is based on dose actually given in blind period. For the blinded period, 2 patterns of analyses on adverse events will be performed, one is on adverse events that occurred between the initial dose and the first dose in the open-label period (or at the completion of study if no dose is given in the open-label period or at the study withdrawal), and another one is on adverse events that occurred within 84 days from the initial dose.

Overall study period (Treatment Emergent AEs)

# Blind phase

- 1. AEs occurred between the initial dose and the first dose in the open-label period (or at the completion of study if no dose is given in the open-label period or at the study withdrawal)
- 2. AEs occurred within 84 days from the initial dose

#### Open-label phase

- 1. AEs occurred during 2nd treatment cycle.
- 2. AEs occurred during 3rd treatment cycle.
- 3. AEs occurred during 4th treatment cycle.

The number and percentages of participants who experience at least one AE will be presented for each category of AE listed as below by treatment group.

- All Treatment Emergent AEs (by SOC and PT, by SOC, PT and Maximum Intensity)
- Common AEs ( $\geq 3\%$ ) (by overall frequency)
- Drug Related AEs (by SOC and PT, by SOC, PT and Maximum Intensity)
- Non-Fatal Serious AEs
- Drug Related Non-Fatal Serious AEs
- AEs Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study (by SOC and PT)
- Most Common Serious Drug Related AEs (by overall frequency)
- Most Common Non-Serious Drug Related AEs (by overall frequency)
- Common (>= 5%) Non-Serious AEs (by SOC and PT)
  - o Number of Participant and Occurrences will be presented.

"Common (>= 3%) AEs" is defined as the percentage of AEs is more than and equal to 3% in either treatment group.

In addition, the items below will be listed.

- All AEs
- Participant Numbers for Individual AEs
- Fatal Serious AEs
- Non-Fatal Serious AEs
- Reasons for Considering as a Serious AE

207660

- AEs Leading Withdrawal from Study/ Permanent Discontinuation of Study Treatment
- Relationship between AE SOC, PT and Verbatim Text.

# 7.2. Adverse Events of Special Interest Analyses

Adverse Events of Special Interest are defined as below.

- Convulsions and Seizures
- Respiratory Adverse Events
- Possible Distant Spread of Toxin

The number and percentage of AESI will be presented by treatment cycle and treatment group. The details of how to identify are described in the Appendix 13.

# 7.3. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 12: List of Data Displays.

These data at Screening Visit, in Blind Phase and at Final Visit will be summarized by visit. Data at all visits will be listed.

Values and change from baseline in Chemistry Laboratory tests and Hematology laboratory tests will be summarized by treatment group and visit.

Worst case results relative to normal range from baseline will be presented for Chemistry, Hematology and Urinalysis.

Shifts from baseline relative to normal range will be summarized by treatment group and visit for Chemistry and Hematology values.

Scatter plot of Chemistry and Hematology at Week 12 versus baseline in Blind Phase will be presented.

The outputs regarding liver events will not be presented unless at least one liver event is observed. See the details in the Appendix 12.

## 7.4. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 12: List of Data Displays.

These above data at Screening Visit, in Blind Phase and at Final Visit will be summarized by visit. Data at all visits will be listed.

207660

ECG findings (Normal, Abnormal – not clinically significant, Abnormal -clinically significant) will be summarized by visit.

Values and changes from baseline in ECG and vital sign data will be summarized by visit.

Values and changes from baseline in SpO2 will be summarized and listed by visit. Data at Screening visit, Visit 1 and 5 in Blind Phase and Final Visit will be summarized and those at all visits will be listed.

# 7.5. Exposure

## • Blind Phase

The number and percentage of participants treated will be presented and the dosage will be summarized by muscle region below, Joint and total. The dosage will be listed by muscle region, subtotal and total.

| Joint | Each muscle region |
|----------|--------------------------------|
| | Biceps brachii |
| Elbow | Brachialis |
| | Brachioradialis |
| Wrist | Flexor carpi radialis |
| Wiist | Flexor carpi ulnaris |
| Finance | Flexor digitorum profundus |
| Finger | Flexor digitorum superficialis |
| Thumb | Flexor pollicis longus |
| ITIUIIID | Adductor pollicis |

#### Open Label Phase

The number and percentage of participants treated will be presented and the dosage will be summarized by treatment phase (2nd, 3rd and 4th treatment), muscle region below, Joint and total. The dosage will be listed by treatment phase and muscle region, Joint and total.

# 207660

| Joint | Each muscle region |
|-----------|--------------------------------|
| | Biceps brachii |
| Elbow | Brachialis |
| | Brachioradialis |
| Wrist | Flexor carpi radialis |
| Wilst | Flexor carpi ulnaris |
| | Flexor digitorum profundus |
| Finger | Flexor digitorum superficialis |
| | Lumbricales interossei |
| | Flexor pollicis longus |
| Thumb | Adductor pollicis |
| | Opponens |
| Forcermo | Pronator teres |
| Forearms | Pronator quadratus |
| | Teres major |
| Shoulder | Latissimus dorsi |
| Silouldei | Pectoralis major |
| | Subscapularis |

207660

# 8. REFERENCES

GlaxoSmithKline Document Number 2017N315029\_02 Study ID 207660. A phase III study (a placebo controlled, randomized, double-blind comparative study and an openlabel, uncontrolled study) to evaluate the efficacy and safety of GSK1358820 in patients with post-stroke upper limb spasticity. Report Date 06-Oct-2017.

Study Reference Manual, Study ID 207660. A phase III study (a placebo controlled, randomized, double-blind comparative study and an open-label, uncontrolled study) to evaluate the efficacy and safety of GSK1358820 in patients with post-stroke upper limb spasticity. Effective Date 29-Jun-2017

207660

# 9. APPENDICES

# 9.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

Per Protocol Population is not defined in this study.

207660

# 9.2. Appendix 2: Schedule of Activities

# 9.2.1. Protocol Defined Schedule of Events

| | Screening <sup>a</sup> | 1)<br>the pa | If<br>rticipa | a par | ticipa<br>Ill mo | Blind phase<br>nt meets the elig<br>we forward to the | ibility at V5/ QRV, e open-label phase | If a p | articipa | int meet<br>move f | s the eli | en-label phase<br>gibility at V5/QR<br>to the next treatme | V, the participant will ent phase | Completion visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Part 1 | | | | Eligibility<br>evaluation <sup>b</sup> | Part 2/Part 3/ Part 4 | | | | | Eligibility<br>evaluation b | Visit | |
| Visit | SV | V1<br>(Day 1) | V2 | V3 | V4 | V5 °<br>(Eligibility<br>evaluation) | QRV | V1 | V2 | V3 | V4 | V5 <sup>a</sup><br>(Eligibility<br>evaluation) | QRV | Final<br>Visit |
| Time from initial injection (Day 1) (Weeks) | - | 0 | 2 | 4 | 6 | 12 | Allowable Week 16 to 36 <sup>e</sup> | | _ | _ | | _ | Allowable Week 24 to 36 e | 48/<br>Withdrawal |
| Time from injection day in each treatment phase (Weeks) | | 0 | 2 | 4 | 6 | 12 | 16/ 20/ 24/ 28/ 32/<br>36 | 0 | 2 | 4 | 6 | 12 | 16/ 20/ 24 | - |
| Acceptable visit windows (days) | | _ | ±4 | ±4 | ±4 | +4 <sup>r</sup> | ±14 <sup>g</sup> | (+4) <sup>v</sup> | ±4 | ±4 | ±4 | +4 1 | ±14 <sup>g</sup> | ±4 |
| Written informed consent | X n | | | | | | | | | | | | | |
| Randomization | | X 1 | | | | | | | | | | | | |
| Injections | | X | | | | | | X | | | | | | |
| Evaluation of eligibility | | | | | | X | X | | | | | X | X | |
| Inclusion/exclusion criteria J | X | X 1 | | | | | | | | | | | | |
| Participant demography | X | | | | | | | | | | | | | |
| MAS <sup>K</sup> | X | X 1 | X | X | X | X | X | X 1,t | X | X | X | X | X | X |
| NRS <sup>1</sup> | | X 1 | X | X | X | X | | $X^{i,t}$ | X | X | X | X | | (X) <sup>r</sup> |
| DAS | | X 1 | X | X | X | X | | X 1,t | X | X | X | X | | (X) <sup>r</sup> |
| CGI by a investigator | | | X | X | X | X | | | X | X | X | X | | (X) <sup>r</sup> |
| CGI by a patient | | | X | X | X | X | | | X | X | X | X | | (X) <sup>r</sup> |
| Time to patient-reported onset of spasticity symptom relief | | | X | | | | | | X | | | | | |
| Patient-reported benefit of injection | | | | X | X | X | | | | X | X | X | | (X) <sup>r</sup> |
| Physical examination (complete version) | X | | | | | | | | | | | | | |
| Physical examination (simplified version) | | X <sup>1</sup> | | | | X | | X 1,t | | | | X | | X |
| Medical history | X | X 1 | | | | | | | | | | | | |
| Vital signs m | X | X 1 | | | | X | | X 1,t | | | | X | | X |
| Height | X | | | | | | | | | | | | | |
| Body weight | X | | | | | X <sup>u</sup> | X <sup>u</sup> | | | | | X <sup>u</sup> | X <sup>u</sup> | |
| Pulmonary function test | X | X | | | | X | X <sup>u</sup> | | | | | X | X u | X |
| Electrocardiogram | X | | | | | X <sup>u</sup> | X <sup>u</sup> | | | | | X <sup>u</sup> | X <sup>u</sup> | |
| Pregnancy test <sup>n</sup> | X | X 1 | | | | X <sup>u</sup> | X u | | | 1 | | X <sup>s, u</sup> | X <sup>u</sup> | X |

207660

| | Screening <sup>a</sup> | 1)<br>the pa | Blind phase 1) If a participant meets the eligibility at V5/ QRV, the participant will move forward to the open-label phase | | | | | Open-label phase If a participant meets the eligibility at V5/QRV, the participant will move forward to the next treatment phase | | | | | | Completion visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Part 1 | | | art 1 | | Eligibility<br>evaluation <sup>b</sup> | Part 2/Part 3/ Part 4 | | | | Part 4 | Eligibility<br>evaluation <sup>b</sup> | |
| Visit | sv | (Day 1) | V2 | V3 | V4 | V5 °<br>(Eligibility<br>evaluation) | QRV | V1 | V2 | V3 | V4 | V5 <sup>a</sup> (Eligibility evaluation) | QRV | Final<br>Visit |
| Laboratory test ° | X | | | | | X | | | | | | X | | X |
| Adverse events p | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant medications/therapies | X | X¹ | X | X | X | X | X | X | X | X | X | X | X | X |
| Testing for neutralising antibodies <sup>q</sup> | X | | | | | X | | | | | | | | X |

- a. Test items for screening must be performed from 4 weeks to 1 weeks before Day 1 visit (±3 days).
- b. Eligibility evaluation (Qualification for Retreatment Visit: QRV) will be performed at V5 as a starting point if a participant does not meet the criteria only. The evaluation is performed at a 4-week interval, V5 as a starting point, The QRV when a participant meets the criteria will be a same day as the injection in the next treatment period.
- c. If a participant is evaluated to meet the eligibility for the injection in the blind phase at V5, the participant will move forward to Part 2 in the open-label phase (Namely, V5 in Part 1 and V1 in Part 2 is a same day). If the participant does not meet the eligibility, QRV will be performed 4 weeks later, at V5 as s starting point.
- d. If a participant is evaluated to meet the eligibility at V5 in the open-label phase, the participant will move forward to the next treatment phase (V5 and V1 in the next treatment phase is a same day). If the participant does not meet the eligibility, QRV is performed 4 weeks later, V5 as a starting point. If V5 in each treatment phase is at Week 48 after initial injection, V5 will be considered to be completion visit (FV). However, for the testing items, pre-scheduled tests at V5 and neutralizing antibody tests will be performed. If V5 in Parts 2 and 3 is performed at Week 36 or later, after completion of V5, completion visit will be performed at Week 48.
- e. QRV is allowable to perform from initial injection to Week 36. Eligibility evaluation (QRV) will not be performed after Week 36.
- f. V5 must be performed at least 84 days after V1.
- g. The acceptable visit windows will be -14 to +4 days if QRV is performed at Week 36.
- h. Must be performed earlier than any other procedures
- i. Must be performed before injection of the product
- j. For inclusion/exclusion criteria, the items to be observed are different between screening phase and Day 1. For details, refer to Protocol Section 6.1 and Section 6.2.

207660

- k. For MAS evaluation, the items to be evaluated differ depending on the treatment phase. For details, refer to Protocol Section 9.1.1.1.
- 1. MAS evaluation will be followed by NRS evaluation. For NRS evaluation, items to be evaluated differ. For details, refer to Protocol Section 9.1.1.2.
- m. Body temperature, heart rate, and blood pressure will be measured as vital signs.
- n. Women of childbearing potential will be only performed. Serum hCG pregnancy test must be performed at screening, and urine hCG pregnancy test after randomization. The tests can be performed beyond the protocol specifications if an investigator considers to be necessary.
- o. For laboratory test items, refer to Protocol Section 12.2. Attachment 2. Fasting is not required for blood collection.
- p. Adverse events and serious adverse events collection period will be from the initial injection day (Day 1) to completion visit (FV).
- q. Neutralizing antibody testing is performed 3 times in each participant. The first test will be performed in screening phase, the second is at V5 in the blind phase, and the third is at completion visit.
- r. A participant who withdraws the study before 12 weeks after last injection will be performed.
- s. Perform if V5 in each treatment phase is at Week 48 after initial injection
- t. Not necessary to perform doubly as V1 assessment if the same assessment is performed at V5 or QRV. If V1 assessment or retreatment cannot be performed on the same day as V5 or QRV, MAS assessment should be performed again on the day of visit for the V1 assessment.
- u. Evaluation of retreatment is performed only when the dosing conditions (1 to 5) of retreatment evaluation are met. If V1 assessment or retreatment cannot be performed on the same day as V5 or QRV, body weight, pulmonary function test, electrocardiogram, and pregnancy test should not be performed again on the day of visit for V1 assessment.
- v. V1 assessment in Part 2 or subsequent parts should be performed as a rule on the same day as V5 or QRS (when eligibility was confirmed) of the previous part. If this is not possible, the V1 assessment may be performed on another day but within the acceptable visit window.

207660

# 9.3. Appendix 3: Assessment Windows

This study does not define Assessment Windows.

207660

# 9.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

## 9.4.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is prior to the date of first treatment |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 9.4.2. Study Phases for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | First Study Treatment Date ≤ AE Start Date ≤ Final Visit Date/Early Withdrawal Date |
| Blind phase (until second dose) | <ul> <li>First Study Treatment Date ≤ AE Start Date ≤ Second Study Treatment Date AND AE Start Time &lt; Second Study Treatment Time IF AE Start Time is collected</li> <li>First Study Treatment Date ≤ AE Start Date &lt; Second Study Treatment Date IF AE Start Time is not collect.</li> </ul> |
| Blind phase (within 84 days) | First Study Treatment Date ≤ AE Start Date ≤ First Study Treatment Date + 84 days AND AE Start Time < Second Study Treatment Time |
| Open-Label<br>Phase (2nd<br>Treatment) | <ul> <li>Second Study Treatment Date ≤ AE Start Date ≤ Third Study Treatment Date AND Second Study Treatment Time ≤ AE Start Time &lt; Third Study Treatment Time IF AE Start Time is collected</li> <li>Second Study Treatment Date ≤ AE Start Date &lt; Third Study Treatment Date IF AE Start Time is not collected</li> </ul> |
| Open-Label<br>Phase (3rd<br>Treatment) | <ul> <li>Third Study Treatment Date ≤ AE Start Date ≤ Fourth Study Treatment Date AND Third Study Time ≤ AE Start Time &lt; Fourth Study Treatment Time IF AE Start Time is collected</li> <li>Third Study Treatment Date ≤ AE Start Date &lt; Fourth Study Treatment Date IF AE Start Time is not collected</li> </ul> |
| Open-Label<br>Phase (4th<br>Treatment) | <ul> <li>Fourth Study Treatment Date ≤ AE Start Date ≤ Final Visit Date AND Fourth Study Time ≤ AE Start Time IF AE Start Time is collected</li> <li>Fourth Study Treatment Date ≤ AE Start Date ≤ Final Visit Date IF AE Start Time is not collected</li> </ul> |
| Drug related | If relationship to Study treatment(GSK1358820/Placebo) is marked 'YES' on CRF OR value is missing. |

## 9.4.2.1. Definition of Adverse Events of Special Interest

AEs of Special Interest are defined in the Appendix 13. If a Preferred Term of AE is included in the list of PTs of the specific AESI, that AE will be considered as AESI. See the details in the Appendix 13.

207660

# 9.5. Appendix 5: Data Display Standards & Handling Conventions

#### 9.5.1. Reporting Process

| Software | |
|---|---|
| The currently supply | The currently supported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server | : US1SALX00259.corpnet2.com |
| HARP Compound | : arenv\arprod\gsk1358820\mid207660 |
| Analysis Datasets | |
| Analysis datasets | Analysis datasets will be created according to Legacy GSK A&R dataset standards. |
| Generation of RTF Files | |
| RTF files will not be generated. | |

# 9.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:
  - https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include participant level listings in the main body of the GSK Clinical Study Report. All
  participant level listings should be located in the modular appendices as ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.

207660

| Unscheduled Visits | Unscheduled Visits |
|---|---|
| Unscheduled visits | Unscheduled visits will not be included in summary tables and/or figures. |
| All unscheduled vis | sits will be included in listings. |
| <b>Descriptive Summary</b> | Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Time to event data | <ul> <li>The number of events and censored case.</li> <li>25<sup>th</sup> and 75<sup>th</sup> percentiles survival time.</li> <li>Median survival time with the associated 95% CIs.</li> <li>95%CIs will be calculated based on Brookmeyer and Crowley method using log-log function as a g-transformation. (This method can be performed using Proc</li> </ul> |
| LIFETEST with no special statement or option (SAS 9.4)) Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

207660

# 9.6. Appendix 6: Derived and Transformed Data

#### 9.6.1. **General**

#### **Study Day**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
- Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

## 9.6.2. Study Population

## Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follow:
  - Any participant with a missing date and month will have this imputed as '30<sup>th</sup> June'.
- Birth date will be presented in listings as 'YYYY'.
- Age will be calculated based on year of the Screening visit as an Age reference date.

#### Age Group

- The following category will be used for Summary of Demography.
  - $\circ \quad \text{Age} \leq 18 \text{ (years)}$
  - o 19 < Age < 64
  - $\circ$  65  $\leq$  Age

#### Age Category

- The following category will be used for Summary of Age Ranges.
  - Age < 17 (years)</li>
  - $\circ$  18  $\leq$  Age  $\leq$  64
  - $\circ$  65  $\leq$  Age  $\leq$  84
  - o 85 ≤ Age

# **Extent of Exposure**

- The total of dosage per treatment cycle will be calculated based on the formula:
  - Total of Dosage per treatment cycle = Sum of (Dosage in each Muscle Region)
- The subtotal of dosage in each joint per treatment cycle will be calculated based on the formula:
   Subtotal of Dosage in the joint per treatment cycle = Sum of (Dosage in each Muscle Region of the Joint)
- Example

Subtotal of Dosage in Elbow = Sum of (Dosage in Biceps brachii, Brachalis and Brachioradialis)

207660

## 9.6.3. Efficacy

#### **Time to Event Data**

#### Time to Qualification for Retreatment

• This time to event data will be derived based on the following formula:

# Time to Event (Days) = Date When a Participant Meets the Criteria for Retreatment – Study Treatment Start Date (Days)

• If a participant is withdrawn from this study, the participant will be regarded as censoring and censored date will be a withdrawal date.

## Time to Patient Reported Onset of Spasticity Symptom Relief

• This time to event data will be derived based on the following formula:

# Time to Event (Days) = Onset Date of the Spasticity Symptom Relief – Study Treatment Start Date (Days)

If a participant is withdrawn from this study, the participant will be regarded as censoring and censored date will be a withdrawal date.

207660

# 9.7. Appendix 7: Reporting Standards for Missing Data

# 9.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Participant study completion (i.e. as specified in the protocol) was defined as those who completed all the study procedures, including a completion visit. |
| | Withdrawn participants were not replaced in the study. |
| | <ul> <li>All available data from participants who were withdrawn from the study will be listed<br/>and all available planned data will be included in summary tables and figures, unless<br/>otherwise specified.</li> </ul> |
| | Withdrawal visits will be slotted as per Appendix 3: Assessment Windows or will be summarised as withdrawal visits. |

# 9.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in participant listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Responder of MAS | If MAS score is missing at the corresponding visit, the participant will be regarded as those who are a non-responder (i.e. non-responder imputation). |

# 9.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in participant listing displays. |
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
207660

# 9.8. Appendix 8: Values of Potential Clinical Importance

This is not applicable to this study.

207660

# 9.9. Appendix 9: Population Pharmacokinetic (PopPK) Analyses

This is not applicable to this study.

207660

# 9.10. Appendix 10: Pharmacokinetic / Pharmacodynamic Analyses

This is not applicable to this study.

207660

# 9.11. Appendix 11: Abbreviations & Trade Marks

## 9.11.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |

207660

| Abbreviation | Description |
|--------------|------------------------------|
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

## 9.11.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies | |
|---------------------------------------------------------|---|
| NONE | 1 |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |

207660

## 9.12. Appendix 12: List of Data Displays

## 9.12.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|--------------|-------------|
| Study Population | 1.1 to 1.18 | |
| Efficacy | 2.1 to 2.49 | 2.1 to 2.56 |
| Safety | 3.1 to 3.132 | 3.1 to 3.2 |
| Section | Listings | |
| ICH Listings | 1 to 61 | |

#### 9.12.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 9.12.3. Deliverables

| Delivery | Description |
|----------|------------------------------------------------|
| IA SAC | Interim Analysis Statistical Analysis Complete |
| SAC | Final Statistical Analysis Complete |

207660

## 9.12.4. Study Population Tables

## 9.12.4.1. Interim Analyses

| Study | Population Tabl | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Partici | pant Disposition | n | | | |
| 1.1. | ITT1 | ES1 | Summary of Participant Disposition for the Participant Conclusion Record (Week 24) | ICH E3, FDAAA, EudraCT Participant disposition at Week 24. | IA SAC |
| 1.2. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | IA SAC |
| 1.3. | Enrolled | NS1 | Summary of Number of Participant by Site ID | EudraCT/Clinical Operations | IA SAC |
| Protoc | ol Deviation | | | | |
| 1.4. | ITT1 | DV1 | Summary of Important Protocol Deviations | ICH E3 | IA SAC |
| Popula | tion Analysed | | | | |
| 1.5. | Screened | SP1 | Summary of Study Populations | IDSL | IA SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.6. | ITT1 | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT<br>Include total arm (240 U + 400 U) | IA SAC |
| 1.7. | Enrolled | DM11 | Summary of Age Ranges | EudraCT | IA SAC |
| 1.8. | Enrolled | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | IA SAC |
| 1.9. | ITT1 | POP_T1 | Summary of Baseline Efficacy Parameters | <ul> <li>MAS scores in finger, thumb, wrist, elbow, pronation of forearm and shoulder flexors</li> <li>Numeric Rating Scale for pain</li> <li>Disability Assessment Scale</li> <li>Include total arm (240 U + 400 U)</li> </ul> | IA SAC |

207660

| Study F | Study Population Tables | | | |
|---|---|---|---|---|
| No. | No. Population IDSL / Example Shell Title Programming Notes Deliverable | | | |
| Prior ar | Prior and Concomitant Medications | | | |
| 1.10. | ITT1 | CM1 | Summary of Prior Medications | IA SAC |
| 1.11. | 1.11. ITT1 CM1 Summary of Concomitant Medications ICH E3 IA SAC | | | |
| 1.12. | ITT1 | POP_T2 | Summary of Rehabilitation | IA SAC |

## 9.12.4.2. Final Analyses

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Particip | ant Disposition | n | | | |
| 1.13. | ITT1 | ES1 | Summary of Participant Disposition for the Participant Conclusion Record | ICH E3, FDAAA, EudraCT | SAC |
| Protoco | ol Deviation | | | | |
| 1.14. | ITT1 | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC |
| Popula | tion Analysed | | | | |
| 1.15. | Screened | SP1 | Summary of Study Populations | IDSL | SAC |
| Prior ar | nd Concomitan | t Medications | | | |
| 1.16. | ITT1 | CM1 | Summary of Prior Medications | | SAC |
| 1.17. | ITT1 | CM1 | Summary of Concomitant Medications | ICH E3 | SAC |
| 1.18. | ITT1 | POP_T2 | Summary of Rehabilitation | | SAC |

207660

## 9.12.5. Efficacy Tables

## 9.12.5.1. Interim Analyses

| Efficacy | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| MAS | | | | | |
| 2.1. | ITT1 | EFF_T1 | Summary of MAS score in Blind Phase | <ul><li>Values and change from baseline</li><li>Summarize data up to Visit 5</li></ul> | IA SAC |
| 2.2. | ITT1 | EFF_T2 | Summary of the Results of Mixed Models for Repeated<br>Measures of Change from Baseline in MAS scores in Blind<br>Phase | Analyse data up to Visit 5 | IA SAC |
| 2.3. | ITT1 | EFF_T3 | Summary of Responder rate of MAS score at Week 6 in Blind Phase | Including subgroup analyses | IA SAC |
| 2.4. | ITT1 | EFF_T4 | Summary of Responder rate of MAS score in Blind Phase | Summarize data up to Visit 5<br>Include Mantel Haenszel estimators | IA SAC |
| 2.5. | ITT2 | EFF_T1 | Summary of MAS score in Open Label Phase (2nd Treatment) | <ul> <li>Values and change from baseline</li> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| 2.6. | ITT2 | EFF_T5 | Summary of Responder rate of MAS score in Open Label Phase (2nd Treatment) | <ul> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |

| Efficacy | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| DAS | | | | | |
| 2.7. | ITT1 | EFF_T1 | Summary of Main Assessment Parameter and All Items of DAS in Blind Phase | <ul><li>Values and change from baseline</li><li>Summarize data up to Visit 5</li></ul> | IA SAC |
| 2.8. | ITT1 | EFF_T2 | Summary of the Results of Mixed Models for Repeated Measures of Main Assessment Parameter of DAS in Blind Phase | Analyse data up to Visit 5 | IA SAC |
| 2.9. | ITT2 | EFF_T1 | Summary of Main Assessment Parameter and All Items of DAS in Open Label Phase (2nd Treatment) | <ul> <li>Values and change from baseline</li> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| NRS for | pain | | | | |
| 2.10. | ITT1 | EFF_T1 | Summary of NRS for pain in Blind Phase | <ul><li>Values and change from baseline</li><li>Summarize data up to Visit 5</li></ul> | IA SAC |
| 2.11. | ITT2 | EFF_T1 | Summary of NRS for pain in Open Label Phase (2nd Treatment) | <ul> <li>Values and change from baseline</li> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |

| Efficacy: | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| CGI of fu | ınctional disal | bility | | | |
| 2.12. | ITT1 | EFF_T1 | Summary of CGI of functional disability by an investigator in Blind Phase | <ul><li>Values and change from baseline</li><li>Summarize data up to Visit 5</li></ul> | IA SAC |
| 2.13. | ITT2 | EFF_T1 | Summary of CGI of functional disability by an investigator in Open Label Phase (2nd Treatment) | <ul> <li>Values and change from baseline</li> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| 2.14. | ITT1 | EFF_T1 | Summary of CGI of functional disability by a patient in Blind Phase | Values and change from baseline Summarize data up to Visit 5 | IA SAC |
| 2.15. | ITT2 | EFF_T1 | Summary of CGI of functional disability by a patient in Open Label Phase (2nd Treatment) | <ul> <li>Values and change from baseline</li> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| Patient-F | Reported Bene | efit of Injection | | · | |
| 2.16. | ITT1 | EFF_T5 | Summary of Patient-Reported Benefit of Injection in Blind Phase | Values and change from baseline Summarize data up to Visit 5 | IA SAC |

| Efficacy | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.17. | ITT2 | EFF_T5 | Summary of Patient-Reported Benefit of Injection in Open Label Phase (2nd Treatment) | <ul> <li>Values and change from baseline</li> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| Time to | Patient-Repor | ted Onset of Spas | ticity Symptom Relief | | |
| 2.18. | ITT1 | EFF_T6 | Summary of Time to Patient-Reported Onset of Spasticity Symptom Relief | | IA SAC |
| 2.19. | ITT1 | EFF_T7 | Summary of Survival Analyses Results of Time to Patient-<br>Reported Onset of Spasticity Symptom Relief in Blind Phase | Survival function estimates will be summarized | IA SAC |
| 2.20. | ITT2 | EFF_T7 | Summary of Survival Analyses Results of Time to Patient-<br>Reported Onset of Spasticity Symptom Relief in Open Label<br>Phase (2nd Treatment) | Survival function estimates will be summarized Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| Time to | Qualification f | or Retreatment | | | |
| 2.21. | ITT1 | EFF_T8 | Summary of Events in Which a Participant Meets the Criteria for Retreatment | | IA SAC |
| 2.22. | ITT1 | EFF_T6 | Summary of Time to Qualification for Retreatment | | IA SAC |
| 2.23. | ITT1 | EFF_T7 | Summary of Survival Analyses Results of Time to Qualification for Retreatment in Blind Phase | Survival function estimates will be summarized Two treatment arms (240 and 400U) | IA SAC |

207660

| Efficacy: | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.24. | ITT2 | EFF_T7 | Summary of Survival Analyses Results of Time to Qualification for Retreatment in Open Label Phase (2nd Treatment) | <ul> <li>Survival function estimates will<br/>be summarized</li> <li>Three treatment arms (240,<br/>400 and 240 + 400U)</li> </ul> | IA SAC |

## 9.12.5.2. Final Analyses

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| MAS | | | | | |
| 2.25. | ITT3 | EFF_T1 | Summary of MAS score in Open Label Phase (3rd Treatment) | Values and change from | SAC |
| 2.26. | ITT4 | EFF_T1 | Summary of MAS score in Open Label Phase (4th Treatment) | <ul> <li>baseline</li> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | SAC |
| 2.27. | ITT3 | EFF_T5 | Summary of Responder rate of MAS score in Open Label Phase (3rd Treatment) | <ul> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | SAC |
| 2.28. | ITT4 | EFF_T5 | Summary of Responder rate of Mas Score in Open Label Phase (4th Treatment) | | SAC |

| Efficacy | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| DAS | • | | | | |
| 2.29. | ITT3 | EFF_T1 | Summary of Main Assessment Parameter and All Items of DAS in Open Label Phase (3rd Treatment) | Values and change from baseline | SAC |
| 2.30. | ITT4 | EFF_T1 | Summary of Main Assessment Parameter and All Items of DAS in Open Label Phase (4th Treatment) | <ul> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | SAC |
| NRS for | pain | | | | |
| 2.31. | ITT3 | EFF_T1 | Summary of NRS for pain in Open Label Phase (3rd Treatment) | Values and change from | SAC |
| 2.32. | ITT4 | EFF_T1 | Summary of NRS for pain in Open Label Phase (4th Treatment) | <ul> <li>baseline</li> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | SAC |
| CGI of fu | unctional disa | bility | | | |
| 2.33. | ITT3 | EFF_T1 | Summary of CGI of functional disability by an investigator in Open Label Phase (3rd Treatment) | Values and change from baseline | SAC |
| 2.34. | ITT4 | EFF_T1 | Summary of CGI of functional disability by an investigator in Open Label Phase (4th Treatment) | <ul> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | SAC |
| 2.35. | ITT3 | EFF_T1 | Summary of CGI of functional disability by a patient in Open Label Phase (3rd Treatment) | Values and change from baseline | SAC |
| 2.36. | ITT4 | EFF_T1 | Summary of CGI of functional disability by a patient in Open Label Phase (4th Treatment) | <ul> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | SAC |

| Efficacy | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Patient-l | Reported Bene | efit of Injection | | | |
| 2.37. | ITT3 | EFF_T5 | Summary of Patient-Reported Benefit of Injection in Open Label Phase (3rd Treatment) | Values and change from baseline | SAC |
| 2.38. | ITT4 | EFF_T5 | Summary of Patient-Reported Benefit of Injection in Open Label Phase (4th Treatment) | <ul> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | SAC |
| Time to | Patient-Repor | ted Onset of Spas | ticity Symptom Relief | | |
| 2.39. | ITT1 | EFF_T6 | Summary of Time to Patient-Reported Onset of Spasticity<br>Symptom Relief | | SAC |
| 2.40. | ITT1 | EFF_T7 | Summary of Survival Analyses Results of Time to Patient-<br>Reported Onset of Spasticity Symptom Relief in Blind Phase | Survival function estimates will<br>be summarized | SAC |
| 2.41. | ITT2 | EFF_T7 | Summary of Survival Analyses Results of Time to Patient-<br>Reported Onset of Spasticity Symptom Relief in Open Label<br>Phase (2nd Treatment) | | SAC |
| 2.42. | ITT3 | EFF_T7 | Summary of Survival Analyses Results of Time to Patient-<br>Reported Onset of Spasticity Symptom Relief in Open Label<br>Phase (3rd Treatment) | Survival function estimates will be summarized Three treatment arms (240, 400 and 240 at 400 l) | SAC |
| 2.43. | ITT4 | EFF_T7 | Summary of Survival Analyses Results of Time to Patient-<br>Reported Onset of Spasticity Symptom Relief in Open Label<br>Phase (4th Treatment) | - 400 and 240 + 400U) - | SAC |
| Time to | Qualification f | or Retreatment | | | |
| 2.44. | ITT1 | EFF_T8 | Summary of Events in Which a Participant Meets the Criteria for Retreatment | | SAC |
| 2.45. | ITT1 | EFF_T6 | Summary of Time to Qualification for Retreatment | | SAC |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.46. | ITT1 | EFF_T7 | Summary of Survival Analyses Results of Time to Qualification for Retreatment in Blind Phase | Survival function estimates will be summarized Two treatment arms (240 and 400U) | SAC |
| 2.47. | ITT2 | EFF_T7 | Summary of Survival Analyses Results of Time to Qualification for Retreatment in Open Label Phase (2nd Treatment) | Survival function estimates will | SAC |
| 2.48. | ITT3 | EFF_T7 | Summary of Survival Analyses Results of Time to Qualification for Retreatment in Open Label Phase (3rd Treatment) | be summarized Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 2.49. | ITT4 | EFF_T7 | Summary of Survival Analyses Results of Time to Qualification for Retreatment in Open Label Phase (4th Treatment) | | SAC |

207660

## 9.12.6. Efficacy Figures

## 9.12.6.1. Interim Analyses

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| MAS | | | | | |
| 2.50. | ITT1 | EFF_F1 | Plot of Mean (95%CI) MAS score Profiles in Blind Phase | <ul> <li>Plot data up to Visit 5</li> <li>Two treatment arms (240 and 400U)</li> </ul> | IA SAC |
| 2.51. | ITT2 | EFF_F1 | Plot of Mean (95%CI) MAS score Profiles in Open Label Phase (2nd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| 2.52. | ITT1 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in MAS score<br>Profiles in Blind Phase | <ul><li>Plot data up to Visit 5</li><li>Two treatment arms (240 and 400U)</li></ul> | IA SAC |
| 2.53. | ITT2 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in MAS score<br>Profiles in Open Label Phase (2nd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| 2.54. | ITT1 | EFF_F2 | Plot of Responder rate of MAS score by Visit in Blind Phase | <ul><li>Plot data up to Visit 5</li><li>Two treatment arms (240 and 400U)</li></ul> | IA SAC |
| 2.55. | ITT2 | EFF_F2 | Plot of Responder rate of MAS score by Visit in Open Label<br>Phase (2nd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| DAS | | | | | |
| 2.56. | ITT1 | EFF_F1 | Plot of Mean (95%CI) DAS score (Main Assessment Parameter)<br>Profiles in Blind Phase | <ul><li>Plot data up to Visit 5</li><li>Two treatment arms (240 and 400U)</li></ul> | IA SAC |
| 2.57. | ITT2 | EFF_F1 | Plot of Mean (95%CI) DAS score (Main Assessment Parameter)<br>Profiles in Open Label Phase (2nd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| 2.58. | ITT1 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in DAS score (Main Assessment Parameter) Profiles in Blind Phase | <ul><li>Plot data up to Visit 5</li><li>Two treatment arms (240 and 400U)</li></ul> | IA SAC |
| 2.59. | ITT2 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in DAS score (Main Assessment Parameter) Profiles in Open Label Phase (2nd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| 2.60. | ITT1 | EFF_F1 | Plot of Mean (95%CI) DAS score Profiles in Blind Phase | <ul> <li>Plot data up to Visit 5</li> <li>Create plots by component of<br/>DAS score</li> <li>Two treatment arms (240 and<br/>400U)</li> </ul> | IA SAC |
| 2.61. | ITT2 | EFF_F1 | Plot of Mean (95%CI) DAS score Profiles in Open Label Phase (2nd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Create plots by component of DAS score</li> <li>Three treatment arms (240 and 400U)</li> </ul> | IA SAC |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.62. | ITT1 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in DAS score<br>Profiles in Blind Phase | <ul> <li>Plot data up to Visit 5</li> <li>Create plots by component of DAS score</li> <li>Two treatment arms (240 and 400U)</li> </ul> | IA SAC |
| 2.63. | ITT2 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in DAS score<br>Profiles in Open Label Phase (2nd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Create plots by component of<br/>DAS score</li> <li>Three treatment arms (240 and<br/>400U)</li> </ul> | IA SAC |
| Numeri | c Rating Scale | for pain | | | |
| 2.64. | ITT1 | EFF_F1 | Plot of Mean (95%CI) NRS for pain Profiles in Blind Phase | <ul> <li>Plot data up to Visit 5</li> <li>Two treatment arms (240 U and 400U)</li> </ul> | IA SAC |
| 2.65. | ITT2 | EFF_F1 | Plot of Mean (95%CI) NRS for pain Profiles in Open Label<br>Phase (2nd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| 2.66. | ITT1 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in NRS for pain Profiles in Blind Phase | <ul> <li>Plot data up to Visit 5</li> <li>Two treatment arms (240 U and 400U)</li> </ul> | IA SAC |
| 2.67. | ITT2 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in NRS for pain<br>Profiles in Open Label Phase (2nd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Clinica | I Global Impres | sion of Change o | f functional disability | | |
| 2.68. | ITT1 | EFF_F1 | Plot of Mean (95%CI) CGI of functional disability Profiles in Blind Phase | <ul><li>Plot data up to Visit 5</li><li>Two treatment arms (240 and 400 U)</li></ul> | IA SAC |
| 2.69. | ITT2 | EFF_F1 | Plot of Mean (95%CI) CGI of functional disability Profiles in Open Label Phase (2nd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400 U)</li> </ul> | IA SAC |
| Time to | Patient-Repor | ted Onset of Spas | ticity Symptom Relief | | |
| 2.70. | ITT1 | EFF_F3 | Kaplan Meier Plot of Time to Patient-Reported Onset of Spasticity Symptom Relief in Blind Phase | Two treatment arm (240 U and 400U) | IA SAC |
| 2.71. | ITT2 | EFF_F3 | Kaplan Meier Plot of Time to Patient-Reported Onset of Spasticity Symptom Relief in Open Label Phase (2nd Treatment) | | IA SAC |
| 2.72. | ITT3 | EFF_F3 | Kaplan Meier Plot of Time to Patient-Reported Onset of Spasticity Symptom Relief in Open Label Phase (3rd Treatment) | Three treatment arms (240, 400, 240 + 400U) | IA SAC |
| 2.73. | ITT4 | EFF_F3 | Kaplan Meier Plot of Time to Patient-Reported Onset of Spasticity Symptom Relief in Open Label Phase (4th Treatment) | | IA SAC |
| Time to | Qualification f | or Retreatment | | | |
| 2.74. | ITT1 | EFF_F3 | Kaplan Meier Plot of Survival Function Estimates of Time to Qualification for Retreatment in Blind Phase | Two treatment arm (240 U, 400U) | IA SAC |

207660

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.75. | ITT2 | EFF_F3 | Kaplan Meier Plot of Survival Function Estimates of Time to Qualification for Retreatment in Open Label Phase (2nd Treatment) | | IA SAC |
| 2.76. | ITT3 | EFF_F3 | Kaplan Meier Plot of Survival Function Estimates of Time to Qualification for Retreatment in Open Label Phase (3rd Treatment) | Three treatment arm (240, 400, 240 + 400U) | IA SAC |
| 2.77. | ITT4 | EFF_F3 | Kaplan Meier Plot of Survival Function Estimates of Time to Qualification for Retreatment in Open Label Phase (4th Treatment) | | IA SAC |

## 9.12.6.2. Final Analyses

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| MAS | | | | | |
| 2.78. | ITT3 | EFF_F1 | Plot of Mean (95%CI) MAS score Profiles in Open Label Phase (3rd Treatment) | <ul><li>Plot data up to Visit 5</li><li>Three treatment arms (240,</li></ul> | SAC |
| 2.79. | ITT4 | EFF_F1 | Plot of Mean (95%CI) MAS score Profiles in Open Label Phase (4th Treatment) | 400 and 240 + 400U) | SAC |
| 2.80. | ITT3 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in MAS score Profiles in Open Label Phase (3rd Treatment) | Plot data up to Visit 5 | SAC |
| 2.81. | ITT4 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in MAS score Profiles in Open Label Phase (4th Treatment) | Three treatment arms (240,<br>400 and 240 + 400U) | SAC |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.82. | ITT3 | EFF_F2 | Plot of Responder rate of MAS score by Visit in Open Label Phase (3rd Treatment) | Plot data up to Visit 5 | SAC |
| 2.83. | ITT4 | EFF_F2 | Plot of Responder rate of MAS score by Visit in Open Label Phase (4th Treatment) | Three treatment arms (240, 400 and 240 + 400U) | SAC |
| DAS | | | | | |
| 2.84. | ITT3 | EFF_F1 | Plot of Mean (95%CI) DAS score (Main Assessment Parameter)<br>Profiles in Open Label Phase (3rd Treatment) | Plot data up to Visit 5 | SAC |
| 2.85. | ITT4 | EFF_F1 | Plot of Mean (95%CI) DAS score (Main Assessment Parameter)<br>Profiles in Open Label Phase (4th Treatment) | Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 2.86. | ITT3 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in DAS score (Main Assessment Parameter) Profiles in Open Label Phase (3rd Treatment) | Plot data up to Visit 5 | SAC |
| 2.87. | ITT4 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in DAS score (Main Assessment Parameter) Profiles in Open Label Phase (4th Treatment) | Three treatment arms (240,<br>400 and 240 + 400U) | SAC |
| 2.88. | ITT3 | EFF_F1 | Plot of Mean (95%CI) DAS score Profiles in Open Label Phase (3rd Treatment) | Plot data up to Visit 5 Create plots by component of | SAC |
| 2.89. | ITT4 | EFF_F1 | Plot of Mean (95%CI) DAS score Profiles in Open Label Phase (4th Treatment) | DAS score Three treatment arms (240 and 400U) | SAC |
| 2.90. | ITT3 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in DAS score<br>Profiles in Open Label Phase (3rd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Create plots by component of DAS score</li> <li>Three treatment arms (240 and 400U)</li> </ul> | SAC |
| 2.91. | ITT4 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in DAS score<br>Profiles in Open Label Phase (4th Treatment) | | SAC |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Numeri | c Rating Scale | for pain | | | |
| 2.92. | ITT3 | EFF_F1 | Plot of Mean (95%CI) NRS for pain Profiles in Open Label Phase (3rd Treatment) | Plot data up to Visit 5 | SAC |
| 2.93. | ITT4 | EFF_F1 | Plot of Mean (95%CI) NRS for pain Profiles in Open Label Phase (4th Treatment) | • Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 2.94. | ITT3 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in NRS for pain Profiles in Open Label Phase (3rd Treatment) | Plot data up to Visit 5 The state of the state of t | SAC |
| 2.95. | ITT4 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in NRS for pain Profiles in Open Label Phase (4th Treatment) | • Three treatment arms (240, 400 and 240 + 400U) | SAC |
| Clinica | Global Impres | sion of Change o | f functional disability | | |
| 2.96. | ITT3 | EFF_F1 | Plot of Mean (95%CI) CGI of functional disability Profiles in Open Label Phase (3rd Treatment) | Plot data up to Visit 5 | SAC |
| 2.97. | ITT4 | EFF_F1 | Plot of Mean (95%CI) CGI of functional disability Profiles in Open Label Phase (4th Treatment) | • Three treatment arms (240, 400 and 240 + 400 U) | SAC |
| Time to | Patient-Repor | ted Onset of Spas | ticity Symptom Relief | | |
| 2.98. | ITT1 | EFF_F3 | Kaplan Meier Plot of Time to Patient-Reported Onset of<br>Spasticity Symptom Relief in Blind Phase | Two treatment arm (240 U and 400U) | SAC |
| 2.99. | ITT2 | EFF_F3 | Kaplan Meier Plot of Time to Patient-Reported Onset of Spasticity Symptom Relief in Open Label Phase (2nd Treatment) | Three treatment arms (240, 400, 240 + 400U) | SAC |
| 2.100. | ITT3 | EFF_F3 | Kaplan Meier Plot of Time to Patient-Reported Onset of Spasticity Symptom Relief in Open Label Phase (3rd Treatment) | | SAC |
| 2.101. | ITT4 | EFF_F3 | Kaplan Meier Plot of Time to Patient-Reported Onset of Spasticity Symptom Relief in Open Label Phase (4th Treatment) | | SAC |

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Time to | Qualification f | or Retreatment | | | |
| 2.102. | ITT1 | EFF_F3 | Kaplan Meier Plot of Survival Function Estimates of Time to Qualification for Retreatment in Blind Phase | Two treatment arm (240 U, 400U) | SAC |
| 2.103. | ITT2 | EFF_F3 | Kaplan Meier Plot of Survival Function Estimates of Time to Qualification for Retreatment in Open Label Phase (2nd Treatment) | Three treatment arm (240, 400, 240 + 400U) | SAC |
| 2.104. | ITT3 | EFF_F3 | Kaplan Meier Plot of Survival Function Estimates of Time to Qualification for Retreatment in Open Label Phase (3rd Treatment) | | SAC |
| 2.105. | ITT4 | EFF_F3 | Kaplan Meier Plot of Survival Function Estimates of Time to Qualification for Retreatment in Open Label Phase (4th Treatment) | | SAC |

207660

# 9.12.7. Safety Tables

## 9.12.7.1. Interim Analyses

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Advers | e Events (AEs) | | | | |
| 3.1. | Safety 1 | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3<br>Treatment Emergent | IA SAC |
| 3.2. | Safety 1 | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term in Blind Phase | Blind Phase (until second dose) See the Section 9.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.3. | Safety 1 | AE1 | Summary of All Adverse Events within 84 days from the initial dose by System Organ Class and Preferred Term | Blind Phase (within 84 days) See the Section 9.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.4. | Safety 2 | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.5. | Safety 1 | AE5A | Summary of All Adverse Events by Maximum Intensity by<br>System Organ Class and Preferred Term | ICH E3 Treatment Emergent Use AE1 or AE1CP if Grade/Intensity not used; otherwise use AE5A/B (with a Total column across all grades/severities, which provides same detail as AE1) | IA SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.6. | Safety 1 | AE5A | Summary of All Adverse Events by Maximum Intensity by<br>System Organ Class and Preferred Term in Blind Phase | Blind Phase (until second dose) See the Section 9.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.7. | Safety 1 | AE5A | Summary of All Adverse Events within 84 days from the initial dose by Maximum Intensity by System Organ Class and Preferred Term | Blind Phase (within 84 days) See the Section 9.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.8. | Safety 2 | AE5A | Summary of All Adverse Events by Maximum Intensity by<br>System Organ Class and Preferred Term in Open Label Phase<br>(2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.9. | Safety 1 | AE3 | Summary of Common (>=3%) Adverse Events by Overall Frequency | ICH E3<br>Treatment Emergent | IA SAC |
| 3.10. | Safety 1 | AE3 | Summary of Common (>=3%) Adverse Events by Overall Frequency in Blind Phase | Blind Phase (until second dose) See the Section 9.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.11. | Safety 1 | AE3 | Summary of Common (>=3%) Adverse Events within 84 days from the initial dose by Overall Frequency | Blind Phase (within 84 days) See the Section 9.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.12. | Safety 2 | AE3 | Summary of Common (>=3%) Adverse Events by Overall Frequency in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.13. | Safety 1 | AE1 | Summary All Drug-Related Adverse Events by System Organ Class and Preferred Term | ICH E3<br>Treatment Emergent | IA SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.14. | Safety 1 | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term in Blind Phase | Blind Phase (until second dose) See the Section 9.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.15. | Safety 1 | AE1 | Summary of All Drug-Related Adverse Events within 84 days from the initial dose by System Organ Class and Preferred Term | Blind Phase (within 84 days) See the Section 9.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.16. | Safety 2 | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term in Open Label Phase in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.17. | Safety 1 | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity | ICH E3 Treatment Emergent AE See the Section 9.4.2 | IA SAC |
| 3.18. | Safety 1 | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity in Blind Phase | Blind Phase (until second dose) See the Section 9.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.19. | Safety 1 | AE5A | Summary of All Drug-Related Adverse Events within 84 days from the initial dose by System Organ Class and Preferred Term and Maximum Intensity | Blind Phase (within 84 days) See the Section 9.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.20. | Safety 2 | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | IA SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.21. | Safety 1 | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Participant and Occurrences) | FDAAA, EudraCT<br>Treatment Emergent AE<br>See the Section 9.4.2 | IA SAC |
| Serious | and Other Sig | nificant Adverse l | Events | | |
| 3.22. | Safety 1 | SAFE_T1 | Summary of Adverse Events of Special Interest | Treatment Emergent AE See the Section 9.4.2 | IA SAC |
| 3.23. | Safety 1 | SAFE_T1 | Summary of Adverse Events of Special Interest in Blind Phase | Blind Phase (until second dose) See the Section 9.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.24. | Safety 1 | SAFE_T1 | Summary of Adverse Events of Special Interest within 84 days from the initial dose | Blind Phase (within 84 days) See the Section 9.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.25. | Safety 2 | SAFE_T1 | Summary of Adverse Events of Special Interest in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 9.4.2 Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.26. | Safety 1 | AE1 | Summary of Non-Fatal Serious Adverse Events | Treatment Emergent AE See the Section 9.4.2 | IA SAC |
| 3.27. | Safety 1 | AE1 | Summary of Non-Fatal Serious Adverse Events in Blind Phase | Blind Phase (until second dose) See the Section 9.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.28. | Safety 1 | AE1 | Summary of Non-Fatal Serious Adverse Events within 84 days from the initial dose | Blind Phase (within 84 days) See the Section 9.4.2. Two treatment arm (240 and 400U) | IA SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.29. | Safety 2 | AE1 | Summary of Non-Fatal Serious Adverse Events in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 9.4.2 Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.30. | Safety 1 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events | Treatment Emergent AE See the Section 9.4.2 | IA SAC |
| 3.31. | Safety 1 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events in Blind Phase | Blind Phase (until second dose) See the Section 9.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.32. | Safety 1 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events within 84 days from the initial dose | Blind Phase (within 84 days) See the Section 9.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.33. | Safety 2 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 9.4.2 Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.34. | Safety 1 | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | FDAAA, EudraCT Treatment Emergent AE See the Section 9.4.2 | IA SAC |
| 3.35. | Safety 1 | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term | IDSL Treatment Emergent AE See the Section 9.4.2 | IA SAC |
| 3.36. | Safety 1 | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term in Blind Phase | Blind Phase (until second dose) See the Section 9.4.2. Two treatment arm (240 and 400U) | IA SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.37. | Safety 1 | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study within 84 days from the initial dose by System Organ Class and Preferred Term | Blind Phase (within 84 days)<br>See the Section 9.4.2.<br>Two treatment arm (240 and 400U) | IA SAC |
| 3.38. | Safety 2 | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| Labora | tory: Chemistry | y | | | |
| 3.39. | Safety 1 | LB1 | Summary of Chemistry by Visit | Summarize data at Screening Visit, in Blind Phase and at Final Visit. | IA SAC |
| 3.40. | Safety 1 | LB1 | Summary of Chemistry Changes from Baseline by Visit | Summarize data at Screening Visit, in Blind Phase and at Final Visit. ICH E3 | IA SAC |
| 3.41. | Safety 1 | LB3 | Summary of Chemistry Shifts from Baseline Relative to Normal Range | | IA SAC |
| 3.42. | Safety 1 | LB15 | Summary of Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 | IA SAC |
| Labora | tory: Hematolo | gy | | | |
| 3.43. | Safety 1 | LB1 | Summary of Haematology by Visit | Summarize data at Screening Visit, in Blind Phase and at Final Visit. | IA SAC |
| 3.44. | Safety 1 | LB1 | Summary of Hematology Changes from Baseline | Summarize data at Screening Visit, in Blind Phase and at Final Visit. ICH E3 | IA SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.45. | Safety 1 | LB3 | Summary of Hematology Shifts from Baseline Relative to Normal Range | | IA SAC |
| 3.46. | Safety 1 | LB15 | Summary of Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 | IA SAC |
| Labora | tory: Urinalysis | ; | | | |
| 3.47. | Safety 1 | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline | ICH E3 | IA SAC |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 3.48. | Safety 1 | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | This display will be presented if liver events occur. | IA SAC |
| 3.49. | Safety 1 | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | IDSL | IA SAC |
| ECG | | | | | |
| 3.50. | Safety 1 | EG1 | Summary of ECG Findings | Summarize data at Screening Visit, in Blind Phase and at Final Visit. IDSL | IA SAC |
| 3.51. | Safety 1 | EG2 | Summary of Change from Baseline in ECG Values by Visit | Summarize data at Screening Visit, in Blind Phase and at Final Visit. IDSL | IA SAC |
| Vital Si | gns | | | | |
| 3.52. | Safety 1 | VS1 | Summary of Change from Baseline in Vital Signs | Summarize data at Screening Visit, in Blind Phase and at Final Visit. ICH E3 | IA SAC |

207660

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| SpO2 | | | | | |
| 3.53. | Safety 1 | SAFE_T2 | Summary of Value and Change from Baseline in SpO2 | | SAC |
| Exposu | re and Treatme | ent Compliance | | | |
| 3.54. | Safety 1 | SAFE_T3 | Summary of Exposure to Study Treatment | ICH E3 | IA SAC |
| 3.55. | Safety 1 | SAFE_T4 | Summary of Extent of Exposure to Study Treatment by Treatment Cycle and Muscle Region | | IA SAC |
| 3.56. | Safety 1 | SAFE_T4 | Summary of Extent of Exposure to Study Treatment by Treatment Cycle and Joint | | IA SAC |

## 9.12.7.2. Final Analyses

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Advers | Adverse Events (AEs) | | | | |
| 3.57. | Safety 1 | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3<br>Treatment Emergent | SAC |
| 3.58. | Safety 1 | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term in Blind Phase | Blind Phase (until second dose) See the Section 9.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.59. | Safety 1 | AE1 | Summary of All Adverse Events within 84 days from the initial dose by System Organ Class and Preferred Term | Blind Phase (within 84 days) See the Section 9.4.2. Two treatment arm (240 and 400U) | SAC |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.60. | Safety 2 | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.61. | Safety 3 | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term in Open Label Phase (3rd Treatment) | Open Label Phase (3rd Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.62. | Safety 4 | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term in Open Label Phase (4th Treatment) | Open Label Phase (4th Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.63. | Safety 1 | AE5A | Summary of All Adverse Events by Maximum Intensity by<br>System Organ Class and Preferred Term | ICH E3<br>Treatment Emergent | SAC |
| 3.64. | Safety 1 | AE5A | Summary of All Adverse Events by Maximum Intensity by<br>System Organ Class and Preferred Term in Blind Phase | Blind Phase (until second dose) See the Section 9.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.65. | Safety 1 | AE5A | Summary of All Adverse Events within 84 days from the initial dose by Maximum Intensity by System Organ Class and Preferred Term | Blind Phase (within 84 days) See the Section 9.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.66. | Safety 2 | AE5A | Summary of All Adverse Events by Maximum Intensity by<br>System Organ Class and Preferred Term in Open Label Phase<br>(2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.67. | Safety 3 | AE5A | Summary of All Adverse Events by Maximum Intensity by<br>System Organ Class and Preferred Term in Open Label Phase<br>(3rd Treatment) | Open Label Phase (3rd Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.68. | Safety 4 | AE5A | Summary of All Adverse Events by Maximum Intensity by<br>System Organ Class and Preferred Term in Open Label Phase<br>(4th Treatment) | Open Label Phase (4th Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.69. | Safety 1 | AE3 | Summary of Common (>=3%) Adverse Events by Overall Frequency | ICH E3<br>Treatment Emergent | SAC |
| 3.70. | Safety 1 | AE3 | Summary of Common (>=3%) Adverse Events by Overall Frequency in Blind Phase | Blind Phase (until second dose) See the Section 9.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.71. | Safety 1 | AE3 | Summary of Common (>=3%) Adverse Events within 84 days from the initial dose by Overall Frequency | Blind Phase (within 84 days) See the Section 9.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.72. | Safety 2 | AE3 | Summary of Common (>=3%) Adverse Events by Overall Frequency in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.73. | Safety 3 | AE3 | Summary of Common (>=3%) Adverse Events by Overall Frequency in Open Label Phase (3rd Treatment) | Open Label Phase (3rd Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.74. | Safety 4 | AE3 | Summary of Common (>=3%) Adverse Events by Overall Frequency in Open Label Phase (4th Treatment) | Open Label Phase (4th Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.75. | Safety 1 | AE1 | Summary All Drug-Related Adverse Events by System Organ Class and Preferred Term | ICH E3<br>Treatment Emergent | SAC |
| 3.76. | Safety 1 | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term in Blind Phase | Blind Phase (until second dose) See the Section 9.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.77. | Safety 1 | AE1 | Summary of All Drug-Related Adverse Events within 84 days from the initial dose by System Organ Class and Preferred Term | Blind Phase (within 84 days) See the Section 9.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.78. | Safety 2 | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term in Open Label Phase in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.79. | Safety 2 | AE1 | Summary of All Drug-Related Adverse Events by System Organ<br>Class and Preferred Term in Open Label Phase in Open Label<br>Phase (3rd Treatment) | Open Label Phase (3rd Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.80. | Safety 2 | AE1 | Summary of All Drug-Related Adverse Events by System Organ<br>Class and Preferred Term in Open Label Phase in Open Label<br>Phase (4th Treatment) | Open Label Phase (4th Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.81. | Safety 1 | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity | ICH E3 Treatment Emergent AE See the Section 9.4.2 | SAC |
| 3.82. | Safety 1 | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity in Blind Phase | Blind Phase (until second dose) See the Section 9.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.83. | Safety 1 | AE5A | Summary of All Drug-Related Adverse Events within 84 days from the initial dose by System Organ Class and Preferred Term and Maximum Intensity | Blind Phase (within 84 days) See the Section 9.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.84. | Safety 2 | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.85. | Safety 2 | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity in Open Label Phase (3rd Treatment) | Open Label Phase (3rd Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.86. | Safety 2 | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity in Open Label Phase (4th Treatment) | Open Label Phase (4th Treatment) See the Section 9.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.87. | Safety 1 | AE3 | Summary of Most Common Serious Drug Related Adverse<br>Events by Overall Frequency | | SAC |
| 3.88. | Safety 1 | AE2 | Summary of Most Common Non-Serious Drug Related Adverse<br>Events by Overall Frequency | | SAC |
| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.89. | Safety 1 | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Participant and Occurrences) | FDAAA, EudraCT<br>Treatment Emergent AE<br>See the Section 9.4.2 | SAC |
| Serious | and Other Sig | nificant Adverse l | Events | | |
| 3.90. | Safety 1 | SAFE_T1 | Summary of Adverse Events of Special Interest | Treatment Emergent AE See the Section 9.4.2 | SAC |
| 3.91. | Safety 1 | SAFE_T1 | Summary of Adverse Events of Special Interest in Blind Phase | Blind Phase (until second dose) See the Section 9.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.92. | Safety 1 | SAFE_T1 | Summary of Adverse Events of Special Interest within 84 days from the initial dose | Blind Phase (within 84 days) See the Section 9.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.93. | Safety 2 | SAFE_T1 | Summary of Adverse Events of Special Interest in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 9.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.94. | Safety 3 | SAFE_T1 | Summary of Adverse Events of Special Interest in Open Label Phase (3rd Treatment) | Open Label Phase (3rd Treatment) See the Section 9.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.95. | Safety 4 | SAFE_T1 | Summary of Adverse Events of Special Interest in Open Label Phase (4th Treatment) | Open Label Phase (4th Treatment) See the Section 9.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.96. | Safety 1 | AE1 | Summary of Non-Fatal Serious Adverse Events | Treatment Emergent AE See the Section 9.4.2 | SAC |
| 3.97. | Safety 1 | AE1 | Summary of Non-Fatal Serious Adverse Events in Blind Phase | Blind Phase (until second dose) See the Section 9.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.98. | Safety 1 | AE1 | Summary of Non-Fatal Serious Adverse Events within 84 days from the initial dose | Blind Phase (within 84 days) See the Section 9.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.99. | Safety 2 | AE1 | Summary of Non-Fatal Serious Adverse Events in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 9.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.100. | Safety 3 | AE1 | Summary of Non-Fatal Serious Adverse Events in Open Label Phase (3rd Treatment) | Open Label Phase (3rd Treatment) See the Section 9.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.101. | Safety 4 | AE1 | Summary of Non-Fatal Serious Adverse Events in Open Label Phase (4th Treatment) | Open Label Phase (4th Treatment) See the Section 9.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.102. | Safety 1 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events | Treatment Emergent AE See the Section 9.4.2 | SAC |
| 3.103. | Safety 1 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events in Blind Phase | Blind Phase (until second dose) See the Section 9.4.2. Two treatment arm (240 and 400U) | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.104. | Safety 1 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events within 84 days from the initial dose | Blind Phase (within 84 days) See the Section 9.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.105. | Safety 2 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 9.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.106. | Safety 3 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events in Open Label Phase (3rd Treatment) | Open Label Phase (3rd Treatment) See the Section 9.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.107. | Safety 4 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events in Open Label Phase (4th Treatment) | Open Label Phase (4th Treatment) See the Section 9.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.108. | Safety 1 | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | FDAAA, EudraCT<br>Treatment Emergent AE<br>See the Section 9.4.2 | SAC |
| 3.109. | Safety 1 | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term | IDSL Treatment Emergent AE See the Section 9.4.2 | SAC |
| 3.110. | Safety 1 | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term in Blind Phase | Blind Phase (until second dose) See the Section 9.4.2. Two treatment arm (240 and 400U) | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.111. | Safety 1 | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study within 84 days from the initial dose by System Organ Class and Preferred Term | Blind Phase (within 84 days) See the Section 9.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.112. | Safety 2 | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.113. | Safety 3 | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term in Open Label Phase (3rd Treatment) | Open Label Phase (3rd Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.114. | Safety 4 | AE1 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term in Open Label Phase (4th Treatment) | Open Label Phase (4th Treatment) See the Section 9.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| Laborat | ory: Chemistry | y | | | |
| 3.115. | Safety 1 | LB1 | Summary of Chemistry by Visit | Summarize data at Screening Visit, in Blind Phase and at Final Visit. | SAC |
| 3.116. | Safety 1 | LB1 | Summary of Chemistry Changes from Baseline by Visit | Summarize data at Screening Visit, in Blind Phase and at Final Visit. ICH E3 | SAC |
| 3.117. | Safety 1 | LB3 | Summary of Chemistry Shifts from Baseline Relative to Normal Range | | SAC |
| 3.118. | Safety 1 | LB15 | Summary of Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Labora | tory: Hematolo | gy | | | |
| 3.119. | Safety 1 | LB1 | Summary of Haematology by Visit | Summarize data at Screening Visit, in Blind Phase and at Final Visit. | SAC |
| 3.120. | Safety 1 | LB1 | Summary of Hematology Changes from Baseline | Summarize data at Screening Visit, in Blind Phase and at Final Visit. ICH E3 | SAC |
| 3.121. | Safety 1 | LB3 | Summary of Hematology Shifts from Baseline Relative to Normal Range | | SAC |
| 3.122. | Safety 1 | LB15 | Summary of Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 | SAC |
| Labora | tory: Urinalysis | <b>,</b> | | | |
| 3.123. | Safety 1 | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline | ICH E3 | SAC |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 3.124. | Safety 1 | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | This display will be presented if liver events occur. | SAC |
| 3.125. | Safety 1 | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | IDSL | SAC |
| ECG | | | | | |
| 3.126. | Safety 1 | EG1 | Summary of ECG Findings | Summarize data at Screening Visit, in Blind Phase and at Final Visit. IDSL | SAC |
| 3.127. | Safety 1 | EG2 | Summary of Change from Baseline in ECG Values by Visit | Summarize data at Screening Visit, in Blind Phase and at Final Visit. IDSL | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Vital Sig | gns | | | | |
| 3.128. | Safety 1 | VS1 | Summary of Change from Baseline in Vital Signs | Summarize data at Screening Visit, in Blind Phase and at Final Visit. ICH E3 | SAC |
| SpO2 | | | | | |
| 3.129. | Safety 1 | SAFE_T1 | Summary of Value and Change from Baseline in SpO2 | | SAC |
| Exposu | re and Treatme | ent Compliance | | | |
| 3.130. | Safety 1 | SAFE_T3 | Summary of Exposure to Study Treatment | ICH E3 | SAC |
| 3.131. | Safety 1 | SAFE_T4 | Summary of Extent of Exposure to Study Treatment by Treatment Cycle and Muscle Region | | SAC |
| 3.132. | Safety 1 | SAFE_T4 | Summary of Extent of Exposure to Study Treatment by Treatment Cycle and Joint | | SAC |

207660

# 9.12.8. Safety Figures

# 9.12.8.1. Interim Analyses

| Safety Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Chemi | Chemistry | | | | |
| 3.1. | Safety1 | SAFE_F1 | Scatter plot of Chemistry at Week 12 versus Baseline in Blind Phase | | IA SAC |
| Hemat | Hematology | | | | |
| 3.2. | Safety1 | SAFE_F1 | Scatter plot of Hematology at Week 12 versus Baseline in Blind Phase | | IA SAC |

207660

# 9.12.9. ICH Listings

# 9.12.9.1. Interim Analyses

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Partici | pant Disposition | | | | · |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | IA SAC |
| 2. | ITT1 | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | IA SAC |
| 3. | Screened | ES9 | Listing of Participants Who Were Rescreened | | IA SAC |
| 4. | ITT1 | BL1 | Listing of Participants for Whom the Treatment Blind was Broken | ICH E3 | IA SAC |
| 5. | ITT1 | TA1 | Listing of Planned and Actual Treatments | IDSL | IA SAC |
| Protoc | ol Deviations | | | | |
| 6. | ITT1 | DV2 | Listing of Important Protocol Deviations | ICH E3 | IA SAC |
| 7. | ITT1 | IE3 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | ICH E3 | IA SAC |
| Popula | ations Analysed | | | | • |
| 8. | Screened | SP3 | Listing of Participants Excluded from Any Population | ICH E3 | IA SAC |
| Demo | graphic and Baseli | ne Characteristics | | | · |
| 9. | ITT1 | DM2 | Listing of Demographic Characteristics | ICH E3 | IA SAC |
| 10. | ITT1 | DM9 | Listing of Race | ICH E3 | IA SAC |
| Prior a | nd Concomitant N | <b>Nedications</b> | | | |
| 11. | ITT1 | CP_CM3 | Listing of Medications | IDSL | IA SAC |
| 12. | ITT1 | POP_L1 | Listing of Rehabilitation | | IA SAC |

| ICH: L | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Expos | Exposure and Treatment Compliance | | | | |
| 13. | ITT1 | POP_L2 | Listing of Exposure Data | ICH E3 | IA SAC |
| Efficac | cy Endpoints | | | | |
| 14. | ITT1 | EFF_L1 | Listing of Modified Ashworth Scales | <ul><li>Values</li><li>Changes from baseline</li><li>Responders</li></ul> | IA SAC |
| 15. | ITT1 | EFF_L1 | Listing of Disability Assessment Scales | <ul><li>Values</li><li>Changes from baseline</li><li>Main Assessment Parameter</li></ul> | IA SAC |
| 16. | ITT1 | EFF_L1 | Listing of Numeric Rating Scale for pain | <ul><li>Values</li><li>Changes from baseline</li></ul> | IA SAC |
| 17. | ITT1 | EFF_L1 | Listing of Clinical Global Impression of Change | <ul><li>CGI by an investigator and a patient</li><li>Values</li></ul> | IA SAC |
| 18. | ITT1 | EFF_L2 | Listing of Patient-Reported Benefit of Injection | | IA SAC |
| 19. | ITT1 | EFF_L3 | Listing of Time to Patient Reported Onset of Spasticity Symptom Relief | | IA SAC |
| 20. | ITT1 | EFF_L3 | Listing of Time to Qualification for Retreatment | | IA SAC |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Advers | se Events | | | | |
| 21. | Safety 1 | AE8 | Listing of All Adverse Events | ICH E3 Including Maximum Intensities, Study Phases for Adverse Events and AESI, SAE flag | IA SAC |
| 22. | Safety 1 | AE7 | Listing of Participant Numbers for Individual Adverse Events | ICH E3 | IA SAC |
| 23. | Safety 1 | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | IA SAC |
| Seriou | s and Other Signi | ficant Adverse Eve | ents | | |
| 24. | Safety 1 | AE8 | Listing of Fatal Serious Adverse Events | ICH E3<br>Including Study Phases for<br>Adverse Events | IA SAC |
| 25. | Safety 1 | AE8 | Listing of Non-Fatal Serious Adverse Events | ICH E3<br>Including Study Phases for<br>Adverse Events | IA SAC |
| 26. | Safety 1 | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | IA SAC |
| 27. | Safety 1 | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3<br>Including Study Phases for<br>Adverse Events | IA SAC |
| Hepato | biliary (Liver) | | | | |
| 28. | Safety 1 | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | This display will be presented if liver events occur. | IA SAC |
| 29. | Safety 1 | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | This display will be presented if liver events occur. | IA SAC |

207660

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| All Lab | oratory | | | • | |
| 30. | Safety 1 | LB5 | Listing of All Laboratory Data for Participants with Any Value Outside Normal Range | ICH E3 | IA SAC |
| 31. | Safety 1 | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | IA SAC |
| 32. | Safety 1 | UR2A | Listing of Urinalysis Data for Participants | ICH E3 | IA SAC |

# 9.12.9.2. Final Analyses

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Partici | pant Disposition | | | - | |
| 33. | ITT1 | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| 34. | Screened | ES9 | Listing of Participants Who Were Rescreened | | SAC |
| 35. | ITT1 | BL1 | Listing of Participants for Whom the Treatment Blind was Broken | ICH E3 | SAC |
| Protoc | ol Deviations | | | | |
| 36. | ITT1 | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC |
| Popula | Populations Analysed | | | | |
| 37. | Screened | SP3 | Listing of Participants Excluded from Any Population | ICH E3 | SAC |

| ICH: L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Demo | graphic and Base | ine Characteristics | | | |
| 38. | ITT1 | DM2 | Listing of Demographic Characteristics | ICH E3 | SAC |
| 39. | ITT1 | DM9 | Listing of Race | ICH E3 | SAC |
| Prior a | and Concomitant I | Medications | | | |
| 40. | ITT1 | CP_CM3 | Listing of Medications | IDSL | SAC |
| 41. | ITT1 | POP_L1 | Listing of Rehabilitation | | SAC |
| Expos | ure and Treatmen | t Compliance | | | |
| 42. | ITT1 | POP_L2 | Listing of Exposure Data | ICH E3 | SAC |
| Efficad | cy Endpoints | | | | |
| 43. | ITT1 | EFF_L1 | Listing of Modified Ashworth Scales | <ul><li>Values</li><li>Changes from baseline</li><li>Responders</li></ul> | SAC |
| 44. | ITT1 | EFF_L1 | Listing of Disability Assessment Scales | <ul><li>Values</li><li>Changes from baseline</li><li>Main Assessment Parameter</li></ul> | SAC |
| 45. | ITT1 | EFF_L1 | Listing of Numeric Rating Scale for pain | Values Changes from baseline | SAC |
| 46. | ITT1 | EFF_L1 | Listing of Clinical Global Impression of Change | <ul> <li>CGI by an investigator and a patient</li> <li>Values</li> </ul> | SAC |
| 47. | ITT1 | EFF_L2 | Listing of Patient-Reported Benefit of Injection | | SAC |
| 48. | ITT1 | EFF_L3 | Listing of Time to Patient Reported Onset of Spasticity Symptom Relief | | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 49. | ITT1 | EFF_L3 | Listing of Time to Qualification for Retreatment | | SAC |
| Advers | se Events | | | | |
| 50. | Safety 1 | AE8 | Listing of All Adverse Events | ICH E3 Including Maximum Intensities, Study Phases for Adverse Events and AESI, SAE flag | SAC |
| 51. | Safety 1 | AE7 | Listing of Participant Numbers for Individual Adverse Events | ICH E3 | SAC |
| 52. | Safety 1 | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | SAC |
| Seriou | s and Other Signi | ificant Adverse Eve | ents | | |
| 53. | Safety 1 | AE8 | Listing of Fatal Serious Adverse Events | ICH E3 Including Study Phases for Adverse Events | SAC |
| 54. | Safety 1 | AE8 | Listing of Non-Fatal Serious Adverse Events | ICH E3 Including Study Phases for Adverse Events | SAC |
| 55. | Safety 1 | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC |
| 56. | Safety 1 | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3<br>Including Study Phases for<br>Adverse Events | SAC |
| Hepato | biliary (Liver) | | | | |
| 57. | Safety 1 | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | This display will be presented if liver events occur. | SAC |
| 58. | Safety 1 | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | This display will be presented if liver events occur. | SAC |
| | | | 1 | II. | |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| All Lab | All Laboratory | | | | |
| 59. | Safety 1 | LB5 | Listing of All Laboratory Data for Participants with Any Value Outside Normal Range | ICH E3 | SAC |
| 60. | Safety 1 | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | SAC |
| 61. | Safety 1 | UR2A | Listing of Urinalysis Data for Participants | ICH E3 | SAC |

207660

#### Appendix 13: List of Preferred Terms / System Organ Class 9.13. of Adverse Events of Special Interest

Adverse Events of Special Interest will be identified based on MedDRA version 20.1.

#### 9.13.1. **Convulsions and Seizures**

This AESI will be identified using Convulsion (SMQ) with narrow scope.

#### 9.13.2. **Respiratory Adverse Events**

This AESI will be identified using the System Organ Class and High Level Term as below.

SOC: "Respiratory, thoracic and mediastinal disorders"

HLT: "Respiratory and pulmonary function diagnostic procedures"

#### 9.13.3. **Possible Distant Spread of Toxin**

This AESI will be identified using the Preferred Term as below.

| Accommodation disorder |
|--------------------------------|
| Aspiration |
| Bradycardia |
| Botulism |
| Bulbar palsy |
| Constipation |
| Cranial nerve palsies multiple |
| Cranial nerve paralysis |
| Diaphragmatic paralysis |
| Diplopia |
| Dry mouth |
| Dysarthria |
| Dysphagia |
| Dysphonia |
| Dyspnoea |
| Extraocular muscle paresis |
| Eyelid function disorder |
| Eyelid ptosis |
| Facial paresis |
| Facial paralysis |

| Hyporeflexia |
|------------------------------|
| Hypotonia |
| Illeus paralytic |
| Muscular weakness |
| Paralysis |
| Paralysis flaccid |
| Paresis cranial nerve |
| Pelvic floor muscle weakness |
| Peripheral nerve palsy |
| Peripheral paralysis |
| Pneumonia aspiration |
| Pupillary reflex impaired |
| Respiratory arrest |
| Respiratory depression |
| Respiratory failure |
| Speech disorder |
| Urinary retention |
| VIIth nerve paralysis |
| Vision blurred |
| Vocal cord paralysis |
| Vocal cord paresis |

## The GlaxoSmithKline group of companies

207660

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | ÷ | Reporting and Analysis Plan for A phase III study (a placebo controlled, randomized, double-blind comparative study and an open-label, uncontrolled study) to evaluate the efficacy and safety of GSK1358820 in patients with post-stroke upper limb spasticity. |
|---|---|---|
| <b>Compound Number</b> | : | GSK1358820 |
| <b>Effective Date</b> | : | 20-AUG-2018 |

# **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 207660.
- This RAP is intended to describe the efficacy and safety analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the interim and final Statistical Analysis Complete (SAC) deliverable.

# **RAP Author(s):**

| Approver | Date | Approval Method |
|-------------------------------------------|------|-----------------|
| PPD | | |
| Lead Statistician (Biostatistics Group 2, | NA | NA |
| Biomedical Data Sciences Dept., Japan) | | |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

207660

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Japan Project Lead (Future Pipelines Discovery Office, Medicines Development, Japan) | 17-Aug-2018 | eSignature |
| Clinical Investigations Lead (Immuno-<br>Inflammation/Oncology TA office, Medicines<br>Development, Japan) | 17-Aug-2018 | eSignature |
| Operations and Science Lead (6, Clinical Operations Dept., Japan) | 17-Aug-2018 | eSignature |
| Data Quality Lead (Data Practice Group,<br>Biomedical Data Sciences Dept., Japan) | 17-Aug-2018 | eSignature |
| Medical Writer (2, Medical Writing Office, Medicines Development, Japan) | 17-Aug-2018 | eSignature |
| Lead Programmer (Statistical Programming & Reporting Group, Biomedical Data Sciences Dept., Japan) | 17-Aug-2018 | eSignature |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Manager (Biostatistics Group 2, Biomedical Data Sciences Dept., Japan) | 20-Aug-2018 | eSignature |
| Department Manager (Biomedical Data Sciences Dept., Japan) | 20-Aug-2018 | eSignature |

207660

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTR( | ODUCTIONRAP Amendments | |
| | 1.1. | NAF Amendments | 0 |
| 2. | SUMN | MARY OF KEY PROTOCOL INFORMATION | |
| | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | 8 |
| | 2.2. | Study Objective(s) and Endpoint(s) | 8 |
| | 2.3. | Study Design | 9 |
| | 2.4. | Statistical Hypotheses / Statistical Analyses | 10 |
| 3. | PLAN | NED ANALYSES | 10 |
| | 3.1. | Interim Analyses | 10 |
| | 3.2. | Final Analyses | 11 |
| 4. | ANAL | YSIS POPULATIONS | 12 |
| | 4.1. | Protocol Deviations | |
| _ | 00110 | DIDEDATIONS FOR DATA ANALYSES AND DATA HANDUNG | |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING /ENTIONS | 13 |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | |
| | 5.2. | Baseline Definitions | |
| | 5.3. | Multicentre Studies | |
| | 5.4. | Examination of Covariates, Other Strata and Subgroups | |
| | | 5.4.1. Covariates and Other Strata | |
| | | 5.4.2. Examination of Subgroups | |
| | 5.5. | Multiple Comparisons and Multiplicity | 15 |
| | 5.6. | Other Considerations for Data Analyses and Data Handling Conventions | 15 |
| | | Conventions | 10 |
| 6. | STUD | Y POPULATION ANALYSES | 15 |
| | 6.1. | Overview of Planned Study Population Analyses | 15 |
| | 6.2. | Participant Disposition and Population | 15 |
| | 6.3. | Protocol Deviation | |
| | 6.4. | Demographic and Baseline Characteristics | |
| | 6.5. | Prior and Concomitant Medications | |
| | 6.6. | Rehabilitation | |
| | 6.7. | Other Surgical Procedure | |
| | 6.8. | Actual dose | 18 |
| 7. | EFFIC | CACY ANALYSES | 19 |
| | 7.1. | Primary Efficacy Analyses | 19 |
| | | 7.1.1. Endpoint / Variables | |
| | | 7.1.2. Summary Measure | |
| | | 7.1.3. Population of Interest | 20 |
| | | 7.1.4. Strategy for Intercurrent (Post-Randomization) Events | 20 |
| | | 7.1.5. Statistical Analyses / Methods | |
| | 7.2. | 7.1.5.1. Statistical Methodology Specification | |
| | 1.4. | Secondary Efficacy Analyses | 21<br>21 |

| | | | 207660 |
|---|---|---|---|
| | | 7.2.2. Summary Measure | 21 |
| | | 7.2.3. Population of Interest | 21 |
| | | 7.2.4. Strategy for Intercurrent (Post-Randomization) Events | 22 |
| | | 7.2.5. Statistical Analyses / Methods | |
| | | 7.2.5.1. Statistical Methodology Specification | |
| | 7.3. | Exploratory Efficacy Analyses | 23 |
| | | 7.3.1. Modified Ashworth Scale (MAS) | 23 |
| | | 7.3.2. Numeric Rating Scale (NRS) for pain | 24 |
| | | 7.3.3. Disability Assessment Scale (DAS) | |
| | | 7.3.4. Clinical Global Impression of Change (CGI) of functional | |
| | | disability | 24 |
| | | 7.3.5. Patient-Reported Benefit of Injection | 24 |
| | | 7.3.6. Time to Patient-Reported Onset of Spasticity Symptom Relief | 25 |
| | | 7.3.7. Time to Qualification for Retreatment | |
| 0 | 0455 | TV ANALYCEC | 00 |
| 8. | | TY ANALYSES | |
| | 8.1.<br>8.2. | Adverse Events Analyses | |
| | 8.3. | Adverse Events of Special Interest Analyses | |
| | o.s.<br>8.4. | Clinical Laboratory Analyses | |
| | 6.4.<br>8.5. | Other Safety Analyses Patient Profiles | |
| | 8.6. | Exposure | |
| | 0.0. | LAPOSUIC | 20 |
| 9. | REFE | RENCES | 31 |
| 10. | APPE | NDICES | 32 |
| | 10.1. | | |
| | | Protocol Population | 32 |
| | 10.2. | Appendix 2: Schedule of Activities | |
| | | 10.2.1. Protocol Defined Schedule of Events | 33 |
| | 10.3. | Appendix 3: Assessment Windows | 36 |
| | | 10.3.1. Definitions of Assessment Windows for Efficacy Analyses (only Final Visit and Withdraw Visit, and only Final | |
| | | Analyses) | 36 |
| | 10.4. | Appendix 4: Study Phases and Treatment Emergent Adverse | |
| | | Events | |
| | | 10.4.1. Study Phases for Concomitant Medication | |
| | | 10.4.2. Study Phases for Adverse Events | 37 |
| | | 10.4.2.1. Definition of Adverse Events of Special Interest | |
| | 10.5. | Appendix 5: Data Display Standards & Handling Conventions | |
| | | 10.5.1. Reporting Process | |
| | | 10.5.2. Reporting Standards | |
| | 10.6. | Appendix 6: Derived and Transformed Data | |
| | | 10.6.1. General | |
| | | 10.6.2. Study Population | |
| | 40.7 | 10.6.3. Efficacy | |
| | 10.7. | Appendix 7: Reporting Standards for Missing Data | |
| | | 10.7.1. Premature Withdrawals | |
| | | 10.7.2. Handling of Missing Data | |
| | 10.8. | 10.7.2.1. Handling of Missing and Partial Dates | |
| | 10.0. | Appondix 0. Values of Fotential cillibal importance | |

207660

# CONFIDENTIAL

| 10.9. | Appendi | x 9: Population Pharmacokinetic (PopPK) Analyses | 45 |
|---|---|---|---|
| | | x 10: Pharmacokinetic / Pharmacodynamic Analyses | |
| | | x 11: Abbreviations & Trade Marks | |
| | 10.11.1. | Abbreviations | 47 |
| | 10.11.2. | Trademarks | 48 |
| 10.12. | Appendi | x 12: List of Data Displays | 49 |
| | 10.12.1. | Data Display Numbering | 49 |
| | 10.12.2. | Mock Example Shell Referencing | 49 |
| | 10.12.3. | Deliverables | 49 |
| | 10.12.4. | Study Population Tables | 50 |
| | | 10.12.4.1. Interim Analyses | |
| | | 10.12.4.2. Final Analyses | 52 |
| | 10.12.5. | Efficacy Tables | |
| | | 10.12.5.1. Interim Analyses | |
| | | 10.12.5.2. Final Analyses | 56 |
| | 10.12.6. | Efficacy Figures | 61 |
| | | 10.12.6.1. Interim Analyses | |
| | | 10.12.6.2. Final Analyses | 65 |
| | 10.12.7. | Safety Tables | |
| | | 10.12.7.1. Interim Analyses | 69 |
| | | 10.12.7.2. Final Analyses | <mark>77</mark> |
| | 10.12.8. | Safety Figures | 90 |
| | | 10.12.8.1. Interim Analyses | |
| | 10.12.9. | ICH Listings | |
| | | 10.12.9.1. Interim Analyses | |
| | | 10.12.9.2. Final Analyses | |
| | 10.12.10 | ).Patient Profiles | 98 |
| | | 10.12.10.1. Final Analyses | 98 |
| 10.13. | | x 13: List of Preferred Terms / System Organ Class of | |
| | | Events of Special Interest | |
| | | Convulsions and Seizures | |
| | | Respiratory Adverse Events | |
| | | Possible Distant Spread of Toxin | |
| 10.14. | Appendi | x 14: Decision Tree to determine Data cutoff visit and date | 102 |

207660

# 1. INTRODUCTION

# 1.1. RAP Amendments

Revision chronology:

| RAP Section | Amendment Details |
|---|---|
| Reporting and Analysis Plan_ | Study207660_Final_V1 02-Apr-2018 |
| Reporting and Analysis Plan_Study207660_Amendment_Final_V1 20-Aug-2018 | |
| Section 2.1. | Added Changes to the Protocol Defined Statistical Analysis Plan |
| Section 3.1.<br>Interim analyses | <ul> <li>Added the definition of the Rehabilitation data used for the interim analysis</li> <li>Changed that Cardiovascular event will not be output in the interim analysis.</li> </ul> |
| Section 5.4.1. | Clarified that a randomization stratum is Baseline MAS value "of the elbow" in this study. |
| Section 6.4. "Summary of Baseline Efficacy Parameter" | <ul> <li>Removed the MAS in the pronation of forearm and shoulder flexors from the summary table since the associated baseline value was not planned to be collected.</li> <li>Clarified a joint location of NRS used for the summary table.</li> <li>Added Baseline MAS score of the elbow as randomization strata in the item list of this summary table.</li> <li>Clarified whether these items are continuous or categorical.</li> </ul> |
| Section 6.7.Section 6.8. | Added the plans for listing of Other Surgical Procedure and displays about actual dose by muscle region and joint. |
| Section 6.6. Category of Frequency | Corrected the category from ">8 days per month" to ">0 and ≤8 days per month" |
| Section 7.1.1. | Clarified which visit the endpoint is. |
| Section 7.2.5.1. Secondary Efficacy Analyses | <ul> <li>Clarified that the Main Assessment Parameter of DAS is used for the secondary efficacy analysis.</li> <li>Clarified whether the fixed effects are categorial or continuous.</li> <li>Clarified the secondary efficacy analysis for the Responder Rate of MAS score.</li> <li>Changed the definition of Responder of MAS in the thumb to that of which denominator does not include the unevaluable thumb.</li> </ul> |
| Section 7.3.1.<br>Modified Ashworth Scale | Removed change from baseline in MAS scores of the pronation of the forearm and should flexors since the corresponding baseline values were not collected. |
| Section 7.3.2.<br>Numeric Rating Scale for Pain | Removed change from baseline in NRS except for that of the elbow since the corresponding baseline values were not collected. |
| Section 7.3.3. Disability Assessment Scale Section 7.3.4. Clinical Global Impression of | Clarified the data used for the summary tables and figures. |

| RAP Section | Amendment Details |
|---|---|
| Change of functional disability | |
| Section 7.3.6. Time to Patient-Reported Onset of Spasticity Symptom Relief | Added the derivation of time to event data in case that the participant does not complete Visit 2 and is withdrawn from study later than the planned date of Visit2. |
| Section 7.3.7. Time to Qualification for retreatment | Removed ITT4 population from the time to qualification for retreatment analysis since participants who were treated 4 times were not assessed to be retreated. |
| Section 8.1. | Added the plan for summary of AE within 84 days by sex and age group. |
| Section 8.3. | Added the details of Worst case urinalysis. |
| Section 8.5. | Added Patient Profiles analysis |
| Section 10.3<br>Assessment Windows | Added the definition of assessment windows for efficacy analyses. The rationale was also added in the section. |
| Section 10.4.1. | Changed the definition of study phases for concomitant medication. |
| Section 10.4.2. | Corrected the definition of Study Phase for AE to that for which AE start time is not used since the previous definition was not that of AE which occurred within 84days. |
| Section 10.5.2. | Added the plan for 95% confidence interval in summary tables for continuous efficacy endpoints. |
| Section 10.6.2<br>Age Category | Changed the definition of Age Category to that of EudraCT requirement. |
| Section 10.12.4. | Corrected the analysis population of "Summary of Race and Racial Combinations" from Enrolled to ITT1 because of baseline characteristics evaluation. |
| Section 10.12.5.2. | Added the summary tables of efficacy endpoints in Open Label Phase (2nd treatment) |
| Section 10.14. | Added the decision tree to determine data cutoff visit and date. |
| Section 10.13. | Removed the two following PT to identify AESI since these were included in the list by mistake. Paralysis flaccid Vilth nerve paralysis |

207660

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There was one change to the originally planned statistical analysis specified in the protocol amendment 02 [(Dated: 06OCT2017)] as the following Table shows:

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Objectives and endpoints | Statistical Analysis Plan | Rationale for Changes |
| Exploratory endpoints Changes in MAS score from baseline in finger, thumb, wrist, elbow, pronation of the forearm and shoulder flexors | Change from baseline in MAS scores of the finger, thumb, wrist and elbow only will be calculated, whereas those of the pronation of the forearm and shoulder will not. | <ul> <li>MAS scores in the pronation of the forearm and shoulder flexors were not collected in Blind Phase.</li> <li>Since baseline value is defined as the latest value prior to the initial treatment, the baseline value would be usually the data at Visit1 in Blind Phase.</li> <li>Therefore, there were not the data of the baseline value in the pronation of the forearm and shoulder flexors, and changes from baseline cannot be calculated.</li> </ul> |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate the efficacy of the injections of 400 units of the product at Week 6 (finger/ wrist flexors: 240 units, elbow flexors: 160 units), comparing to that of 240 units (finger/ wrist flexors: 240 units, elbow flexors: placebo). | The responder rate: The rate of the participants that Modified Ashworth Scale (MAS) score was reduced at least 1 from baseline in the elbow flexors. |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the efficacy of 400 units of the product, comparing to | The responder rate of MAS score from baseline in<br>the finger, thumb and wrist flexors |
| 240 units of the product | Changes in MAS score from baseline in the finger,<br>thumb, wrist and elbow flexors |
| | Changes in Disability Assessment Scale (DAS) from baseline |
| To evaluate the safety and | Adverse events |
| tolerability of the product of 400 | Physical examinations |
| units, comparing to 240 units of the | Clinical laboratory tests (haematology, blood |
| product/ To evaluate the safety | biochemistry, urinalysis) |

207660

| Objectives | Endpoints |
|---|---|
| and tolerability of 400 units of the | Vital signs (heart rate, blood pressure, body |
| product | temperature) |
| Exploratory Objectives | Exploratory Endpoints |
| To evaluate the efficacy of 400 units of the product | Changes in MAS score from baseline in finger,<br>thumb, wrist, elbow, pronation of the forearm and<br>shoulder flexors |
| To evaluate the other efficacy of<br>the product of 400 units, | Changes in Numeric Rating Scale (NRS) for pain from baseline |
| comparing to 240 units of the | Changes in other items of DAS from baseline |
| product/ To evaluate the other | Clinical Global Impression of Change (CGI) of |
| efficacy of 400 units of the product | functional disability by an investigator |
| | CGI of functional disability by a patient |
| | Time to patient-reported onset of spasticity symptom relief |
| | Patient-reported benefit of injection |
| | Time to qualification for retreatment |
| To evaluate neutralizing antibody production | Testing for neutralizing antibody |

# 2.3. Study Design



207660

| Overview of S | Overview of Study Design and Key Features |
|---|---|
| | <ul> <li>muscles that act on the finger (including thumb flexors) and wrist flexors, and 160 units into the muscles that act on the elbow flexors. A total of 400 units of the product will be injected.</li> <li>In the 240-unit group, 240 units of the product will be injected into the muscles that act on the finger (including thumb flexors) and wrist flexors. Placebo will be injected into the muscles that act on the elbow flexors. A total of 240 units of the product will be injected.</li> <li>In the Open-label phase, a total of 400 units will be injected in both groups.</li> <li>The product can be injected up to 3 times after completion of Part 1 in the blind phase. Participants whom the investigator considers as eligible for the injections will be treated. The next injections cannot be performed until the eligibility of the participant has been confirmed by the investigator.</li> <li>The muscle to be injected and the dose will be decided by the investigator based on the patient's symptoms, and a total dose of 400 units of the product will be injected in a divided dose. For the muscles that the investigator considers as unnecessary to be treated, an injection may be skipped. The involving muscle and the dose do not have to be same each time always.</li> </ul> |
| Treatment<br>Assignment | <ul> <li>Number of participants (randomized participants): 120 (60 per group)</li> <li>GSK RandAll NG will be used to generate the randomization schedule.</li> <li>The randomization will be stratified by the MAS score (3 or 4) in the elbow flexors at Day1</li> </ul> |
| Interim<br>Analysis | Interim analysis is planned in this study as described in 3.1. |

# 2.4. Statistical Hypotheses / Statistical Analyses

No formal hypothesis will not be tested.

# 3. PLANNED ANALYSES

# 3.1. Interim Analyses

The interim planned primary analyses will be performed after the completion of the following sequential steps:

1. All participants (except for early termination) complete the visit at Week 24 of the initial dose as defined in the protocol. The participants who complete that visit are defined as below.

The participant is re-treated at Week 12 visit in Blind Phase and completes the Week 12 visit in Open-label Phase.

The participant is re-treated at Week 16 visit in Blind Phase and completes the Week 12 visit in Open-label Phase.

207660

The participant is re-treated at Week 20 visit in Blind Phase and completes the Week 4 visit in Open-label Phase.

The participant completes the Week 24 visit in Blind Phase.

- 2. All required database cleaning activities have been completed and interim database release and database freeze has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG procedures.
- 5. Interim analyses will be performed.

The interim analyses will be performed for regulatory submission. However subject level data will not be disclosed to people who work at the sites including investigators.

All planned interim analyses (i.e. Study population, Efficacy and Safety analyses) will be performed using data up to Week 24 visit for all participants.

For Rehabilitations, the data at Screening visit and Week 12 visit will be used for the interim analysis.

For Adverse Events, Liver Events and Medication, the data up to Week 24 visit is defined by using the start date. If the start date of these data is earlier than or same as the date of Week 24 visit defined above, these data will be included in the data up to Week 24 visit. Otherwise the data will not. See the decision tree (Appendix 14) to determine the Week 24 visit and date of the participant.

Cardiovascular Events will not be output in the interim analysis.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. Final analyses will be performed.

207660

#### **ANALYSIS POPULATIONS** 4.

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | Comprise of all screened participants | Study Population |
| Enrolled | Comprise of all participants who meet the eligibility criteria at a screening and Day 1 visit. | Study Population |
| Intent-To-Treat 1 | This population consists of all participants who | Study Population |
| (ITT1) | are randomized in the study and who have at least 1 post-baseline efficacy assessment: | Efficacy |
| | ITT is the primary efficacy analysis population,<br>and the participants will be analyzed in line<br>with the randomized treatment group | |
| | Any participant who receives a study treatment<br>randomization number will be considered to<br>have been randomized. | |
| ITT2 | This population consists of all participants in | Study Population |
| | ITT1 population, who have at least 2 study | Efficacy |
| | treatments and who have at least 1 efficacy assessment after the 2nd treatment. | |
| ITT3 | This population consists of all participants in | Study Population |
| | ITT2 population, who have at least <b>3</b> study treatments and who have at least 1 efficacy | Efficacy |
| | assessment after the 3rd treatment. | · |
| ITT4 | This population consists of all participants in | Study Population |
| | ITT3 population, who have <b>4</b> study treatments and who have at least 1 efficacy assessment after the 4th treatment. | Efficacy |
| Safety1 | This population consists of all participants who are randomized in the study and who receive | Safety |
| | study treatment at least once | |
| | The participants will be analyzed based on the treatment actually given. | |
| Safety2 | This population consists of all participants in<br>Safety1 population, who receive study<br>treatment at least twice. | Safety |
| | The participants will be analyzed based on the treatment actually given. | |
| Safety3 | This population consists of all participants who are randomized in the study and who receive study treatment at least three times | Safety |
| | The participants will be analyzed based on the | |

207660

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | treatment actually given. | |
| Safety4 | This population consists of all participants in<br>Safety1 population, who receive study<br>treatment four times. | Safety |
| | The participants will be analyzed based on the treatment actually given. | |

#### NOTES:

 Please refer to Appendix 12: List of Data Displays which details the population to be used for each displays being generated.

## 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided. This listing will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | Reporting | |
| Code | Description | Description | Order in TLF |
| Α | GSK1358820 240U | GSK1358820 240U | 1 |
| В | GSK1358820 400U | GSK1358820 400U | 2 |

Treatment comparisons will be displayed as follows using the descriptors as specified:

1. GSK1358820 400U vs GSK1358820 240U

207660

## 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline. These baseline values will be used for all analyses in both Blind Phase and Open Label Phase.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

## 5.3. Multicentre Studies

No data will be analysed by center.

# 5.4. Examination of Covariates, Other Strata and Subgroups

## 5.4.1. Covariates and Other Strata

The list of covariates and other strata may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses. Additional covariates and other strata of clinical interest may also be considered.

| Category | Details |
|----------|------------------------------------------|
| Strata | Baseline MAS value of the elbow (3 or 4) |

#### 5.4.2. Examination of Subgroups

The list of subgroups may be used in descriptive summaries and statistical analyses. Additional subgroups of clinical interest may also be considered.

- If the percentage of participants is small within a particular subgroup, then the subgroup categories may be refined prior to unblinding the trial.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.

| Subgroup | Categories |
|---|---|
| Baseline MAS value of the elbow | 3 or 4 |
| Baseline Rehabilitation | |
| Task-specific practice | Yes, or No |
| Muscle strengthening exercise | The subgroup analyses will be conducted by each rehabilitation use. |
| Stretching/Range of motion | |
| exercise | |
| Splinting/Orthoses | |
| Taping | |
| Positioning aids | |

207660

# 5.5. Multiple Comparisons and Multiplicity

No multiplicity adjustment is considered in this study because no statistical hypothesis will be tested.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---|---|
| Section 10.3 | Appendix 3: Assessment Windows |
| Section 10.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| Section 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| Section 10.6 | Appendix 6: Derived and Transformed Data |
| Section 10.7 | Appendix 7: Reporting Standards for Missing Data |
| Section 10.8 | Appendix 8: Values of Potential Clinical Importance |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Screened, Enrolled and ITT populations, unless otherwise specified.

Study population analyses including analyses of participant's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and rehabilitations will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 12: List of Data Displays.

# 6.2. Participant Disposition and Population

The number and percentage of those participants below will be presented by treatment group and total.

- Participants who completed the Week 24 and who withdrew early from study by Week 24 (including the reasons for early withdrawal)
- Participants who completed the study and who withdrew early from study (including the reasons for early withdrawal)
- Participants who passed screening and who failed screening (including the reasons for screen failure)
- Participants at each centre
- Participants included in each population defined in the Section 4.

207660

These items below will be listed.

- The reasons for early withdrawal and screen failure.
- Participants who were rescreened.
- Participants for whom the treatment blind was broken.
- Planned and actual treatments
- Participants excluded from any population defined in the Section 4.

## 6.3. Protocol Deviation

The number and percentage of participants with important protocol deviation will be presented by treatment group. This summary will not include subcategories

Important protocol deviations and participants with inclusion/exclusion criteria deviation will be listed.

# 6.4. Demographic and Baseline Characteristics

These parameters as below will be summarized by treatment group and total.

- Demographic data (age, sex, ethnicity, weight, height, body mass index(BMI), race and racial combinations)
- Baseline Efficacy Parameter
  - o Continuous variable
    - Modified Ashworth Scales in finger, thumb, wrist and elbow
    - Numeric Rating Scale for pain in elbow
    - Disability Assessment Scale (Main Assessment Parameter)
    - Disability Assessment Scale (Hygiene, Pain, Dressing and Limb posture)
  - o Categorical variable
    - Baseline MAS score of the elbow (3 or 4, original values) as randomization strata
    - The selected item as a Main Assessment Parameter of DAS out of the 4 items
      - Hygiene
      - Pain
      - Dressing
      - Limb posture

207660

## 6.5. Prior and Concomitant Medications

All medication used in this study will be coded according to drug name as defined in the GSK Drug Dictionary. The relationship between the ATC level 1 and ingredient will be summarized for the all prior and concomitant medications, respectively.

## 6.6. Rehabilitation

Screening

The number and percentage of Rehabilitations will be presented.

• Treatment phase

The category and frequency of Rehabilitations will be collected on eCRF. The number and percentage of each Rehabilitation will be presented in Blind Phase. The category and frequency of Rehabilitations in all treatment phase will be listed.

• Category and Frequency

The categories of Rehabilitation are as below:

- Task-specific practice
- Muscle strengthening exercise
- Stretching/Range of motion exercise
- Splinting/Orthoses
- Taping
- Positioning aids

The category of frequency which will be collected on CRF is defined as below:

- No practice
- $\circ$  > 0 and  $\leq$  8 days per month
- $\circ$  > 8 and  $\leq$  16 days per month
- $\circ$  > 16 and  $\leq$  24 days per month
- $\circ$  > 24 days per month

# 6.7. Other Surgical Procedure

The other surgical procedure except for Rehabilitation will be listed by treatment group.

207660

# 6.8. Actual dose

The dosage in each muscle and joint to which more than 0 unit of GSK1358820 is administered will be summarized by treatment group and treatment cycle. The Relationship between Muscle Region and Joint is shown below in each treatment phase.

## • Muscle Region

If a muscle region of a participant is not treated, the muscle will not be included when calculating the summary statistics.

| Example | Dosage of Biceps brachii (unit) | Mean |
|---|---|---|
| Subject PPD | 0 | |
| Subject | 40 | (40 + 80 + 120) / 3 = 80 units |
| Subject | 80 | (40 + 80 + 120) / 3 - 80 units |
| Subject | 120 | |

## • Joint

If no muscle region of a Joint of a Participant is treated, the corresponding joint will not be included when calculating the summary statistics.

| <b>Example</b> | Muscle Region | Dosage of each Muscle (unit) | Dosage of<br>Elbow (unit) | Mean |
|---|---|---|---|---|
| SubjectPPD | Biceps brachii | 0 | | |
| | Brachialis | 0 | 0 | |
| | Brachioradialis | 0 | | |
| Subject | Biceps brachii | 0 | | |
| | Brachialis | 20 | 100 | (100 + 110 + |
| | Brachioradialis | 80 | | (100 + 110 + 180) / 3 = 130 |
| Subject | Biceps brachii | 10 | | units |
| | Brachialis | 40 | 110 | units |
| | Brachioradialis | 60 | | |
| Subject | Biceps brachii | 40 | | |
| | Brachialis | 60 | 180 | |
| | Brachioradialis | 80 | | |

## • Blind Phase

| Joint | Each muscle region |
|-------|-----------------------|
| | Biceps brachii |
| Elbow | Brachialis |
| | Brachioradialis |
| VA/-: | Flexor carpi radialis |
| Wrist | Flexor carpi ulnaris |

207660

| Joint | Each muscle region |
|----------|--------------------------------|
| Finger | Flexor digitorum profundus |
| Finger | Flexor digitorum superficialis |
| Thursela | Flexor pollicis longus |
| Thumb | Adductor pollicis |

# • Open Label Phase

| Joint | Each muscle region |
|----------|--------------------------------|
| | Biceps brachii |
| Elbow | Brachialis |
| | Brachioradialis |
| VAL::-4 | Flexor carpi radialis |
| Wrist | Flexor carpi ulnaris |
| | Flexor digitorum profundus |
| Finger | Flexor digitorum superficialis |
| | Lumbricales interossei |
| | Flexor pollicis longus |
| Thumb | Adductor pollicis |
| | Opponens |
| F | Pronator teres |
| Forearms | Pronator quadratus |
| | Teres major |
| Shoulder | Latissimus dorsi |
| Snoulder | Pectoralis major |
| | Subscapularis |

# 7. EFFICACY ANALYSES

# 7.1. Primary Efficacy Analyses

# 7.1.1. Endpoint / Variables

The primary endpoint is the responder rate of MAS score in the elbow flexors at Week 6 of the initial dose.

# 7.1.2. Summary Measure

The summary measure is the difference in the responder rate of MAS score in the elbow flexors.

207660

## 7.1.3. Population of Interest

The primary efficacy analyses will be based on the Intent-To-Treat 1 population, unless otherwise specified.

# 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

Intercurrent event: early withdrawal from study

Strategy: if MAS score is missing because of an early withdrawal from the study, the participant will be regarded as a non-responder.

# 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics and listed.

## 7.1.5.1. Statistical Methodology Specification

### **Endpoint / Variables**

Responder Rate of MAS in the elbow flexors at Week 6 of the initial dose

## **Model Specification**

- To summarize the primary endpoint without statistical model
  - The primary endpoint will be calculated as the proportion of participants whose MAS score decreased by at least 1 level from the baseline in the ITT1 population.
  - The intergroup difference in the responder rate and its 95% confidence interval (Waldtype) will be computed.

#### **Data Convention**

• The MAS scores, 0, 1, 1+, 2, 3 and 4 will be encoded to 0, 1, 2, 3, 4 and 5, respectively, for the analyses.

## **Definition of Responder and Responder rate**

"Responder" is defined as a participant whose MAS score decrease by at least 1 level from the baseline.

Responder Rate will be calculated as below.

Responder Rate (%) = (Number of Responders) / (Number of participants in ITT1 population) x 100

• If MAS score of a given participant is missing at Week 6, then this participant will be regarded as a non-responder.

## **Model Results Presentation**

The difference in the responder rate (400 units – 240 units) and its associated 95% CI will be presented.
207660

#### **Subgroup Analyses (Rehabilitation)**

- Subgroup analyses will be performed by baseline rehabilitation in the Section 5.4.
- The difference (400 units 240 units) and its 95% CI will be presented.

#### **Subgroup Analyses (baseline MAS score)**

- Subgroup analyses will be performed by baseline MAS score of the elbow (3 or 4) used as randomization strata.
- The difference (400 units 240 units) and its 95% CI will be presented.

#### **Supportive Analyses**

- The difference in the responder rate will be estimated using Mantel-Haenszel method to consider a stratification factor, that is baseline MAS score of the elbow (3 or 4).
- Mantel-Haenszel rate difference (400 units 240 units) and its 95% CI will be calculated.

## 7.2. Secondary Efficacy Analyses

#### 7.2.1. Endpoint / Variables

Secondary Efficacy Endpoints are the following items in Blind Phase:

- MAS scores in the elbow, finger, thumb and wrist flexors.
- Change from baseline in MAS scores
- Responder rate of MAS in the elbow, finger, thumb and wrist flexors.
- DAS score (Main Assessment Parameter)
- Change from baseline in DAS score (Main Assessment Parameter)

#### 7.2.2. Summary Measure

Summary Measures are as below.

- The differences in the responder rate of MAS scores
- The differences in the least square means of changes from baseline in MAS scores
- The differences in the least square means of changes from baseline in DAS scores

#### 7.2.3. Population of Interest

The secondary efficacy analyses will be based on the Intent-To-Treat 1 population, unless otherwise specified.

The secondary efficacy analyses will be performed for only double blind phase. All efficacy analyses for open -label phase and other endpoints for double blind phase will be done as exploratory.

207660

Unless specified otherwise, the data up to Week 12 of treatment will be summarized during the double-blind period. This is because this study allows to re-treat. In other words, after 12 weeks, only participants who have a smaller MAS score would remain and the difference of the change from baseline in MAS between 240 units and 400 units would be attenuated. Therefore, the data up to Week 12 of initial treatment will be analysed as secondary statistical analyses. This is the case for exploratory analyses for open label period (i.e. the data up to week 12 of re-treatment will be summarized). Listing will include the data after week 12 of treatment/re-treatment.

#### 7.2.4. Strategy for Intercurrent (Post-Randomization) Events

Intercurrent event: early withdrawal from study.

Strategy for dichotomous data: the participant will be regarded as a non-responder.

Strategy for continuous data: the missing data will be removed from the analyses.

#### 7.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented and listed.

#### 7.2.5.1. Statistical Methodology Specification

#### Secondary Efficacy Analysis

#### **Endpoint / Variables**

• Change from baseline in MAS in each joint and DAS (Main Assessment Parameter) scores

#### **Model Specification**

- The endpoint will be analyzed using a mixed model for repeated measures (MMRM)
- Terms fitted in the MMRM will include the items below as fixed effects.
  - Categorical effect
    - Treatment
    - o Visit
    - Treatment-by-visit interaction
  - Continuous effect
    - o Baseline value in MAS of each joint or in DAS (Main Assessment Parameter)
    - Baseline-by-visit interaction
- An unstructured variance structure will be used to model the within-participant errors, shared across treatments.
- The empirical sandwich estimator will be used to estimate the standard errors.

#### **Model Checking & Diagnostics**

• If the model will not converge with unstructured variance. AR(1) variance structure can be

207660

#### **Secondary Efficacy Analysis**

used.

#### Model Results Presentation

Adjusted means (least square means) and corresponding standard errors of means will be
presented for each treatment by visit, together with estimated treatment differences (400 units

– 240 units) and the corresponding 95% CI.

#### **Data included in Model**

The dataset including only data until week 12 after the first treatment will be used.

#### **Secondary Efficacy Analysis**

#### **Endpoint / Variables**

- Responder Rate of MAS score in each joint at all visit
- Responder is defined as well as primary endpoint.
- For the elbow, finger and wrist flexors.
  - Responder rate (%) = (Number of Responders) / (Number of participants in ITT1 population) x 100
- For the thumb flexors
  - Responder rate (%) = (Number of Responders) / (Number of Participants in ITT1 population, except for the participants of which thumb was not evaluable, x 100.
  - In case that the thumb was not evaluable, MAS score data will be entered as "Not Applicable".

#### **Model Specification**

See primary endpoint section.

#### **Data Convention**

See primary endpoint section.

#### **Supportive Statistical Analyses**

- See supportive statistical analyses for primary efficacy analyses section.
- Baseline MAS score of the elbow as a stratification factor will be used for the Mantel Haenszel Estimator, regardless of the Responder rate of MAS score in the other joint.

## 7.3. Exploratory Efficacy Analyses

#### 7.3.1. Modified Ashworth Scale (MAS)

These analyses will be based on ITT 2, 3 and 4 populations.

Values and changes from baseline in MAS scores in finger, thumb, wrist and elbow will be summarised using descriptive statistics, graphically presented and listed by visit and treatment cycle. In addition, the number and percentage of Responder in MAS score of each joint will be presented by visit and treatment cycle including graphically. The

207660

Responder rate will be the proportion of the responder in the corresponding population, except for the participant of which joint was not evaluable. MAS score values in pronation of the forearm and shoulder flexors will be summarised using descriptive statistics, graphically presented and listed by visit and treatment cycle. Data up to Week 12 in each treatment cycle will be used for summary tables and Figures, whereas all data will be listed.

#### 7.3.2. Numeric Rating Scale (NRS) for pain

These analyses will be based on ITT 1, 2, 3 and 4 populations.

Values and changes from baseline in NRS of the elbow for pain will be summarised using descriptive statistics, graphically presented and listed by visit, treatment cycle and evaluated part. NRS values except for that of elbow flexors will be summarised using descriptive statistics, graphically presented and listed by visit and treatment cycle. Data up to Week 12 in each treatment cycle will be used for summary tables and Figures, whereas all data will be listed.

#### 7.3.3. Disability Assessment Scale (DAS)

These analyses will be based on ITT 1, 2, 3 and 4 populations.

Values and changes from baseline in all items of DAS will be summarised using descriptive statistics, graphically presented and listed by visit and treatment cycle. Data up to Week 12 in each treatment cycle will be used for summary tables and Figures, whereas all data will be listed.

## 7.3.4. Clinical Global Impression of Change (CGI) of functional disability

These analyses will be based on ITT 1, 2, 3 and 4 populations.

Values of the variables below will be summarised using descriptive statistics, graphically presented and listed by visit and treatment cycle. Data up to Week 12 in each treatment cycle will be used for summary tables and Figures, whereas all data will be listed.

CGI of functional disability by an investigator

CGI of functional disability by a patient

#### 7.3.5. Patient-Reported Benefit of Injection

These analyses will be based on ITT 1, 2, 3 and 4 populations.

The number and percentage of patient-reported benefit of injection will be presented and listed by visit and treatment cycle.

207660

#### 7.3.6. Time to Patient-Reported Onset of Spasticity Symptom Relief

These analyses will be based on ITT 1, 2, 3 and 4 populations.

Time to event data will be summarized using the descriptive statistics below and listed.

- The number of events and censored cases.
- Median survival time with the associated 95% CI.
- 25% and 75% survival time.

Survival analyses will be conducted using a Kaplan-Meier method. To graphically compare the survival functions between 400 units and 240 units, the analysis will be conducted based on ITT 1 population whereas the analyses will be based on ITT 2, 3 and 4 populations to assess the survival time by treatment cycle. Participants who are withdrawn from this study before Visit 2 are censored at the withdrawal date. All other participants who do not experience the event and is not withdrawn from study or of whom the date of Visit 2 is missing and is not withdrawn from study before the planned date of Visit 2 are censored at the Visit 2.

Survival function estimates will be summarized (survival probabilities and the number of participants at risk per time to event, and median in survival time) based on Kaplan Meier method. Kaplan Meier plots will be presented.

#### 7.3.7. Time to Qualification for Retreatment

These analyses will be based on ITT 1, 2 and 3 populations.

The number and percentage of event of interest will be presented by visit. Time to event data will be summarized using the descriptive statistics below and listed.

- The number of events and censored cases.
- Median survival time with the associated 95% CI.
- 25% and 75% survival time.

Survival analyses will be conducted using a Kaplan-Meier method. To graphically compare the survival functions between 400 units and 240 units, the analysis will be conducted based on ITT 1 population whereas the analyses will be based on ITT 2 and 3 populations to assess the survival time by treatment cycle. Participants who are withdrawn from this study before the events are censored at the withdrawal date. All other participants who do not experience the event and is not withdrawn from study are censored at the Last Observed Visit at the interim analyses or the final analyses.

Survival function estimates will be summarized (survival probabilities and the number of participants at risk per time to event, and median in survival time) based on Kaplan Meier method. Kaplan Meier plots will be presented.

Note that the retreatment is not allowed within 83 days from the previous treatment. Therefore, this event will not occur before 83 days later after the treatment/re-treatment.

207660

#### 8. SAFETY ANALYSES

The safety analyses will be based on the Safety 1, 2, 3 and 4 populations, unless otherwise specified.

## 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 12: List of Data Displays.

Adverse events that occurred in the overall study period, blinded period and open-label period will be summarized for each treatment group. The treatment group is based on dose actually given in blind period. For the blinded period, 2 patterns of analyses on adverse events will be performed, one is on adverse events that occurred between the initial dose and the first dose in the open-label period (or at the completion of study if no dose is given in the open-label period or at the study withdrawal), and another one is on adverse events that occurred within 84 days from the initial dose.

Overall study period (Treatment Emergent AEs)

#### Blind phase

- 1. AEs occurred between the initial dose and the first dose in the open-label period (or at the completion of study if no dose is given in the open-label period or at the study withdrawal)
- 2. AEs occurred within 84 days from the initial dose

#### Open-label phase

- 3.01. AEs occurred during 2nd treatment cycle.
- 3.02. AEs occurred during 3rd treatment cycle.
- 3.03. AEs occurred during 4th treatment cycle.

The number and percentages of participants who experience at least one AE will be presented for each category of AE listed as below by treatment group.

- All Treatment Emergent AEs (by SOC and PT, by SOC, PT and Maximum Intensity)
- Common AEs ( $\geq 3\%$ ) (by overall frequency)
- Drug Related AEs (by SOC and PT, by SOC, PT and Maximum Intensity)
- Non-Fatal Serious AEs
- Drug Related Non-Fatal Serious AEs
- AEs Leading to Withdrawal from Study (by SOC and PT)
- Most Common Serious Drug Related AEs (by overall frequency)
- Most Common Non-Serious Drug Related AEs (by overall frequency)
- Common ( $\geq$  5%) Non-Serious AEs (by SOC and PT)
  - o Number of Participant and Occurrences will be presented.

207660

The number and percentages of participants wo experience at least one AE will be presented for AEs below. This summary will include only AE occurred within 84 days in Blind Phase.

- Common AEs (>= 3%) within 84 days in Blind Phase by Sex (by overall frequency)
- Common AEs (>= 3%) within 84 days in Blind Phase by Age group (Age < 65, Age >= 65) (by overall frequency)

"Common (>= 3%) AEs" is defined as the percentage of AEs is more than and equal to 3% in either treatment group.

In addition, the items below will be listed.

- All AEs
- Participant Numbers for Individual AEs
- Fatal Serious AEs
- Non-Fatal Serious AEs
- Reasons for Considering as a Serious AE
- AEs Leading to Withdrawal from Study
- Relationship between AE SOC, PT and Verbatim Text.

## 8.2. Adverse Events of Special Interest Analyses

Adverse Events of Special Interest are defined as below.

- Convulsions and Seizures
- Respiratory Adverse Events
- Possible Distant Spread of Toxin

The number and percentage of AESI will be presented by treatment cycle and treatment group. The details of how to identify are described in the Appendix 13.

## 8.3. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 12: List of Data Displays.

These data at Screening Visit, in Blind Phase and at Final Visit will be summarized by visit. Data at all visits for participants with any value outside normal range will be listed.

Values and change from baseline in Chemistry Laboratory tests and Hematology laboratory tests will be summarized by treatment group and visit.

Worst case results relative to normal range from baseline will be presented for Chemistry, Hematology and Urinalysis. Worst case urinalysis results relative to baseline for protein (category: NEG, TRA, 1+, 2+, 3+, 4+) and occult blood (category: NEG, TRA, 1+, 2+, 3+) urinalysis only will be summarized by treatment group. The categories for worst case

207660

are: No Change/Decreased, Any Increase, Increase to TRA, Increase to 1+, Increase to 2+, Increase to 3+, Increase to 4+. The categorization is determined by comparing the baseline category to the worst case post-baseline category. The determination of the worst case post-baseline takes into account both planned and unscheduled assessments. The percentages are based on the number of subjects in the treatment group with data for the test post-baseline. Subjects with missing baseline value are to be assumed to have normal/within range baseline value.

Shifts from baseline relative to normal range will be summarized by treatment group and visit for Chemistry and Hematology values.

Scatter plot of Chemistry and Hematology at Week 12 versus baseline in Blind Phase will be presented.

The outputs regarding liver events will not be presented unless at least one liver event is observed. See the details in the Appendix 12.

#### 8.4. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 12: List of Data Displays.

These above data at Screening Visit, in Blind Phase and at Final Visit will be summarized by visit. These analyses will not include the data at QRV, in Open Label Phase and at Early Withdrawal, whereas all the data at all visit will be listed for final analyses.

ECG findings (Normal, Abnormal – not clinically significant, Abnormal -clinically significant) will be summarized by visit.

Values and changes from baseline in ECG and vital sign data will be summarized by visit.

Values and changes from baseline in SpO2 will be summarized and listed by visit. Data at Screening visit, Visit 1 and 5 in Blind Phase and Final Visit will be summarized and those at all visits will be listed including values and changes from baseline.

#### 8.5. Patient Profiles

Listing for patient profiles will be produced at only Final Analyses if at least one event is reported below.

CV event (

Arrhythmias,

Congestive Heart Failure,

Cerebrovascular Events/Stroke and Transient Ischemic Attack,

Deep Vein Thrombosis (DVT)/ Pulmonary Embolism (PE),

Myocardial Infarction (MI)/ Unstable Angina (UA),

207660

Peripheral Arterial Thromboembolism, Pulmonary Hypertension, Revascularization, Valvulopathy) And Death.

## 8.6. Exposure

The number and percentage of participants treated will be presented by the number of injection.

#### Blind Phase

The dosage will be summarized by muscle region below, Joint and total. The dosage will be listed by muscle region, joint and total.

| Joint | Each muscle region |
|---------|--------------------------------|
| | Biceps brachii |
| Elbow | Brachialis |
| | Brachioradialis |
| Wrist | Flexor carpi radialis |
| WHSt | Flexor carpi ulnaris |
| Einger | Flexor digitorum profundus |
| Finger | Flexor digitorum superficialis |
| Thumb | Flexor pollicis longus |
| indillo | Adductor pollicis |

## • Open Label Phase

The dosage will be summarized by treatment phase (2nd, 3rd and 4th treatment), muscle region below, Joint and total. The dosage will be listed by treatment phase and muscle region, Joint and total.

| Joint | Each muscle region |
|--------|--------------------------------|
| | Biceps brachii |
| Elbow | Brachialis |
| | Brachioradialis |
| Wrist | Flexor carpi radialis |
| WHSt | Flexor carpi ulnaris |
| | Flexor digitorum profundus |
| Finger | Flexor digitorum superficialis |
| | Lumbricales interossei |
| Thumb | Flexor pollicis longus |

## 207660

| Joint | Each muscle region |
|----------|--------------------|
| | Adductor pollicis |
| | Opponens |
| Forcermo | Pronator teres |
| Forearms | Pronator quadratus |
| | Teres major |
| Chaulder | Latissimus dorsi |
| Shoulder | Pectoralis major |
| | Subscapularis |

207660

## 9. REFERENCES

GlaxoSmithKline Document Number 2017N315029\_02 Study ID 207660. A phase III study (a placebo controlled, randomized, double-blind comparative study and an openlabel, uncontrolled study) to evaluate the efficacy and safety of GSK1358820 in patients with post-stroke upper limb spasticity. Report Date 06-Oct-2017.

Study Reference Manual, Study ID 207660. A phase III study (a placebo controlled, randomized, double-blind comparative study and an open-label, uncontrolled study) to evaluate the efficacy and safety of GSK1358820 in patients with post-stroke upper limb spasticity. Effective Date 01-Jun-2018

207660

## 10. APPENDICES

## 10.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

Per Protocol Population is not defined in this study.

207660

## 10.2. Appendix 2: Schedule of Activities

## 10.2.1. Protocol Defined Schedule of Events

| | Screening <sup>a</sup> | label phase | | | | | | | Open-label phase If a participant meets the eligibility at V5/QRV, the participant will move forward to the next treatment phase | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Pa | art 1 | | Eligibility<br>evaluation <sup>b</sup> | Part 2/Part 3/ Part 4 | | | | | Eligibility<br>evaluation <sup>b</sup> | |
| Visit | SV | V1<br>(Day<br>1) | V2 | V3 | V4 | V5 °<br>(Eligibility<br>evaluation) | QRV | V1 | V2 | V3 | V4 | V5 d<br>(Eligibility<br>evaluation) | QRV | Final<br>Visit |
| Time from initial injection (Day 1) (Weeks) | _ | 0 | 2 | 4 | 6 | 12 | Allowable Week 16 to 36e | _ | _ | _ | _ | _ | Allowable Week 24 to 36 e | 48/<br>Withdrawal |
| Time from injection day<br>in each treatment phase<br>(Weeks) | _ | 0 | 2 | 4 | 6 | 12 | 16/ 20/ 24/ 28/<br>32/ 36 | 0 | 2 | 4 | 6 | 12 | 16/ 20/ 24 | - |
| Acceptable visit windows (days) | | _ | ±4 | ±4 | ±4 | +4 <sup>f</sup> | ±14 <sup>g</sup> | (+4) <sup>v</sup> | ±4 | ±4 | ±4 | +4 <sup>f</sup> | ±14 <sup>g</sup> | ±4 |
| Written informed consent | X h | | | | | | | | | | | | | |
| Randomization | | X i | | | | | | | | | | | | |
| Injections | | X | | | | | | X | | | | | | |
| Evaluation of eligibility | | | | | | X | X | | | | | X | X | |
| Inclusion/exclusion criteria j | X | X i | | | | | | | | | | | | |
| Participant demography | X | | | | | | | | | | | | | |
| MAS <sup>k</sup> | X | X i | X | X | X | X | X | X i,t | X | X | X | X | X | X |
| NRS <sup>1</sup> | | X i | X | X | X | X | | X i,t | X | X | X | X | | (X) r |
| DAS | | $X^{i}$ | X | X | X | X | | $X^{i,t}$ | X | X | X | X | | (X) r |
| CGI by a investigator | | | X | X | X | X | | | X | X | X | X | | (X) r |
| CGI by a patient | | | X | X | X | X | | | X | X | X | X | | (X) r |
| Time to patient-reported onset of spasticity symptom relief | | | X | | | | | | X | | | | | |
| Patient-reported benefit of injection | | | | X | X | X | | | | X | X | X | | (X) <sup>r</sup> |
| Physical examination | X | | | | | | | | | | | | | |

207660

| | Screening <sup>a</sup> | label phase | | | | | | Open-label phase If a participant meets the eligibility at V5/QRV, the participant will move forward to the next treatment phase | | | | | | Completion visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Pa | art 1 | | Eligibility<br>evaluation <sup>b</sup> | Part 2/Part 3/ Part 4 Eligibility evaluation b | | | | Eligibility<br>evaluation <sup>b</sup> | | |
| Visit | SV | V1<br>(Day<br>1) | V2 | V3 | V4 | V5 °<br>(Eligibility<br>evaluation) | QRV | V1 | V2 | V3 | V4 | V5 <sup>d</sup><br>(Eligibility<br>evaluation) | QRV | Final<br>Visit |
| (complete version) | | | | | | | | | | | | | | |
| Physical examination (simplified version) | | X i | | | | X | | X i,t | | | | X | | X |
| Medical history | X | X i | | | | | | | | | | | | |
| Vital signs m | X | Xi | | | | X | | $X^{i,t}$ | | | | X | | X |
| Height | X | | | | | | | | | | | | | |
| Body weight | X | | | | | X <sup>u</sup> | X <sup>u</sup> | | | | | X <sup>u</sup> | X <sup>u</sup> | |
| Pulmonary function test | X | X | | | | X | X <sup>u</sup> | | | | | X | X <sup>u</sup> | X |
| Electrocardiogram | X | | | | | X <sup>u</sup> | X <sup>u</sup> | | | | | X <sup>u</sup> | X <sup>u</sup> | |
| Pregnancy test n | X | X i | | | | X <sup>u</sup> | X <sup>u</sup> | | | | | X <sup>s, u</sup> | X <sup>u</sup> | X |
| Laboratory test o | X | | | | | X | | | | | | X | | X |
| Adverse events p | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant medications/therapies | X | X i | X | X | X | X | X | X | X | X | X | X | X | X |
| Testing for neutralising antibodies q | X | | | | | X | | | | | | | | X |

- a. Test items for screening must be performed from 4 weeks to 1 weeks before Day 1 visit (±3 days).
- b. Eligibility evaluation (Qualification for Retreatment Visit: QRV) will be performed at V5 as a starting point if a participant does not meet the criteria only. The evaluation is performed at a 4-week interval, V5 as a starting point, The QRV when a participant meets the criteria will be a same day as the injection in the next treatment period.
- c. If a participant is evaluated to meet the eligibility for the injection in the blind phase at V5, the participant will move forward to Part 2 in the open-label phase (Namely, V5 in Part 1 and V1 in Part 2 is a same day). If the participant does not meet the eligibility, QRV will be performed 4 weeks later, at V5 as s starting point.
- d. If a participant is evaluated to meet the eligibility at V5 in the open-label phase, the participant will move forward to the next treatment phase (V5 and V1 in the next treatment phase is a same day). If the participant does not meet the eligibility, QRV is performed 4 weeks later, V5 as a starting point. If V5 in each treatment phase is at Week 48 after initial injection, V5 will be considered to be completion visit (FV). However, for the testing items, pre-scheduled tests at

207660

V5 and neutralizing antibody tests will be performed. If V5 in Parts 2 and 3 is performed at Week 36 or later, after completion of V5, completion visit will be performed at Week 48.

- e. QRV is allowable to perform from initial injection to Week 36. Eligibility evaluation (QRV) will not be performed after Week 36.
- f. V5 must be performed at least 84 days after V1.
- g. The acceptable visit windows will be -14 to +4 days if QRV is performed at Week 36.
- h. Must be performed earlier than any other procedures
- i. Must be performed before injection of the product
- j. For inclusion/exclusion criteria, the items to be observed are different between screening phase and Day 1. For details, refer to Protocol Section 6.1 and Section 6.2.
- k. For MAS evaluation, the items to be evaluated differ depending on the treatment phase. For details, refer to Protocol Section 9.1.1.1.
- 1. MAS evaluation will be followed by NRS evaluation. For NRS evaluation, items to be evaluated differ. For details, refer to Protocol Section 9.1.1.2.
- m. Body temperature, heart rate, and blood pressure will be measured as vital signs.
- n. Women of childbearing potential will be only performed. Serum hCG pregnancy test must be performed at screening, and urine hCG pregnancy test after randomization. The tests can be performed beyond the protocol specifications if an investigator considers to be necessary.
- o. For laboratory test items, refer to Protocol Section 12.2. Attachment 2. Fasting is not required for blood collection.
- p. Adverse events and serious adverse events collection period will be from the initial injection day (Day 1) to completion visit (FV).
- q. Neutralizing antibody testing is performed 3 times in each participant. The first test will be performed in screening phase, the second is at V5 in the blind phase, and the third is at completion visit.
- r. A participant who withdraws the study before 12 weeks after last injection will be performed.
- s. Perform if V5 in each treatment phase is at Week 48 after initial injection
- t. Not necessary to perform doubly as V1 assessment if the same assessment is performed at V5 or QRV. If V1 assessment or retreatment cannot be performed on the same day as V5 or QRV, MAS assessment should be performed again on the day of visit for the V1 assessment.
- u. Evaluation of retreatment is performed only when the dosing conditions (1 to 5) of retreatment evaluation are met. If V1 assessment or retreatment cannot be performed on the same day as V5 or QRV, body weight, pulmonary function test, electrocardiogram, and pregnancy test should not be performed again on the day of visit for V1 assessment.
- v. V1 assessment in Part 2 or subsequent parts should be performed as a rule on the same day as V5 or QRS (when eligibility was confirmed) of the previous part. If this is not possible, the V1 assessment may be performed on another day but within the acceptable visit window.

207660

## 10.3. Appendix 3: Assessment Windows

## 10.3.1. Definitions of Assessment Windows for Efficacy Analyses (only Final Visit and Withdraw Visit, and only Final Analyses)

If the Visit 5 in last treatment cycle coincides with Final Visit (e.g., Visit 5 in 3rd treatment cycle is achieved on Week 48 from the initial dose), the efficacy data will be entered as Final Visit, not the last visit in the treatment cycle. However, actually the data at the last visit is not missing. Therefore, in the following cases, the Final Visit data will be treated as the Visit 5 in the last treatment cycle for the efficacy analyses.

Where the participant (except for the withdrawn from study) who was qualified for retreatment:

- At Week 12 in Blind Phase, 2nd and 3rd Open Label Phase
- At Week 12 in Blind Phase and at Week 24 in 2nd Open Label Phase.
- At Week 16 in Blind Phase and at Week 20 in 2nd Open Label Phase.
- At Week 20 in Blind Phase and at Week 16 in 2nd Open Label Phase.
- At Week 24 in Blind Phase and at Week 12 in 2nd Open Label Phase.
- At Week 36 in Blind Phase.

207660

## 10.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

## 10.4.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|-------------|--------------------------------------------------------------|
| Prior | "Taken prior to study?" is marked "Yes" on eCRF OR |
| | Medication Start Date < First Study Treatment Date <b>OR</b> |
| | Medication Start Date is missing. |
| Concomitant | "Ongoing medication?" is marked "Yes" or missing on eCRF OR |
| | Medication End Date ≥ First Study Treatment Date <b>OR</b> |
| | Medication End Date is missing |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

## 10.4.2. Study Phases for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | • First Study Treatment Date ≤ AE Start Date ≤ Final Visit Date/Early Withdrawal Date |
| Blind phase (until second dose) | <ul> <li>First Study Treatment Date ≤ AE Start Date ≤ Second Study Treatment Date AND AE Start Time &lt; Second Study Treatment Time IF AE Start Time is collected</li> <li>First Study Treatment Date ≤ AE Start Date &lt; Second Study Treatment Date IF AE Start Time is not collect.</li> </ul> |
| Blind phase (within 84 days) | • First Study Treatment Date ≤ AE Start Date ≤ First Study Treatment Date + 83 days |
| Open-Label<br>Phase (2nd<br>Treatment) | <ul> <li>Second Study Treatment Date ≤ AE Start Date ≤ Third Study Treatment Date</li> <li>AND Second Study Treatment Time ≤ AE Start Time &lt; Third Study Treatment</li> <li>Time IF AE Start Time is collected</li> </ul> |
| | <ul> <li>Second Study Treatment Date ≤ AE Start Date &lt; Third Study Treatment Date IF AE Start Time is not collected</li> </ul> |
| Open-Label<br>Phase (3rd<br>Treatment) | <ul> <li>Third Study Treatment Date ≤ AE Start Date ≤ Fourth Study Treatment Date AND Third Study Time ≤ AE Start Time &lt; Fourth Study Treatment Time IF AE Start <p>Time is collected </p></li> </ul> |
| | Third Study Treatment Date ≤ AE Start Date < Fourth Study Treatment Date IF AE Start Time is not collected |
| Open-Label<br>Phase (4th<br>Treatment) | <ul> <li>Fourth Study Treatment Date ≤ AE Start Date ≤ Final Visit Date AND Fourth Study Time ≤ AE Start Time IF AE Start Time is collected</li> <li>Fourth Study Treatment Date ≤ AE Start Date ≤ Final Visit Date IF AE Start Time</li> </ul> |
| Drug related | <ul> <li>is not collected</li> <li>If relationship to Study treatment(GSK1358820/Placebo) is marked 'YES' on CRF OR value is missing.</li> </ul> |

207660

## 10.4.2.1. Definition of Adverse Events of Special Interest

AEs of Special Interest are defined in the Appendix 13. If a Preferred Term of AE is included in the list of PTs of the specific AESI, that AE will be considered as AESI. See the details in the Appendix 13.

207660

## 10.5. Appendix 5: Data Display Standards & Handling Conventions

#### 10.5.1. Reporting Process

| Software | Software |
|---|---|
| The currently supply | The currently supported versions of SAS software will be used. |
| Reporting Area | Reporting Area |
| HARP Server | : US1SALX00259.corpnet2.com |
| HARP Compound | : arenv\arprod\gsk1358820\mid207660 |
| Analysis Datasets | Analysis Datasets |
| Analysis datasets will be created according to Legacy GSK A&R dataset standards. | |
| Generation of RTF Files | |
| RTF files will not b | e generated. |

#### 10.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:
  - https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include participant level listings in the main body of the GSK Clinical Study Report. All participant level listings should be located in the modular appendices as ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

## Planned and Actual Time

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.

207660

| Unscheduled Visits | |
|---|---|
| <ul> <li>Unscheduled visits</li> </ul> | Unscheduled visits will not be included in summary tables and/or figures. |
| All unscheduled vi | sits will be included in listings. |
| Descriptive Summary | Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| | For continuous efficacy endpoints, 95%Confidence Interval will be calculated based on t-distribution. |
| Categorical Data | N, n, frequency, % |
| Time to event data | The number of events and censored case. |
| | 25 <sup>th</sup> and 75 <sup>th</sup> percentiles survival time. |
| | Median survival time with the associated 95% Cls. |
| | 95%Cls will be calculated based on Brookmeyer and Crowley method using log-log function as a g-transformation. (This method can be performed using Proc LIFETEST with no special statement or option (SAS 9.4)) |
| Graphical Displays | |
| Refer to IDSL State | Refer to IDSL Statistical Principals 7.01 to 7.13. |

207660

#### 10.6. Appendix 6: Derived and Transformed Data

#### 10.6.1. General

#### **Study Day**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
- Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

## 10.6.2. Study Population

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follow:
  - o Any participant with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Age will be calculated based on year of the Screening visit as an Age reference date.

#### Age Group

- The following category will be used for Summary of Demography.
  - Age  $\leq$  18 (years)
  - o 19 < Age < 65
  - $\circ$  65  $\leq$  Age

#### Age Category

- The following category will be used for Summary of Age Ranges.
  - In utero
  - Preterm newborn infants (gestational age <37 weeks)</li>
  - Newborns (0-27 days)
  - o Infants and toddlers (28 days-23 months)
  - Children (2-11 years)
  - Adolescents (12-17 years)
  - Adult (18-64 years)
  - >=65-84 years
  - >=85 years

#### **Extent of Exposure**

- The total of dosage per treatment cycle will be calculated based on the formula:
  - Total of Dosage per treatment cycle = Sum of (Dosage in each Muscle Region)
- The subtotal of dosage in each joint per treatment cycle will be calculated based on the formula:
   Subtotal of Dosage in the joint per treatment cycle = Sum of (Dosage in each Muscle Region of the Joint)
- Example

Subtotal of Dosage in Elbow = Sum of (Dosage in Biceps brachii, Brachalis and Brachioradialis)

207660

## 10.6.3. Efficacy

#### **Time to Event Data**

#### Time to Qualification for Retreatment

• This time to event data will be derived based on the following formula:

## Time to Event (Days) = Date When a Participant Meets the Criteria for Retreatment – Study Treatment Start Date (Days)

• If a participant is withdrawn from this study, the participant will be regarded as censoring and censored date will be a withdrawal date.

#### Time to Patient Reported Onset of Spasticity Symptom Relief

• This time to event data will be derived based on the following formula:

## Time to Event (Days) = Onset Date of the Spasticity Symptom Relief – Study Treatment Start Date (Days)

If a participant is withdrawn from this study, the participant will be regarded as censoring and censored date will be a withdrawal date.

207660

## 10.7. Appendix 7: Reporting Standards for Missing Data

## 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Participant study completion (i.e. as specified in the protocol) was defined as those who completed all the study procedures, including a completion visit. |
| | Withdrawn participants were not replaced in the study. |
| | <ul> <li>All available data from participants who were withdrawn from the study will be listed<br/>and all available planned data will be included in summary tables and figures, unless<br/>otherwise specified.</li> </ul> |
| | Withdrawal visits will be slotted as per Appendix 3: Assessment Windows or will be summarised as withdrawal visits. |

## 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in participant listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Responder of MAS | If MAS score is missing at the corresponding visit, the participant will be regarded as those who are a non-responder (i.e. non-responder imputation). |

## 10.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in participant listing displays. |
| Concomitant<br>Medications<br>and Surgery | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

207660

## 10.8. Appendix 8: Values of Potential Clinical Importance

This is not applicable to this study.

207660

## 10.9. Appendix 9: Population Pharmacokinetic (PopPK) Analyses

This is not applicable to this study.

207660

# 10.10. Appendix 10: Pharmacokinetic / Pharmacodynamic Analyses

This is not applicable to this study.

207660

#### **Appendix 11: Abbreviations & Trade Marks** 10.11.

## 10.11.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | |
| DOB | Database Release Date of Birth |
| DP | Decimal Places |
| eCRF | |
| | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| MMRM | Mixed Model for Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |

207660

| Abbreviation | Description |
|--------------|------------------------------|
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

## 10.11.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| NONE |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |

207660

## 10.12. Appendix 12: List of Data Displays

## 10.12.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|--------------|-------------|
| Study Population | 1.1 to 1.22 | |
| Efficacy | 2.1 to 2.53 | 2.1 to 2.55 |
| Safety | 3.1 to 3.138 | 3.1 to 3.2 |
| Section | Listings | |
| ICH Listings | 1 to 78 | |

## 10.12.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 10.12.3. Deliverables

| Delivery | Description |
|----------|------------------------------------------------|
| IA SAC | Interim Analysis Statistical Analysis Complete |
| SAC | Final Statistical Analysis Complete |

207660

## 10.12.4. Study Population Tables

## 10.12.4.1. Interim Analyses

| Study I | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Particip | oant Dispositio | n | | | |
| 1.01. | ITT1 | ES1 | Summary of Participant Disposition for the Participant Conclusion Record (Week 24) | ICH E3, FDAAA, EudraCT Participant disposition at Week 24. Include total arm (240 U + 400 U) | IA SAC |
| 1.02. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | IA SAC |
| 1.03. | Enrolled | NS1 | Summary of Number of Participant by Site ID | EudraCT/Clinical Operations | IA SAC |
| Protoc | ol Deviation | | | | |
| 1.04. | ITT1 | DV1 | Summary of Important Protocol Deviations | ICH E3<br>Include total arm (240 U + 400 U) | IA SAC |
| Popula | tion Analysed | | | | |
| 1.05. | Screened | SP1 | Summary of Study Populations | IDSL | IA SAC |
| Demog | raphic and Bas | eline Characteris | tics | | • |
| 1.06. | ITT1 | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT<br>Include total arm (240 U + 400 U) | IA SAC |
| 1.07. | Enrolled | DM11 | Summary of Age Ranges | EudraCT | IA SAC |
| 1.08. | ITT1 | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | IA SAC |

207660

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 1.09. | ITT1 | POP_T1 | Summary of Baseline Efficacy Parameters | <ul> <li>MAS scores in finger, thumb, wrist and elbow</li> <li>Randomization Strata</li> <li>Numeric Rating Scale for pain</li> <li>Disability Assessment Scale</li> <li>Include total arm (240 U + 400 U)</li> </ul> | IA SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 1.10. | ITT1 | CM1 | Summary of Prior Medications | Include total arm (240 U + 400 U) | IA SAC |
| 1.11. | ITT1 | CM1 | Summary of Concomitant Medications | ICH E3<br>Include total arm (240 U + 400 U) | IA SAC |
| 1.12. | ITT1 | POP_T2 | Summary of Rehabilitation | Include total arm (240 U + 400 U) | IA SAC |
| 1.13. | ITT1 | SAFE_T4 | Summary of Actual Dosage in Exposed Muscle Region by Treatment Cycle and Muscle Region. | | IA SAC |
| 1.14. | ITT1 | SAFE_T4 | Summary of Actual Dosage in Exposed Joint by Treatment Cycle and Joint | | IA SAC |

207660

## 10.12.4.2. Final Analyses

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Particip | ant Disposition | n | | | |
| 1.15. | ITT1 | ES1 | Summary of Participant Disposition for the Participant Conclusion Record | ICH E3, FDAAA, EudraCT<br>Include total arm (240 U + 400 U) | SAC |
| Protoc | ol Deviation | | | | |
| 1.16. | ITT1 | DV1 | Summary of Important Protocol Deviations | ICH E3<br>Include total arm (240 U + 400 U) | SAC |
| Popula | tion Analysed | | | | |
| 1.17. | Screened | SP1 | Summary of Study Populations | IDSL | SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 1.18. | ITT1 | CM1 | Summary of Prior Medications | Include total arm (240 U + 400 U) | SAC |
| 1.19. | ITT1 | CM1 | Summary of Concomitant Medications | ICH E3<br>Include total arm (240 U + 400 U) | SAC |
| 1.20. | ITT1 | POP_T2 | Summary of Rehabilitation | Include total arm (240 U + 400 U) | SAC |
| Actual | Actual dose | | | | |
| 1.21. | ITT1 | SAFE_T4 | Summary of Actual Dosage in Exposed Muscle Region by Treatment Cycle and Muscle Region. | | SAC |
| 1.22. | ITT1 | SAFE_T4 | Summary of Actual Dosage in Exposed Joint by Treatment Cycle and Joint | | SAC |

207660

## 10.12.5. Efficacy Tables

## 10.12.5.1. Interim Analyses

| Efficacy | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| MAS | | | | | |
| 2.01. | ITT1 | EFF_T1 | Summary of MAS score in Blind Phase | <ul><li>Values and change from baseline</li><li>Summarize data up to Visit 5</li></ul> | IA SAC |
| 2.02. | ITT1 | EFF_T2 | Summary of the Results of Mixed Models for Repeated<br>Measures of Change from Baseline in MAS scores in Blind<br>Phase | Analyse data up to Visit 5 | IA SAC |
| 2.03. | ITT1 | EFF_T3 | Summary of Responder rate of MAS score at Week 6 in Blind Phase | Including subgroup analyses | IA SAC |
| 2.04. | ITT1 | EFF_T4 | Summary of Responder rate of MAS score in Blind Phase | Summarize data up to Visit 5<br>Include Mantel Haenszel estimators | IA SAC |
| 2.05. | ITT2 | EFF_T1 | Summary of MAS score in Open Label Phase (2nd Treatment) | <ul> <li>Values and change from baseline</li> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| 2.06. | ITT2 | EFF_T5 | Summary of Responder rate of MAS score in Open Label Phase (2nd Treatment) | <ul> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |

207660

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| DAS | | | | | |
| 2.07. | ITT1 | EFF_T1 | Summary of Main Assessment Parameter and All Items of DAS in Blind Phase | <ul><li>Values and change from baseline</li><li>Summarize data up to Visit 5</li></ul> | IA SAC |
| 2.08. | ITT1 | EFF_T2 | Summary of the Results of Mixed Models for Repeated<br>Measures of Change from Baseline in Main Assessment<br>Parameter of DAS in Blind Phase | Analyse data up to Visit 5 | IA SAC |
| 2.09. | ITT2 | EFF_T1 | Summary of Main Assessment Parameter and All Items of DAS in Open Label Phase (2nd Treatment) | <ul> <li>Values and change from baseline</li> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| NRS for | pain | | | | |
| 2.10. | ITT1 | EFF_T1 | Summary of NRS for pain in Blind Phase | <ul><li>Values and change from baseline</li><li>Summarize data up to Visit 5</li></ul> | IA SAC |
| 2.11. | ITT2 | EFF_T1 | Summary of NRS for pain in Open Label Phase (2nd Treatment) | <ul> <li>Values in each joint and change from baseline in only elbow.</li> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |

207660

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| CGI of functional disability | | | | | |
| 2.12. | ITT1 | EFF_T1 | Summary of CGI of functional disability by an investigator in Blind Phase | <ul><li> Values only</li><li> Summarize data up to Visit 5</li></ul> | IA SAC |
| 2.13. | ITT2 | EFF_T1 | Summary of CGI of functional disability by an investigator in Open Label Phase (2nd Treatment) | <ul> <li>Values only</li> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| 2.14. | ITT1 | EFF_T1 | Summary of CGI of functional disability by a patient in Blind Phase | Values only Summarize data up to Visit 5 | IA SAC |
| 2.15. | ITT2 | EFF_T1 | Summary of CGI of functional disability by a patient in Open Label Phase (2nd Treatment) | <ul> <li>Values only</li> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| Patient- | Reported Bene | efit of Injection | | | |
| 2.16. | ITT1 | EFF_T5 | Summary of Patient-Reported Benefit of Injection in Blind Phase | Summarize data up to Visit 5 | IA SAC |
| 2.17. | ITT2 | EFF_T5 | Summary of Patient-Reported Benefit of Injection in Open Label Phase (2nd Treatment) | <ul> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| Time to | Patient-Repor | ted Onset of Spas | sticity Symptom Relief | <u>, </u> | |
| 2.18. | ITT1 | EFF_T6 | Summary of Time to Patient-Reported Onset of Spasticity Symptom Relief | | IA SAC |
| 2.19. | ITT1 | EFF_T7 | Summary of Survival Analyses Results of Time to Patient-<br>Reported Onset of Spasticity Symptom Relief in Blind Phase | Survival function estimates will<br>be summarized | IA SAC |

207660

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.20. | ITT2 | EFF_T7 | Summary of Survival Analyses Results of Time to Patient-<br>Reported Onset of Spasticity Symptom Relief in Open Label<br>Phase (2nd Treatment) | Survival function estimates will<br>be summarized | IA SAC |
| | | | | • Three treatment arms (240, 400 and 240 + 400U) | |
| Time to | Time to Qualification for Retreatment | | | | |
| 2.21. | ITT1 | EFF_T8 | Summary of Events in Which a Participant Meets the Criteria for Retreatment | | IA SAC |
| 2.22. | ITT1 | EFF_T6 | Summary of Time to Qualification for Retreatment | | IA SAC |
| 2.23. | ITT1 | EFF_T7 | Summary of Survival Analyses Results of Time to Qualification for Retreatment in Blind Phase | <ul> <li>Survival function estimates will<br/>be summarized</li> <li>Two treatment arms (240 and<br/>400U)</li> </ul> | IA SAC |

## 10.12.5.2. Final Analyses

| Efficacy: Tables | | | | | | | | | |
|---|---|---|---|---|---|--|--|--|--|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable | | | | |
| MAS | | | | | | | | | |
| 2.24. | ITT2 | EFF_T1 | Summary of MAS score in Open Label Phase (2nd Treatment) | <ul> <li>Values and change from baseline</li> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | SAC | | | | |
| 2.25. | ITT3 | EFF_T1 | Summary of MAS score in Open Label Phase (3rd Treatment) | | SAC | | | | |
| 2.26. | ITT4 | EFF_T1 | Summary of MAS score in Open Label Phase (4th Treatment) | | SAC | | | | |
| Efficacy | Efficacy: Tables | | | | | | | |
|---|---|---|---|---|---|--|--|--|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable | | | |
| 2.27. | ITT2 | EFF_T5 | Summary of Responder rate of MAS score in Open Label Phase (2nd Treatment) | <ul> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | SAC | | | |
| 2.28. | ITT3 | EFF_T5 | Summary of Responder rate of MAS score in Open Label Phase (3rd Treatment) | | SAC | | | |
| 2.29. | ITT4 | EFF_T5 | Summary of Responder rate of Mas Score in Open Label Phase (4th Treatment) | | SAC | | | |

| Efficacy | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| DAS | • | | | | |
| 2.30. | ITT2 | EFF_T1 | Summary of Main Assessment Parameter and All Items of DAS in Open Label Phase (2nd Treatment) | Values and change from baseline | SAC |
| 2.31. | ITT3 | EFF_T1 | Summary of Main Assessment Parameter and All Items of DAS in Open Label Phase (3rd Treatment) | Summarize data up to Visit 5 | SAC |
| 2.32. | ITT4 | EFF_T1 | Summary of Main Assessment Parameter and All Items of DAS in Open Label Phase (4th Treatment) | • Three treatment arms (240, 400 and 240 + 400U) | SAC |
| NRS for | pain | | | | |
| 2.33. | ITT2 | EFF_T1 | Summary of NRS for pain in Open Label Phase (2nd Treatment) | Values in each joint and | SAC |
| 2.34. | ITT3 | EFF_T1 | Summary of NRS for pain in Open Label Phase (3rd Treatment) | change from baseline in only elbow. | SAC |
| 2.35. | ITT4 | EFF_T1 | Summary of NRS for pain in Open Label Phase (4th Treatment) | <ul> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | SAC |
| CGI of fo | unctional disa | bility | | | |
| 2.36. | ITT2 | EFF_T1 | Summary of CGI of functional disability by an investigator in Open Label Phase (2nd Treatment) | Values only | SAC |
| 2.37. | ITT3 | EFF_T1 | Summary of CGI of functional disability by an investigator in Open Label Phase (3rd Treatment) | <ul> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240,</li> </ul> | SAC |
| 2.38. | ITT4 | EFF_T1 | Summary of CGI of functional disability by an investigator in Open Label Phase (4th Treatment) | 400 and 240 + 400U) | SAC |
| 2.39. | ITT2 | EFF_T1 | Summary of CGI of functional disability by a patient in Open Label Phase (2nd Treatment) | <ul><li>Values only</li><li>Summarize data up to Visit 5</li><li>Three treatment arms (240,</li></ul> | SAC |
| 2.40. | ITT3 | EFF_T1 | Summary of CGI of functional disability by a patient in Open Label Phase (3rd Treatment) | | SAC |

| Efficacy | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.41. | ITT4 | EFF_T1 | Summary of CGI of functional disability by a patient in Open Label Phase (4th Treatment) | 400 and 240 + 400U) | SAC |
| Patient-I | Reported Bene | efit of Injection | | | |
| 2.42. | ITT2 | EFF_T5 | Summary of Patient-Reported Benefit of Injection in Open Label Phase (2nd Treatment) | Comments data and North 5 | SAC |
| 2.43. | ITT3 | EFF_T5 | Summary of Patient-Reported Benefit of Injection in Open Label Phase (3rd Treatment) | <ul> <li>Summarize data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | SAC |
| 2.44. | ITT4 | EFF_T5 | Summary of Patient-Reported Benefit of Injection in Open Label Phase (4th Treatment) | 400 and 240 + 4000) | SAC |
| Time to | Patient-Repor | ted Onset of Spas | ticity Symptom Relief | | |
| 2.45. | ITT1 | EFF_T6 | Summary of Time to Patient-Reported Onset of Spasticity Symptom Relief | | SAC |
| 2.46. | ITT2 | EFF_T7 | Summary of Survival Analyses Results of Time to Patient-<br>Reported Onset of Spasticity Symptom Relief in Open Label<br>Phase (2nd Treatment) | | SAC |
| 2.47. | ITT3 | EFF_T7 | Summary of Survival Analyses Results of Time to Patient-<br>Reported Onset of Spasticity Symptom Relief in Open Label<br>Phase (3rd Treatment) | Survival function estimates will be summarized Three treatment arms (240, 400 and 240 + 400 ll) | SAC |
| 2.48. | ITT4 | EFF_T7 | Summary of Survival Analyses Results of Time to Patient-<br>Reported Onset of Spasticity Symptom Relief in Open Label<br>Phase (4th Treatment) | - 400 and 240 + 400U) | SAC |
| Time to | Qualification f | or Retreatment | | | |
| 2.49. | ITT1 | EFF_T8 | Summary of Events in Which a Participant Meets the Criteria for Retreatment | | SAC |
| 2.50. | ITT1 | EFF_T6 | Summary of Time to Qualification for Retreatment | | SAC |

| Efficacy | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.51. | ITT1 | EFF_T7 | Summary of Survival Analyses Results of Time to Qualification for Retreatment in Blind Phase | Survival function estimates will be summarized Two treatment arms (240 and 400U) | SAC |
| 2.52. | ITT2 | EFF_T7 | Summary of Survival Analyses Results of Time to Qualification for Retreatment in Open Label Phase (2nd Treatment) | Survival function estimates will<br>be summarized | SAC |
| 2.53. | ITT3 | EFF_T7 | Summary of Survival Analyses Results of Time to Qualification for Retreatment in Open Label Phase (3rd Treatment) | • Three treatment arms (240, 400 and 240 + 400U) | SAC |

207660

# 10.12.6. Efficacy Figures

## 10.12.6.1. Interim Analyses

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| MAS | | | | | |
| 2.01. | ITT1 | EFF_F1 | Plot of Mean (95%CI) MAS score Profiles in Blind Phase | <ul> <li>Plot data up to Visit 5</li> <li>Two treatment arms (240 and 400U)</li> </ul> | IA SAC |
| 2.02. | ITT2 | EFF_F1 | Plot of Mean (95%CI) MAS score Profiles in Open Label Phase (2nd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| 2.03. | ITT1 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in MAS score<br>Profiles in Blind Phase | <ul><li>Plot data up to Visit 5</li><li>Two treatment arms (240 and 400U)</li></ul> | IA SAC |
| 2.04. | ITT2 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in MAS score<br>Profiles in Open Label Phase (2nd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| 2.05. | ITT1 | EFF_F2 | Plot of Responder rate of MAS score by Visit in Blind Phase | <ul><li>Plot data up to Visit 5</li><li>Two treatment arms (240 and 400U)</li></ul> | IA SAC |
| 2.06. | ITT2 | EFF_F2 | Plot of Responder rate of MAS score by Visit in Open Label Phase (2nd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| DAS | • | | | | |
| 2.07. | ITT1 | EFF_F1 | Plot of Mean (95%CI) DAS score (Main Assessment Parameter)<br>Profiles in Blind Phase | <ul><li>Plot data up to Visit 5</li><li>Two treatment arms (240 and 400U)</li></ul> | IA SAC |
| 2.08. | ITT2 | EFF_F1 | Plot of Mean (95%CI) DAS score (Main Assessment Parameter)<br>Profiles in Open Label Phase (2nd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| 2.09. | ITT1 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in DAS score (Main Assessment Parameter) Profiles in Blind Phase | <ul><li>Plot data up to Visit 5</li><li>Two treatment arms (240 and 400U)</li></ul> | IA SAC |
| 2.10. | ITT2 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in DAS score (Main Assessment Parameter) Profiles in Open Label Phase (2nd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| 2.11. | ITT1 | EFF_F1 | Plot of Mean (95%CI) DAS score Profiles in Blind Phase | <ul> <li>Plot data up to Visit 5</li> <li>Create plots by component of DAS score</li> <li>Two treatment arms (240 and 400U)</li> </ul> | IA SAC |
| 2.12. | ITT2 | EFF_F1 | Plot of Mean (95%CI) DAS score Profiles in Open Label Phase (2nd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Create plots by component of<br/>DAS score</li> <li>Three treatment arms (240 and<br/>400U)</li> </ul> | IA SAC |

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.13. | ITT1 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in DAS score<br>Profiles in Blind Phase | <ul> <li>Plot data up to Visit 5</li> <li>Create plots by component of DAS score</li> <li>Two treatment arms (240 and 400U)</li> </ul> | IA SAC |
| 2.14. | ITT2 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in DAS score<br>Profiles in Open Label Phase (2nd Treatment) | Plot data up to Visit 5 Create plots by component of DAS score Three treatment arms (240 and 400U) | IA SAC |
| Numeri | c Rating Scale | for pain | | | |
| 2.15. | ITT1 | EFF_F1 | Plot of Mean (95%CI) NRS for pain Profiles in Blind Phase | <ul> <li>Plot data up to Visit 5</li> <li>Two treatment arms (240 U and 400U)</li> </ul> | IA SAC |
| 2.16. | ITT2 | EFF_F1 | Plot of Mean (95%CI) NRS for pain Profiles in Open Label<br>Phase (2nd Treatment) | <ul> <li>Plot data of the elbow only up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | IA SAC |
| 2.17. | ITT1 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in NRS for pain Profiles in Blind Phase | <ul> <li>Plot data up to Visit 5</li> <li>Two treatment arms (240 U and 400U)</li> </ul> | IA SAC |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Clinica | Clinical Global Impression of Change of functional disability | | | | |
| 2.18. | ITT1 | EFF_F1 | Plot of Mean (95%CI) CGI of functional disability Profiles in Blind Phase | <ul><li>Plot data up to Visit 5</li><li>Two treatment arms (240 and 400 U)</li></ul> | IA SAC |
| 2.19. | ITT2 | EFF_F1 | Plot of Mean (95%CI) CGI of functional disability Profiles in Open Label Phase (2nd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400 U)</li> </ul> | IA SAC |
| Time to | Patient-Repor | ted Onset of Spas | ticity Symptom Relief | | |
| 2.20. | ITT1 | EFF_F3 | Kaplan Meier Plot of Time to Patient-Reported Onset of Spasticity Symptom Relief in Blind Phase | Two treatment arm (240 U and 400U) | IA SAC |
| 2.21. | ITT2 | EFF_F3 | Kaplan Meier Plot of Time to Patient-Reported Onset of Spasticity Symptom Relief in Open Label Phase (2nd Treatment) | Three treatment arms (240, 400, 240 + 400U) | IA SAC |
| Time to | Qualification f | for Retreatment | | | |
| 2.22. | ITT1 | EFF_F3 | Kaplan Meier Plot of Survival Function Estimates of Time to Qualification for Retreatment in Blind Phase | Two treatment arm (240 U, 400U) | IA SAC |

207660

# 10.12.6.2. Final Analyses

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| MAS | • | | | , | |
| 2.23. | ITT2 | EFF_F1 | Plot of Mean (95%CI) MAS score Profiles in Open Label Phase (2nd Treatment) | Plot data up to Visit 5 Three treatment arms (240, | SAC |
| 2.24. | ITT3 | EFF_F1 | Plot of Mean (95%CI) MAS score Profiles in Open Label Phase (3rd Treatment) | 400 and 240 + 400U) ` | SAC |
| 2.25. | ITT4 | EFF_F1 | Plot of Mean (95%CI) MAS score Profiles in Open Label Phase (4th Treatment) | | SAC |
| 2.26. | ITT2 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in MAS score<br>Profiles in Open Label Phase (2nd Treatment) | 51 | SAC |
| 2.27. | ITT3 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in MAS score<br>Profiles in Open Label Phase (3rd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Three treatment arms (240, 400 l)</li> </ul> | SAC |
| 2.28. | ITT4 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in MAS score<br>Profiles in Open Label Phase (4th Treatment) | 400 and 240 + 400U) | SAC |
| 2.29. | ITT2 | EFF_F2 | Plot of Responder rate of MAS score by Visit in Open Label Phase (2nd Treatment) | D1.1.1.1.1.1.1.1.1.1.1.1.1.1.1.1.1.1.1. | SAC |
| 2.30. | ITT3 | EFF_F2 | Plot of Responder rate of MAS score by Visit in Open Label Phase (3rd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Three treatment arms (240, 400 l)</li> </ul> | SAC |
| 2.31. | ITT4 | EFF_F2 | Plot of Responder rate of MAS score by Visit in Open Label Phase (4th Treatment) | 400 and 240 + 400U) | SAC |
| DAS | | | | | |
| 2.32. | ITT2 | EFF_F1 | Plot of Mean (95%CI) DAS score (Main Assessment Parameter)<br>Profiles in Open Label Phase (2nd Treatment) | Plot data up to Visit 5 | SAC |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 2.33. | ITT3 | EFF_F1 | Plot of Mean (95%CI) DAS score (Main Assessment Parameter)<br>Profiles in Open Label Phase (3rd Treatment) | • Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 2.34. | ITT4 | EFF_F1 | Plot of Mean (95%CI) DAS score (Main Assessment Parameter)<br>Profiles in Open Label Phase (4th Treatment) | | SAC |
| 2.35. | ITT2 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in DAS score (Main Assessment Parameter) Profiles in Open Label Phase (2nd Treatment) | | SAC |
| 2.36. | ITT3 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in DAS score (Main Assessment Parameter) Profiles in Open Label Phase (3rd Treatment) | <ul> <li>Plot data up to Visit 5</li> <li>Three treatment arms (240, 400 and 240 + 400U)</li> </ul> | SAC |
| 2.37. | ITT4 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in DAS score (Main Assessment Parameter) Profiles in Open Label Phase (4th Treatment) | 100 and 2 10 × 1000) | SAC |
| 2.38. | ITT2 | EFF_F1 | Plot of Mean (95%CI) DAS score Profiles in Open Label Phase (2nd Treatment) | Plot data up to Visit 5 | SAC |
| 2.39. | ITT3 | EFF_F1 | Plot of Mean (95%CI) DAS score Profiles in Open Label Phase (3rd Treatment) | Create plots by component of DAS score The state of the state of | SAC |
| 2.40. | ITT4 | EFF_F1 | Plot of Mean (95%CI) DAS score Profiles in Open Label Phase (4th Treatment) | Three treatment arms (240 and 400U) | SAC |
| 2.41. | ITT2 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in DAS score<br>Profiles in Open Label Phase (2nd Treatment) | Plot data up to Visit 5 Create plots by component of DAS score Three treatment arms (240 and 400U) | SAC |
| 2.42. | ITT3 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in DAS score<br>Profiles in Open Label Phase (3rd Treatment) | | SAC |
| 2.43. | ITT4 | EFF_F1 | Plot of Mean (95%CI) Change from Baseline in DAS score<br>Profiles in Open Label Phase (4th Treatment) | | SAC |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Numeri | Numeric Rating Scale for pain | | | | |
| 2.44. | ITT2 | EFF_F1 | Plot of Mean (95%CI) NRS for pain Profiles in Open Label<br>Phase (2nd Treatment) | Plot data of the elbow only up | SAC |
| 2.45. | ITT3 | EFF_F1 | Plot of Mean (95%CI) NRS for pain Profiles in Open Label Phase (3rd Treatment) | to Visit 5 Three treatment arms (240, | SAC |
| 2.46. | ITT4 | EFF_F1 | Plot of Mean (95%CI) NRS for pain Profiles in Open Label<br>Phase (4th Treatment) | 400 and 240 + 400U) | SAC |
| Clinical | Global Impres | sion of Change of | f functional disability | | |
| 2.47. | ITT2 | EFF_F1 | Plot of Mean (95%CI) CGI of functional disability Profiles in Open Label Phase (2nd Treatment) | 51 | SAC |
| 2.48. | ITT3 | EFF_F1 | Plot of Mean (95%CI) CGI of functional disability Profiles in Open Label Phase (3rd Treatment) | Plot data up to Visit 5 Three treatment arms (240, | SAC |
| 2.49. | ITT4 | EFF_F1 | Plot of Mean (95%CI) CGI of functional disability Profiles in Open Label Phase (4th Treatment) | 400 and 240 + 400 U) | SAC |
| Time to | Patient-Repor | ted Onset of Spas | ticity Symptom Relief | | |
| 2.50. | ITT2 | EFF_F3 | Kaplan Meier Plot of Time to Patient-Reported Onset of Spasticity Symptom Relief in Open Label Phase (2nd Treatment) | | SAC |
| 2.51. | ITT3 | EFF_F3 | Kaplan Meier Plot of Time to Patient-Reported Onset of Spasticity Symptom Relief in Open Label Phase (3rd Treatment) | Three treatment arms (240, 400, 240 + 400U) | SAC |
| 2.52. | ITT4 | EFF_F3 | Kaplan Meier Plot of Time to Patient-Reported Onset of Spasticity Symptom Relief in Open Label Phase (4th Treatment) | | SAC |

| Efficacy: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Time to | Qualification 1 | for Retreatment | | | |
| 2.53. | ITT1 | EFF_F3 | Kaplan Meier Plot of Survival Function Estimates of Time to Qualification for Retreatment in Blind Phase | Two treatment arm (240 U, 400U) | SAC |
| 2.54. | ITT2 | EFF_F3 | Kaplan Meier Plot of Survival Function Estimates of Time to Qualification for Retreatment in Open Label Phase (2nd Treatment) | Three treatment arm (240, 400, 240 + 400U) | SAC |
| 2.55. | ITT3 | EFF_F3 | Kaplan Meier Plot of Survival Function Estimates of Time to Qualification for Retreatment in Open Label Phase (3rd Treatment) | | SAC |

207660

# 10.12.7. Safety Tables

# 10.12.7.1. Interim Analyses

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Adverse | e Events (AEs) | | | | |
| 3.01. | Safety 1 | AE1 | Summary of All Adverse Events until Week 24 visit by System<br>Organ Class and Preferred Term | ICH E3 Treatment Emergent Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.02. | Safety 1 | AE1 | Summary of All Adverse Events until Week 24 visit by System<br>Organ Class and Preferred Term in Blind Phase | Blind Phase (until second dose) See the Section 10.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.03. | Safety 1 | AE1 | Summary of All Adverse Events within 84 days from the initial dose by System Organ Class and Preferred Term in Blind Phase | Blind Phase (within 84 days) See the Section 10.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.04. | Safety 2 | AE1 | Summary of All Adverse Events until Week 24 visit by System Organ Class and Preferred Term in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.05. | Safety 1 | AE5A | Summary of All Adverse Events until Week 24 visit by Maximum Intensity by System Organ Class and Preferred Term | ICH E3 Treatment Emergent Use AE1 or AE1CP if Grade/Intensity not used; otherwise use AE5A/B (with a Total column across all grades/severities, which provides same detail as AE1) | IA SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.06. | Safety 1 | AE5A | Summary of All Adverse Events until Week 24 visit by Maximum Intensity by System Organ Class and Preferred Term in Blind Phase | Blind Phase (until second dose) See the Section 10.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.07. | Safety 1 | AE5A | Summary of All Adverse Events within 84 days from the initial dose by Maximum Intensity by System Organ Class and Preferred Term in Blind Phase | Blind Phase (within 84 days) See the Section 10.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.08. | Safety 2 | AE5A | Summary of All Adverse Events until Week 24 visit by Maximum Intensity by System Organ Class and Preferred Term in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.09. | Safety 1 | AE3 | Summary of Common (>=3%) Adverse Events until Week 24 visit by Overall Frequency | ICH E3 Treatment Emergent Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.10. | Safety 1 | AE3 | Summary of Common (>= 3%) Adverse Events within 84 days from the initial dose by Overall Frequency in Blind Phase (by Sex) | Three treatment arms (240, 400 and total) | IA SAC |
| 3.11. | Safety 1 | AE3 | Summary of Common (>= 3%) Adverse Events within 84 days from the initial dose by Overall Frequency in Blind Phase (by Age Group) | Three treatment arms (240, 400 and total) Age group (Age < 65 or Age >= 65) | IA SAC |
| 3.12. | Safety 1 | AE3 | Summary of Common (>=3%) Adverse Events until Week 24 visit by Overall Frequency in Blind Phase | Blind Phase (until second dose) See the Section 10.4.2. Two treatment arm (240 and 400U) | IA SAC |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.13. | Safety 1 | AE3 | Summary of Common (>=3%) Adverse Events within 84 days from the initial dose by Overall Frequency in Blind Phase | Blind Phase (within 84 days) See the Section 10.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.14. | Safety 2 | AE3 | Summary of Common (>=3%) Adverse Events until Week 24 visit by Overall Frequency in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.15. | Safety 1 | AE1 | Summary of All Drug-Related Adverse Events until Week 24 visit by System Organ Class and Preferred Term | ICH E3 Treatment Emergent Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.16. | Safety 1 | AE1 | Summary of All Drug-Related Adverse Events until Week 24 visit by System Organ Class and Preferred Term in Blind Phase | Blind Phase (until second dose) See the Section 10.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.17. | Safety 1 | AE1 | Summary of All Drug-Related Adverse Events within 84 days from the initial dose by System Organ Class and Preferred Term in Blind Phase | Blind Phase (within 84 days) See the Section 10.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.18. | Safety 2 | AE1 | Summary of All Drug-Related Adverse Events until Week 24 visit by System Organ Class and Preferred Term in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | IA SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.19. | Safety 1 | AE5A | Summary of All Drug-Related Adverse Events until Week 24 visit by System Organ Class and Preferred Term and Maximum Intensity | ICH E3 Treatment Emergent AE See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.20. | Safety 1 | AE5A | Summary of All Drug-Related Adverse Events until Week 24 visit by System Organ Class and Preferred Term and Maximum Intensity in Blind Phase | Blind Phase (until second dose) See the Section 10.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.21. | Safety 1 | AE5A | Summary of All Drug-Related Adverse Events within 84 days from the initial dose by System Organ Class and Preferred Term and Maximum Intensity in Blind Phase | Blind Phase (within 84 days) See the Section 10.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.22. | Safety 2 | AE5A | Summary of All Drug-Related Adverse Events until Week 24 visit by System Organ Class and Preferred Term and Maximum Intensity in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.23. | Safety 1 | AE15 | Summary of Common (>=5%) Non-serious Adverse Events until Week 24 visit by System Organ Class and Preferred Term (Number of Participant and Occurrences) | FDAAA, EudraCT Treatment Emergent AE See the Section 10.4.2 | IA SAC |
| Serious | s and Other Sig | nificant Adverse | Events | | |
| 3.24. | Safety 1 | SAFE_T1 | Summary of Adverse Events of Special Interest until Week 24 visit | Treatment Emergent AE See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | IA SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.25. | Safety 1 | SAFE_T1 | Summary of Adverse Events of Special Interest until Week 24 visit in Blind Phase | Blind Phase (until second dose) See the Section 10.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.26. | Safety 1 | SAFE_T1 | Summary of Adverse Events of Special Interest within 84 days from the initial dose in Blind Phase | Blind Phase (within 84 days) See the Section 10.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.27. | Safety 2 | SAFE_T1 | Summary of Adverse Events of Special Interest until Week 24 visit in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.28. | Safety 1 | AE1 | Summary of Non-Fatal Serious Adverse Events until Week 24 visit | Treatment Emergent AE See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.29. | Safety 1 | AE1 | Summary of Non-Fatal Serious Adverse Events until Week 24 visit in Blind Phase | Blind Phase (until second dose) See the Section 10.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.30. | Safety 1 | AE1 | Summary of Non-Fatal Serious Adverse Events within 84 days from the initial dose in Blind Phase | Blind Phase (within 84 days) See the Section 10.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.31. | Safety 2 | AE1 | Summary of Non-Fatal Serious Adverse Events until Week 24 visit in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | IA SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.32. | Safety 1 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events until Week 24 visit | Treatment Emergent AE See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.33. | Safety 1 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events until Week 24 visit in Blind Phase | Blind Phase (until second dose) See the Section 10.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.34. | Safety 1 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events within 84 days from the initial dose in Blind Phase | Blind Phase (within 84 days) See the Section 10.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.35. | Safety 2 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events until Week 24 visit in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.36. | Safety 1 | AE16 | Summary of Serious Adverse Events until Week 24 visit by System Organ Class and Preferred Term (Number of Participants and Occurrences) | FDAAA, EudraCT Treatment Emergent AE See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| 3.37. | Safety 1 | AE1 | Summary of Adverse Events until Week 24 visit Leading to Withdrawal from Study by System Organ Class and Preferred Term | IDSL Treatment Emergent AE See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | IA SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.38. | Safety 1 | AE1 | Summary of Adverse Events until Week 24 visit Leading to Withdrawal from Study by System Organ Class and Preferred Term in Blind Phase | Blind Phase (until second dose) See the Section 10.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.39. | Safety 1 | AE1 | Summary of Adverse Events Leading to Withdrawal from Study within 84 days from the initial dose by System Organ Class and Preferred Term | Blind Phase (within 84 days) See the Section 10.4.2. Two treatment arm (240 and 400U) | IA SAC |
| 3.40. | Safety 2 | AE1 | Summary of Adverse Events until Week 24 visit Leading to Withdrawal from Study by System Organ Class and Preferred Term in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | IA SAC |
| Labora | tory: Chemistry | 1 | | | |
| 3.41. | Safety 1 | LB1 | Summary of Chemistry by Visit | Summarize data at Screening Visit and in Blind Phase. | IA SAC |
| 3.42. | Safety 1 | LB1 | Summary of Chemistry Changes from Baseline by Visit | Summarize data in Blind Phase. ICH E3 | IA SAC |
| 3.43. | Safety 1 | LB3 | Summary of Chemistry Shifts from Baseline Relative to Normal Range | | IA SAC |
| 3.44. | Safety 1 | LB15 | Summary of Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 | IA SAC |
| Labora | tory: Hematolo | gy | | | |
| 3.45. | Safety 1 | LB1 | Summary of Haematology by Visit | Summarize data at Screening Visit and in Blind Phase. | IA SAC |
| 3.46. | Safety 1 | LB1 | Summary of Hematology Changes from Baseline | Summarize data in Blind Phase. ICH E3 | IA SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.47. | Safety 1 | LB3 | Summary of Hematology Shifts from Baseline Relative to Normal Range | | IA SAC |
| 3.48. | Safety 1 | LB15 | Summary of Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 | IA SAC |
| Labora | tory: Urinalysis | • | | | |
| 3.49. | Safety 1 | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline | ICH E3 | IA SAC |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 3.50. | Safety 1 | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | This display will be presented if liver events occur. | IA SAC |
| 3.51. | Safety 1 | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | IDSL | IA SAC |
| ECG | | | | | |
| 3.52. | Safety 1 | EG1 | Summary of ECG Findings | Summarize data at Screening Visit and in Blind Phase. IDSL | IA SAC |
| 3.53. | Safety 1 | EG2 | Summary of ECG Values | Summarize data at Screening Visit, in Blind Phase and at Final Visit. | IA SAC |
| 3.54. | Safety 1 | EG2 | Summary of Change from Baseline in ECG Values by Visit | Summarize data in Blind Phase.<br>IDSL | IA SAC |
| Vital Si | gns | | | | |
| 3.55. | Safety 1 | VS1 | Summary of Vital Signs | Summarize data at Screening Visit and in Blind Phase. | IA SAC |
| 3.56. | Safety 1 | VS1 | Summary of Change from Baseline in Vital Signs | Summarize data in Blind Phase.<br>ICH E3 | IA SAC |

207660

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| SpO2 | | | | | |
| 3.57. | Safety 1 | SAFE_T2 | Summary of Value and Change from Baseline in SpO2 | | IA SAC |
| Exposu | re and Treatmo | ent Compliance | | | |
| 3.58. | Safety 1 | SAFE_T3 | Summary of Exposure to Study Treatment | ICH E3 | IA SAC |
| 3.59. | Safety 1 | SAFE_T4 | Summary of Extent of Exposure to Study Treatment by Treatment Cycle and Muscle Region | Include total arm in Open label phase only | IA SAC |
| 3.60. | Safety 1 | SAFE_T4 | Summary of Extent of Exposure to Study Treatment by Treatment Cycle and Joint | Include total arm in Open label phase only | IA SAC |

## 10.12.7.2. Final Analyses

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Advers | e Events (AEs) | | | | |
| 3.61. | Safety 1 | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term in Overall Study Period | ICH E3 Treatment Emergent Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.62. | Safety 1 | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term in Blind Phase | Blind Phase (until second dose) See the Section 10.4.2. Two treatment arm (240 and 400U) | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.63. | Safety 1 | AE1 | Summary of All Adverse Events within 84 days from the initial dose by System Organ Class and Preferred Term in Blind Phase | Blind Phase (within 84 days) See the Section 10.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.64. | Safety 2 | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.65. | Safety 3 | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term in Open Label Phase (3rd Treatment) | Open Label Phase (3rd Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.66. | Safety 4 | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term in Open Label Phase (4th Treatment) | Open Label Phase (4th Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.67. | Safety 1 | AE5A | Summary of All Adverse Events by Maximum Intensity by<br>System Organ Class and Preferred Term in Overall Study<br>Period | ICH E3 Treatment Emergent Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.68. | Safety 1 | AE5A | Summary of All Adverse Events by Maximum Intensity by<br>System Organ Class and Preferred Term in Blind Phase | Blind Phase (until second dose) See the Section 10.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.69. | Safety 1 | AE5A | Summary of All Adverse Events within 84 days from the initial dose by Maximum Intensity by System Organ Class and Preferred Term in Blind Phase | Blind Phase (within 84 days) See the Section 10.4.2. Two treatment arm (240 and 400U) | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.70. | Safety 2 | AE5A | Summary of All Adverse Events by Maximum Intensity by<br>System Organ Class and Preferred Term in Open Label Phase<br>(2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.71. | Safety 3 | AE5A | Summary of All Adverse Events by Maximum Intensity by<br>System Organ Class and Preferred Term in Open Label Phase<br>(3rd Treatment) | Open Label Phase (3rd Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.72. | Safety 4 | AE5A | Summary of All Adverse Events by Maximum Intensity by System Organ Class and Preferred Term in Open Label Phase (4th Treatment) | Open Label Phase (4th Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.73. | Safety 1 | AE3 | Summary of Common (>=3%) Adverse Events by Overall Frequency in Overall Study Period | ICH E3 Treatment Emergent Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.74. | Safety 1 | AE3 | Summary of Common (>=3%) Adverse Events by Overall Frequency in Blind Phase | Blind Phase (until second dose) See the Section 10.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.75. | Safety 1 | AE3 | Summary of Common (>=3%) Adverse Events within 84 days from the initial dose by Overall Frequency in Blind Phase | Blind Phase (within 84 days) See the Section 10.4.2. Two treatment arm (240 and 400U) | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.76. | Safety 2 | AE3 | Summary of Common (>=3%) Adverse Events by Overall Frequency in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.77. | Safety 3 | AE3 | Summary of Common (>=3%) Adverse Events by Overall Frequency in Open Label Phase (3rd Treatment) | Open Label Phase (3rd Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.78. | Safety 4 | AE3 | Summary of Common (>=3%) Adverse Events by Overall Frequency in Open Label Phase (4th Treatment) | Open Label Phase (4th Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.79. | Safety 1 | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term in Overall Study Period | ICH E3 Treatment Emergent Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.80. | Safety 1 | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term in Blind Phase | Blind Phase (until second dose) See the Section 10.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.81. | Safety 1 | AE1 | Summary of All Drug-Related Adverse Events within 84 days from the initial dose by System Organ Class and Preferred Term in Blind Phase | Blind Phase (within 84 days) See the Section 10.4.2. Two treatment arm (240 and 400U) | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.82. | Safety 2 | AE1 | Summary of All Drug-Related Adverse Events by System Organ<br>Class and Preferred Term in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.83. | Safety 2 | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term in Open Label Phase (3rd Treatment) | Open Label Phase (3rd Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.84. | Safety 2 | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term in Open Label Phase (4th Treatment) | Open Label Phase (4th Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.85. | Safety 1 | AE5A | Summary of All Drug-Related Adverse Events by System Organ<br>Class and Preferred Term and Maximum Intensity in Overall<br>Study Period | ICH E3 Treatment Emergent AE See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.86. | Safety 1 | AE5A | Summary of All Drug-Related Adverse Events by System Organ<br>Class and Preferred Term and Maximum Intensity in Blind<br>Phase | Blind Phase (until second dose) See the Section 10.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.87. | Safety 1 | AE5A | Summary of All Drug-Related Adverse Events within 84 days from the initial dose by System Organ Class and Preferred Term and Maximum Intensity in Blind Phase | Blind Phase (within 84 days) See the Section 10.4.2. Two treatment arm (240 and 400U) | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.88. | Safety 2 | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.89. | Safety 2 | AE5A | Summary of All Drug-Related Adverse Events by System Organ<br>Class and Preferred Term and Maximum Intensity in Open Label<br>Phase (3rd Treatment) | Open Label Phase (3rd Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.90. | Safety 2 | AE5A | Summary of All Drug-Related Adverse Events by System Organ<br>Class and Preferred Term and Maximum Intensity in Open Label<br>Phase (4th Treatment) | Open Label Phase (4th Treatment) See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.91. | Safety 1 | AE3 | Summary of Most Common Serious Drug Related Adverse<br>Events by Overall Frequency in Overall Study Period | Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.92. | Safety 1 | AE2 | Summary of Most Common Non-Serious Drug Related Adverse Events by Overall Frequency in Overall Study Period | Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.93. | Safety 1 | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Participant and Occurrences) in Overall Study Period | FDAAA, EudraCT Treatment Emergent AE See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Serious | and Other Sig | nificant Adverse | Events | | |
| 3.94. | Safety 1 | SAFE_T1 | Summary of Adverse Events of Special Interest in Overall Study Period | Treatment Emergent AE See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.95. | Safety 1 | SAFE_T1 | Summary of Adverse Events of Special Interest in Blind Phase | Blind Phase (until second dose) See the Section 10.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.96. | Safety 1 | SAFE_T1 | Summary of Adverse Events of Special Interest within 84 days from the initial dose in Blind Phase | Blind Phase (within 84 days) See the Section 10.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.97. | Safety 2 | SAFE_T1 | Summary of Adverse Events of Special Interest in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.98. | Safety 3 | SAFE_T1 | Summary of Adverse Events of Special Interest in Open Label Phase (3rd Treatment) | Open Label Phase (3rd Treatment) See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.99. | Safety 4 | SAFE_T1 | Summary of Adverse Events of Special Interest in Open Label Phase (4th Treatment) | Open Label Phase (4th Treatment) See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.100. | Safety 1 | AE1 | Summary of Non-Fatal Serious Adverse Events in Overall Study<br>Period | Treatment Emergent AE See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.101. | Safety 1 | AE1 | Summary of Non-Fatal Serious Adverse Events in Blind Phase | Blind Phase (until second dose) See the Section 10.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.102. | Safety 1 | AE1 | Summary of Non-Fatal Serious Adverse Events within 84 days from the initial dose in Blind Phase | Blind Phase (within 84 days) See the Section 10.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.103. | Safety 2 | AE1 | Summary of Non-Fatal Serious Adverse Events in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.104. | Safety 3 | AE1 | Summary of Non-Fatal Serious Adverse Events in Open Label Phase (3rd Treatment) | Open Label Phase (3rd Treatment) See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.105. | Safety 4 | AE1 | Summary of Non-Fatal Serious Adverse Events in Open Label Phase (4th Treatment) | Open Label Phase (4th Treatment) See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.106. | Safety 1 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events in<br>Overall Study Period | Treatment Emergent AE See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.107. | Safety 1 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events in Blind Phase | Blind Phase (until second dose) See the Section 10.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.108. | Safety 1 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events within 84 days from the initial dose in Blind Phase | Blind Phase (within 84 days) See the Section 10.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.109. | Safety 2 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events in Open Label Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.110. | Safety 3 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events in Open Label Phase (3rd Treatment) | Open Label Phase (3rd Treatment) See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.111. | Safety 4 | AE1 | Summary of Drug-Related Non-Fatal Serious Adverse Events in Open Label Phase (4th Treatment) | Open Label Phase (4th Treatment) See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.112. | Safety 1 | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) in Overall Study Period | FDAAA, EudraCT Treatment Emergent AE See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.113. | Safety 1 | AE1 | Summary of Adverse Events Leading to Withdrawal from Study<br>by System Organ Class and Preferred Term in Overall Study<br>Period | IDSL Treatment Emergent AE See the Section 10.4.2 Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.114. | Safety 1 | AE1 | Summary of Adverse Events Leading to Withdrawal from Study by System Organ Class and Preferred Term in Blind Phase | Blind Phase (until second dose) See the Section 10.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.115. | Safety 1 | AE1 | Summary of Adverse Events Leading to Withdrawal from Study within 84 days from the initial dose by System Organ Class and Preferred Term in Blind Phase | Blind Phase (within 84 days) See the Section 10.4.2. Two treatment arm (240 and 400U) | SAC |
| 3.116. | Safety 2 | AE1 | Summary of Adverse Events Leading to Withdrawal from Study<br>by System Organ Class and Preferred Term in Open Label<br>Phase (2nd Treatment) | Open Label Phase (2nd Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| 3.117. | Safety 3 | AE1 | Summary of Adverse Events Leading to Withdrawal from Study<br>by System Organ Class and Preferred Term in Open Label<br>Phase (3rd Treatment) | Open Label Phase (3rd Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.118. | Safety 4 | AE1 | Summary of Adverse Events Leading to Withdrawal from Study by System Organ Class and Preferred Term in Open Label Phase (4th Treatment) | Open Label Phase (4th Treatment) See the Section 10.4.2. Three treatment arms (240, 400 and 240 + 400U) | SAC |
| Laborat | ory: Chemistry | 1 | | | |
| 3.119. | Safety 1 | LB1 | Summary of Chemistry by Visit | Summarize data at Screening Visit, in Blind Phase and at Final Visit. | SAC |
| 3.120. | Safety 1 | LB1 | Summary of Chemistry Changes from Baseline by Visit | Summarize data in Blind Phase and at Final Visit. ICH E3 | SAC |
| 3.121. | Safety 1 | LB3 | Summary of Chemistry Shifts from Baseline Relative to Normal Range | | SAC |
| 3.122. | Safety 1 | LB15 | Summary of Worst Case Chemistry Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 | SAC |
| Laborat | ory: Hematolo | gy | | | |
| 3.123. | Safety 1 | LB1 | Summary of Hematology by Visit | Summarize data at Screening Visit, in Blind Phase and at Final Visit. | SAC |
| 3.124. | Safety 1 | LB1 | Summary of Hematology Changes from Baseline | Summarize data in Blind Phase and at Final Visit. ICH E3 | SAC |
| 3.125. | Safety 1 | LB3 | Summary of Hematology Shifts from Baseline Relative to Normal Range | | SAC |
| 3.126. | Safety 1 | LB15 | Summary of Worst Case Hematology Results Relative to Normal Range Post-Baseline Relative to Baseline | ICH E3 | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Laborat | ory: Urinalysis | <b>5</b> | | | |
| 3.127. | Safety 1 | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline | ICH E3 | SAC |
| Laborat | tory: Hepatobil | iary (Liver) | | | |
| 3.128. | Safety 1 | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | This display will be presented if liver events occur. | SAC |
| 3.129. | Safety 1 | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | IDSL | SAC |
| ECG | | | | | |
| 3.130. | Safety 1 | EG1 | Summary of ECG Findings | Summarize data at Screening Visit, in Blind Phase and at Final Visit. IDSL | SAC |
| 3.131. | Safety 1 | EG2 | Summary of ECG Values | Summarize data at Screening Visit, in Blind Phase and at Final Visit. | SAC |
| 3.132. | Safety 1 | EG2 | Summary of Change from Baseline in ECG Values by Visit | Summarize data in Blind Phase and at Final Visit. IDSL | SAC |
| Vital Sig | gns | | | | |
| 3.133. | Safety 1 | VS1 | Summary of Vital Signs | Summarize data at Screening Visit, in Blind Phase and at Final Visit. | SAC |
| 3.134. | Safety 1 | VS1 | Summary of Change from Baseline in Vital Signs | Summarize data in Blind Phase and at Final Visit. ICH E3 | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| SpO2 | | | | | |
| 3.135. | Safety 1 | SAFE_T1 | Summary of Value and Change from Baseline in SpO2 | | SAC |
| Exposu | re and Treatme | ent Compliance | | | |
| 3.136. | Safety 1 | SAFE_T3 | Summary of Exposure to Study Treatment | ICH E3 | SAC |
| 3.137. | Safety 1 | SAFE_T4 | Summary of Extent of Exposure to Study Treatment by Treatment Cycle and Muscle Region | Include total arm in Open label phase only | SAC |
| 3.138. | Safety 1 | SAFE_T4 | Summary of Extent of Exposure to Study Treatment by Treatment Cycle and Joint | Include total arm in Open label phase only | SAC |

207660

# 10.12.8. Safety Figures

## 10.12.8.1. Interim Analyses

| Safety | Safety Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Chemi | Chemistry | | | | |
| 3.1. | Safety1 | SAFE_F1 | Scatter plot of Chemistry at Week 12 versus Baseline in Blind Phase | | IA SAC |
| Hemat | Hematology | | | | |
| 3.2. | Safety1 | SAFE_F1 | Scatter plot of Hematology at Week 12 versus Baseline in Blind Phase | | IA SAC |

207660

# 10.12.9. ICH Listings

## 10.12.9.1. Interim Analyses

| ICH: L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Partic | ipant Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | IA SAC |
| 2. | ITT1 | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | IA SAC |
| 3. | Screened | ES9 | Listing of Participants Who Were Rescreened | | IA SAC |
| 4. | ITT1 | BL1 | Listing of Participants for Whom the Treatment Blind was Broken | ICH E3 | IA SAC |
| 5. | ITT1 | TA1 | Listing of Planned and Actual Treatments | IDSL | IA SAC |
| Protoc | col Deviations | | | | |
| 6. | ITT1 | DV2 | Listing of Important Protocol Deviations | ICH E3 | IA SAC |
| 7. | ITT1 | IE3 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | ICH E3 | IA SAC |
| Popul | ations Analysed | | | | |
| 8. | Enrolled | SP3 | Listing of Participants Excluded from Any Population | ICH E3 | IA SAC |
| Demo | graphic and Baselir | ne Characteristics | | | |
| 9. | ITT1 | DM2 | Listing of Demographic Characteristics | ICH E3 | IA SAC |
| 10. | ITT1 | DM9 | Listing of Race | ICH E3 | IA SAC |
| Prior a | and Concomitant M | edications | | | |
| 11. | ITT1 | CM3 | Listing of Medications | IDSL | IA SAC |
| 12. | ITT1 | POP_L1 | Listing of Rehabilitation | | IA SAC |

| ICH: L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 13. | ITT1 | Study Specific | Listing of Other Surgical Procedure | | IA SAC |
| Expos | ure and Treatment | Compliance | | | |
| 14. | ITT1 | POP_L2 | Listing of Exposure Data | ICH E3 | IA SAC |
| Efficac | y Endpoints | | | | |
| 15. | ITT1 | EFF_L1 | Listing of Modified Ashworth Scales | <ul><li>Values</li><li>Changes from baseline</li><li>Responders</li></ul> | IA SAC |
| 16. | ITT1 | EFF_L1 | Listing of Disability Assessment Scales | <ul><li>Values</li><li>Changes from baseline</li><li>Main Assessment Parameter</li></ul> | IA SAC |
| 17. | ITT1 | EFF_L1 | Listing of Numeric Rating Scale for pain | <ul><li>Values in each joint</li><li>Changes from baseline in only elbow joint</li></ul> | IA SAC |
| 18. | ITT1 | EFF_L1 | Listing of Clinical Global Impression of Change | CGI by an investigator and a patient Values | IA SAC |
| 19. | ITT1 | EFF_L2 | Listing of Patient-Reported Benefit of Injection | | IA SAC |
| 20. | ITT1 | EFF_L3 | Listing of Time to Patient Reported Onset of Spasticity Symptom Relief | | IA SAC |
| 21. | ITT1 | EFF_L3 | Listing of Time to Qualification for Retreatment | | IA SAC |

| ICH: L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Adver | se Events | | | | |
| 22. | Safety 1 | AE8 | Listing of All Adverse Events until Week 24 visit | ICH E3<br>Including Maximum Intensities,<br>Study Phases for Adverse Events<br>and AESI, SAE flag | IA SAC |
| 23. | Safety 1 | AE7 | Listing of Participant Numbers for Individual Adverse Events until Week 24 visit | ICH E3 | IA SAC |
| 24. | Safety 1 | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | IA SAC |
| Seriou | s and Other Signifi | icant Adverse Eve | nts | | |
| 25. | Safety 1 | AE8 | Listing of Fatal Serious Adverse Events until Week 24 visit | ICH E3<br>Including Study Phases for<br>Adverse Events | IA SAC |
| 26. | Safety 1 | AE8 | Listing of Non-Fatal Serious Adverse Events until Week 24 visit | ICH E3<br>Including Study Phases for<br>Adverse Events | IA SAC |
| 27. | Safety 1 | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | IA SAC |
| 28. | Safety 1 | AE8 | Listing of Adverse Events Leading to Withdrawal from Study until Week 24 visit | ICH E3<br>Including Study Phases for<br>Adverse Events | IA SAC |
| Hepat | obiliary (Liver) | | | | |
| 29. | Safety 1 | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | This display will be presented if liver events occur. | IA SAC |
| 30. | Safety 1 | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | This display will be presented if liver events occur. | IA SAC |
| | | • | · | • | |

207660

| ICH: L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| All Lal | ooratory | • | | | |
| 31. | Safety 1 | LB5 | Listing of All Laboratory Data for Participants with Any Value Outside Normal Range | ICH E3 | IA SAC |
| 32. | Safety 1 | LB14 | Listing of Laboratory Data with Character Results | ICH E3 Except for urinalysis data | IA SAC |
| 33. | Safety 1 | UR2A | Listing of Urinalysis Data for Participants | ICH E3 | IA SAC |
| SpO2 | | | | | |
| 34. | Safety 1 | VS4 | Listing of SpO2 | | IA SAC |

## 10.12.9.2. Final Analyses

| ICH: L | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Partic | ipant Disposition | | | | |
| 35. | ITT1 | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| 36. | Screened | ES9 | Listing of Participants Who Were Rescreened | | SAC |
| 37. | ITT1 | BL1 | Listing of Participants for Whom the Treatment Blind was Broken | ICH E3 | SAC |
| Protoc | Protocol Deviations | | | | |
| 38. | ITT1 | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC |

| ICH: L | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| Popula | ations Analysed | | | | |
| 39. | Enrolled | SP3 | Listing of Participants Excluded from Any Population | ICH E3 | SAC |
| Demo | graphic and Baselin | e Characteristics | | | |
| 40. | ITT1 | DM2 | Listing of Demographic Characteristics | ICH E3 | SAC |
| 41. | ITT1 | DM9 | Listing of Race | ICH E3 | SAC |
| Prior a | and Concomitant Me | edications | | | |
| 42. | ITT1 | CM3 | Listing of Medications | IDSL | SAC |
| 43. | ITT1 | POP_L1 | Listing of Rehabilitation | | SAC |
| 44. | ITT1 | Study Specific | Listing of Other Surgical Procedure | | SAC |
| Expos | ure and Treatment | Compliance | | | |
| 45. | ITT1 | POP_L2 | Listing of Exposure Data | ICH E3 | SAC |
| Efficad | cy Endpoints | | | | |
| 46. | ITT1 | EFF_L1 | Listing of Modified Ashworth Scales | <ul><li>Values</li><li>Changes from baseline</li><li>Responders</li></ul> | SAC |
| 47. | ITT1 | EFF_L1 | Listing of Disability Assessment Scales | <ul><li>Values</li><li>Changes from baseline</li><li>Main Assessment Parameter</li></ul> | SAC |
| 48. | ITT1 | EFF_L1 | Listing of Numeric Rating Scale for pain | <ul><li>Values in each joint</li><li>Changes from baseline in only elbow joint</li></ul> | SAC |

| ICH: L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 49. | ITT1 | EFF_L1 | Listing of Clinical Global Impression of Change | CGI by an investigator and a patient Values | SAC |
| 50. | ITT1 | EFF_L2 | Listing of Patient-Reported Benefit of Injection | | SAC |
| 51. | ITT1 | EFF_L3 | Listing of Time to Patient Reported Onset of Spasticity Symptom Relief | | SAC |
| 52. | ITT1 | EFF_L3 | Listing of Time to Qualification for Retreatment | | SAC |
| Advers | se Events | | | | |
| 53. | Safety 1 | AE8 | Listing of All Adverse Events | ICH E3 Including Maximum Intensities, Study Phases for Adverse Events and AESI, SAE flag | SAC |
| 54. | Safety 1 | AE7 | Listing of Participant Numbers for Individual Adverse Events | ICH E3 | SAC |
| 55. | Safety 1 | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | SAC |
| Seriou | s and Other Signifi | cant Adverse Eve | nts | | |
| 56. | Safety 1 | AE8 | Listing of Fatal Serious Adverse Events | ICH E3<br>Including Study Phases for<br>Adverse Events | SAC |
| 57. | Safety 1 | AE8 | Listing of Non-Fatal Serious Adverse Events | ICH E3<br>Including Study Phases for<br>Adverse Events | SAC |
| 58. | Safety 1 | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC |

| ICH: L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 59. | Safety 1 | AE8 | Listing of Adverse Events Leading to Withdrawal from Study | ICH E3<br>Including Study Phases for<br>Adverse Events | SAC |
| Hepate | obiliary (Liver) | | | | |
| 60. | Safety 1 | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | This display will be presented if liver events occur. | SAC |
| 61. | Safety 1 | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | This display will be presented if liver events occur. | SAC |
| All Lal | ooratory | | | | |
| 62. | Safety 1 | LB5 | Listing of All Laboratory Data for Participants with Any Value Outside Normal Range | ICH E3 | SAC |
| 63. | Safety 1 | LB14 | Listing of Laboratory Data with Character Results | ICH E3 Except for urinalysis data | SAC |
| 64. | Safety 1 | UR2A | Listing of Urinalysis Data for Participants | ICH E3 | SAC |
| Other | Safety | | | | |
| 65. | Safety 1 | EG3 | Listing of All ECG values | | SAC |
| 66. | Safety 1 | EG5 | Listing of All ECG Findings | | SAC |
| 67. | Safety 1 | VS4 | Listing of Vital Signs | | SAC |
| SpO2 | | | | | |
| 68. | Safety 1 | VS4 | Listing of SpO2 | | SAC |

207660

## 10.12.10. Patient Profiles

## 10.12.10.1. Final Analyses

| Patient | Profiles Listing | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable |
| 69. | Safety1 | IDSL standard | Listing of Investigator Reported Cardiovascular Events: Arrhythmias | This display will be presented if at least one event occurs. | SAC |
| 70. | Safety1 | IDSL standard | Listing of Investigator Reported Cardiovascular Events:<br>Congestive Heart Failure | This display will be presented if at least one event occurs | SAC |
| 71. | Safety1 | IDSL standard | Listing of Investigator Reported Cardiovascular Events:<br>Cerebrovascular Events/ Stroke and Transient Ischemic Attack | This display will be presented if at least one event occurs | SAC |
| 72. | Safety1 | IDSL standard | Listing of Investigator Reported Cardiovascular Events: Deep Vein Thrombosis/ Pulmonary Embolism | This display will be presented if at least one event occurs | SAC |
| 73. | Safety1 | IDSL standard | Listing of Investigator Reported Cardiovascular Events:<br>Myocardial Infarction/ Unstable Angina | This display will be presented if at least one event occurs | SAC |
| 74. | Safety1 | IDSL standard | Listing of Investigator Reported Cardiovascular Events: Peripheral Arterial Thromboembolism | This display will be presented if at least one event occurs | SAC |
| 75. | Safety1 | IDSL standard | Listing of Investigator Reported Cardiovascular Events: Pulmonary Hypertension | This display will be presented if at least one event occurs | SAC |
| 76. | Safety1 | IDSL standard | Listing of Investigator Reported Cardiovascular Events: Revascularization | This display will be presented if at least one event occurs | SAC |
| 77. | Safety1 | IDSL standard | Listing of Investigator Reported Cardiovascular Events: Valvulopathy | This display will be presented if at least one event occurs | SAC |
| 78. | Safety1 | IDSL standard | Listing of Investigator Reported Events: Deaths | This display will be presented if at least one event occurs | SAC |

207660

# 10.13. Appendix 13: List of Preferred Terms / System Organ Class of Adverse Events of Special Interest

Adverse Events of Special Interest will be identified based on MedDRA version 20.1.

#### 10.13.1. Convulsions and Seizures

This AESI will be identified using Convulsions (SMQ) with narrow scope.

## 10.13.2. Respiratory Adverse Events

This AESI will be identified using the System Organ Class and High Level Term as below.

SOC: "Respiratory, thoracic and mediastinal disorders"

HLT: "Respiratory and pulmonary function diagnostic procedures"

#### 10.13.3. Possible Distant Spread of Toxin

This AESI will be identified using the Preferred Term as below.

| Accommodation disorder |
|--------------------------------|
| Aspiration |
| Bradycardia |
| Botulism |
| Bulbar palsy |
| Constipation |
| Cranial nerve palsies multiple |
| Cranial nerve paralysis |
| Diaphragmatic paralysis |
| Diplopia |
| Dry mouth |
| Dysarthria |

| Dysphagia |
|------------------------------|
| Dysphonia |
| Dyspnoea |
| Extraocular muscle paresis |
| Eyelid function disorder |
| Eyelid ptosis |
| Facial paresis |
| Facial paralysis |
| Hyporeflexia |
| Hypotonia |
| Illeus paralytic |
| Muscular weakness |
| Paralysis |
| Paresis cranial nerve |
| Pelvic floor muscle weakness |
| Peripheral nerve palsy |
| Peripheral paralysis |
| Pneumonia aspiration |
| Pupillary reflex impaired |
| Respiratory arrest |
| Respiratory depression |
| Respiratory failure |
| Speech disorder |
| Urinary retention |

| Vision blurred |
|----------------------|
| Vocal cord paralysis |
| Vocal cord paresis |

207660

## 10.14. Appendix 14: Decision Tree to determine Data cutoff visit and date

